## **Reporting and Analysis Plan**

**Study ID: 200304** 

**Official Title of Study:** Reporting and Analysis Plan Amendment for 200304: A Phase 3b, randomised, open-label study of the antiviral activity and safety of dolutegravir compared to lopinavir/ritonavir both administered with dual nucleoside reverse transcriptase inhibitor therapy in HIV-1 infected adult subjects with treatment failure on first line therapy

**EudraCT**: 2014-001057-17

**Date of Document**: 31-Jan-2022

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | Ξ | Reporting and Analysis Plan Amendment for 200304: A Phase 3b, randomised, open-label study of the antiviral activity and safety of dolutegravir compared to lopinavir/ritonavir both administered with dual nucleoside reverse transcriptase inhibitor therapy in HIV-1 infected adult subjects with treatment failure on first line therapy |
|---|---|---|
| Compound Number | : | GSK1349572 |
| Effective Date | : | Refer to Document date |

## Description:

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 200304.
- This RAP is intended to describe the planned efficacy, safety & tolerability, virology and health outcome analyses required for the study.
- This RAP will be provided to the study team members to convey the content of IDMC, the Week 24 (interim) and Week 48 (primary) Statistical Analysis Complete (SAC) deliverables.
- This RAP is to provide details of planned analyses and data displays for End of Study (EoS) reporting. These analyses may be included in regulatory submissions, study reports and publications.

#### Author's Name and Functional Area:

| PPD |
|----------------------------------|
| Senior Biostatistician (Parexel) |

### Approved by:

| Approver | Date |
|-------------------------------|------|
| PPD | |
| Senior Manager, Biostatistics | |

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.s

## **TABLE OF CONTENTS**

| TAE | BLE OF CONTENTS | 2 |
|---|---|---|
| 1. | REPORTING & ANALYSIS PLAN SYNPOSIS | 6 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION 2.1. Changes to the Protocol Defined Statistical Analysis Plan 2.2. Study Objective(s) and Endpoint(s) 2.3. Study Design 2.4. Statistical Hypotheses | 8<br>8<br>11 |
| 3. | PLANNED ANALYSES 3.1. Interim Analyses 3.1.1. Week 24 data cut 3.1.2. IDMC interim analyses 3.2. Primary Analyses 3.3. Final Analyses | 12<br>12<br>12 |
| 4. | ANALYSIS POPULATIONS 4.1. Protocol Deviations | |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS | 17 |
| 6. | STUDY POPULATION ANALYSES | |
| 7. | PRIMARY STATISTICAL ANALYSES | 21<br>21 |
| 8. | SECONDARY STATISTICAL ANALYSES 8.1. Efficacy Analyses 8.1.1. Overview of Planned Efficacy Analyses 8.1.2. Planned Efficacy Statistical Analyses 8.2. Safety Analyses 8.2.1. Overview of Planned Analyses 8.2.2. Planned Safety Statistical Analyses | 28<br>30<br>34 |
| 9. | OTHER STATISTICAL ANALYSES 9.1. Health Outcomes Analyses 9.1.1. Overview of Planned Analyses 9.1.2. Planned Health Outcomes Statistical Analyses 9.2. Virology Analyses 9.2.1. Overview of Planned Analyses | 40<br>41<br>43 |
| 10. | REFERENCES | 45 |
| 11. | APPENDICES | 46 |

| 11.1. | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population | 47 |
|---|---|---|
| | 11.1.1. Exclusions from Per Protocol Population | |
| 44.0 | | |
| 11.2. | Appendix 2: Time & Events | |
| 11 2 | Appendix 3: Assessment Windows | |
| 11.3. | • • • | |
| 44.4 | 11.3.1. Definitions of Assessment Windows for Analyses | |
| 11.4. | Appendix 4: Treatment States and Phases | |
| | 11.4.1. Study Phases | |
| | 11.4.3. Post-treatment Assessments and Phases | |
| 11.5. | | |
| 11.5. | Appendix 5: Data Display Standards & Handling Conventions | |
| | 11.5.2. Baseline Definition & Derivations | |
| 44.0 | 11.5.3. Reporting Process & Standards | |
| 11.6. | Appendix 6: Derived and Transformed Data | |
| | 11.6.1. Week 24 cut off date | |
| | 11.6.2. General | |
| | 11.6.3. Study Population | |
| | 11.6.4. Safety | |
| | 11.6.5. Efficacy | |
| | 11.6.6. Virology | |
| 44.7 | 11.6.7. Health Outcomes | |
| 11.7. | Appendix 7: Premature Withdrawals & Handling of Missing Data | |
| | 11.7.1. Premature Withdrawals | |
| 44.0 | 11.7.2. Handling of Missing Data | |
| 11.8. | Appendix 8: Values of Potential Clinical Importance | |
| 11.9. | Appendix 9: Multicenter Studies | |
| 44.40 | 11.9.1. Methods for Handling Centres | |
| 11.10. | Appendix 10: Examination of Covariates, Subgroups & Other Strata | |
| 44.44 | 11.10.1. Handling of Covariates, Subgroups & Other Strata | |
| | Appendix 11: Handling of Multiple Comparisons & Multiplicity | 80 |
| 11.12. | Appendix 12: Model Checking and Diagnostics for Statistical | 07 |
| | Analyses | |
| 44.40 | 11.12.1. Statistical Analysis Assumptions | |
| | Appendix 13: Snapshot | 00 |
| 11.14. | Appendix 14 – Q2 Creatinine Assay Accuracy Issue | |
| 44.45 | 11.14.1. Sensitivity Analyses | 91 |
| 11.15. | Appendix 15 – Abbreviations & Trade Marks | 92 |
| | 11.15.1. Abbreviations | |
| 44.40 | 11.15.2. Trademarks | |
| | Appendix 16 – Example SAS code for Additional Estimand 2 | |
| 11.17. | Appendix 17 – End of Study Analysis | |
| | 11.17.1. General considerations for data analyses | |
| | 11.17.2. Study Population | |
| | 11.17.3. Efficacy Analysis | |
| | 11.17.4. Safety Analysis | |
| | 11.17.5. Virology analysis | 104 |
| | 11.17.6. COVID - 19 analysis | |
| | 11.17.7. Data Displays for End of Study Final Report | |
| 44.40 | 11.17.8. Abbreviations and Trademarks | |
| 11.18. | Appendix 18 –List of Data Displays | 132 |


| | 200304 |
|-----------------------------------------|--------|
| 11.18.1. Data Display Numbering | 132 |
| 11.18.2. Mock Example Shell Referencing | 132 |
| 11.18.3. Deliverable | 133 |
| 11.18.4. Study Population | 134 |
| 11.18.5. Efficacy | |
| 11.18.6. Safety | 153 |
| 11.18.7. Virology | |
| 11.18.8. Health Outcomes | 166 |
| 11.18.9. ICH Listings | 171 |
| 11.18.10. Non-ICH Listings. | |

## Revision History:

The purpose of the latest update (RAP Amendment 2 with EoS Analysis) is to describe the analyses to be included in the End of Study Clinical Study Report based on Study 200304 protocol amendment 3 (19-JUN-2018) - (GlaxoSmithKline Document No.: 2013N172672\_03).

| Revision Chronology: | | |
|---|---|---|
| RAP | 30-Apr-2014 | Reporting and Analysis Plan for Study MID200304 |
| RAP Amendment 1 | 05-Oct-2015 | Amendment to Reporting and Analysis Plan for Study MID200304 (HIV TSQ and Week 48 Snapshot) |
| RAP Amendment 2 | 09-Apr-2017 | Amendment to Reporting and Analysis Plan for Study MID200304 (Switch LPV/RTV to DTG) |
| RAP Amendment 3<br>with EoS Analysis | PPD | Amendment to Reporting and Analysis Plan with End of<br>Study Analysis for Study MID200304 (Appendix 11.17<br>Added) |

## 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP details all planned analyses and outputs required for the Week 24 and Week 48 Clinical Study Reports (CSR) of study 200304. |
| Protocol | This RAP is based on the protocol amendment No. 1 (Dated: 30-APR-2014) of study 200304 (GlaxoSmithKline Document No. : 2013N172672_01) and eCRF Version (Insert Version). |
| Primary<br>Objective | To demonstrate non-inferior antiviral activity at 48 weeks of a DTG containing regimen (DTG 50 mg once daily + two NRTIs) compared to a WHO-recommended standard of care regimen for second line treatment, LPV/RTV + two NRTIs, in HIV-1 infected patients failing first line therapy. |
| Primary<br>Endpoint | <ul> <li>Proportion of subjects with plasma HIV-1 RNA &lt;50 c/mL at Week 48 using the<br/>Snapshot algorithm (Missing, Switch or Discontinuation = Failure) for the intent-<br/>to-treat exposed (ITT-E) population</li> </ul> |
| Study<br>Design | Phase IIIb, randomised, open-label, active-controlled, multicenter, parallel group, non-inferiority study |
| | <ul> <li>Approximately 612 adult patients with confirmed virologic failure (HIV-1 RNA<br/>≥400 c/mL on two occasions) on their first antiretroviral regimen consisting of<br/>one NNRTI + two NRTIs will be recruited.</li> </ul> |
| | <ul> <li>Assuming a true response rate of 70% for both DTG and LPV/r arms, the study<br/>requires 306 subjects per arm to have 90% power with a 12% non-inferiority<br/>margin and a one-sided 2.5% significance level (see Section 8.2.1).</li> </ul> |
| | <ul> <li>Subjects will be randomised 1:1 to receive DTG 50 mg once daily or LPV/RTV (800/200 mg once daily or 400/100 mg twice daily, in accordance with investigator decision and local label), each added to an investigator selected background regimen consisting of two NRTIs with at least one fully active NRTI. In consultation with the medical monitor, 3TC may be added as a third NRTI to a dual-NRTI background regimen in subjects with chronic HBV infection and evidence of HIV resistance to 3TC (e.g. M184V)</li> </ul> |
| Planned<br>Analyses | The primary analysis at Week 48 will take place after the last subject completes 52 weeks on therapy (Day 1 to Week 48 plus a 4-week treatment extension). |
| | An interim analysis and data cut will be conducted after the last subject completes 24 weeks on therapy, with the intent to provide an earlier assessment of efficacy to inform the Sponsor and clinicians. |
| | An IDMC will be instituted to perform periodic reviews of the accumulating data to ensure that subjects are not being sub-optimally treated. |
| Analysis<br>Populations | The 'Intent-to-Treat Exposed Population' (ITT-E) consisting of all randomised subjects who receive at least one dose of study medication, assessed according to their randomised treatment regardless of the treatment they receive, will be the primary analysis population for evaluating efficacy. |

| Overview | Key Elements of the RAP |
|---|---|
| | The 'Per-Protocol Population' consisting of subjects in the ITT-E population with the exception of major protocol violators, e.g. violations that could affect the assessment of antiviral activity will be used for sensitivity analyses of the primary efficacy endpoint. |
| | The 'Safety Population' consisting of all subjects who receive at least one dose of IP, assessed according to the actual treatment received, will be used for evaluating safety and tolerability. Subjects will be analyzed according to the actual treatments received. |
| | The 'Intent-to-Treat Population' consisting of all randomised subjects, assessed according to their randomised treatment even if no study treatment was taken or the wrong treatment was received, will be used for sensitivity analyses of the primary efficacy endpoint. |
| Hypothesis | This study is designed to show that the antiviral effect of a regimen of DTG (administered once daily) + two NRTIs is non-inferior to LPV/RTV + two NRTIs; non-inferiority will be declared if the lower bound of the two-sided 95% CI for the difference in snapshot response rates (DTG – LPV/RTV) is greater than - 12%. The primary analysis will be based on the ITT-E population using the Snapshot dataset at Week 48. The primary comparison will be made at a one-sided 2.5% level of significance. |
| Primary<br>Analyses | The primary endpoint will be analysed using a Cochran-Mantel-Haenszel stratified analysis, adjusting for baseline stratification factors. A point estimate and corresponding 95% confidence interval will be constructed for the adjusted difference in response rates between DTG and LPV/RTV treatment groups. |
| Secondary<br>Analyses | Secondary analyses will be conducted for additional efficacy, safety, health outcomes, and virologic endpoints. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 1 (Dated: 30/APR/2014).

The main changes included in RAP Amendment 1 are:

#### HIV TSQ

The original RAP described analyses for the 10-item HIV TSQ, however the 14-item HIV TSQ is being used in this study.

## • Suspect Creatinine Samples

An issue was identified with the creatinine testing at the central laboratory. Sensitivity analyses will be conducted excluding any suspect creatinine samples from laboratory summaries including creatinine.

## • Week 48 snapshot

Including a summary of week 48 snapshot outcomes in the Week 24 interim.

• Phenotype & genotype data for China subjects

Phenotype data may not be available for all subjects in China at the time of the Week 24 analyses. The China subjects may also have genotype data from Q2 and/or Monogram. In the event that subjects have both Q2 and Monogram data at a timepoint, the Monogram data will be used.

The main changes in RAP Amendment 2 are:

Following Protocol Amendment 2 (Dated: 19/Apr/2017) additional analyses have been included to account for subjects that switch from LPV/RTV to DTG or withdraw from the study due to the IDMC recommendation.

The planned summary by-visit CSSR has been replaced with the IDSL recommended summary.

Other minor changes have been included.

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To demonstrate non-inferior antiviral activity at 48 weeks of a DTG containing regimen (DTG 50 mg once daily + two NRTIs) compared to a WHO-recommended standard of care regimen for second line treatment, LPV/RTV + two NRTIs, in HIV-1 | Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm (Missing, Switch or Discontinuation = Failure) for the ITT-E population |

| Objectives | Endpoints |
|---|---|
| infected patients failing first line therapy. | |
| Secondary Objectives | Secondary Endpoints |
| To demonstrate non-inferior antiviral activity at 24 weeks of a DTG containing regimen (DTG 50 mg once daily + two NRTIs) compared to a recommended WHO standard of care regimen for second line treatment, LPV/RTV + two NRTIs, in HIV-1 infected patients failing first line therapy | Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 24 using the Snapshot algorithm |
| To evaluate the antiviral and immunological activity and incidence of disease progression (HIV-associated conditions, AIDS and death) of DTG compared to LPV/RTV over time | <ul> <li>Proportion of subjects with plasma HIV-1 RNA &lt;400 c/mL at Weeks 24 and 48 using the Snapshot algorithm;</li> <li>Proportion of subjects without virologic or tolerability failure by Weeks 24 and 48, where failure equals treatment-related discontinuation (meeting confirmed virologic withdrawal criteria, treatment-related adverse event, safety stopping criteria, and lack of efficacy);</li> <li>Time to viral suppression (HIV-1 RNA &lt;50 c/mL);</li> <li>Absolute values and changes from Baseline in CD4+ cell counts at Weeks 24 and 48;</li> <li>Incidence of disease progression (HIV-associated conditions, AIDS and death).</li> </ul> |
| To assess the development of viral<br>resistance in subjects meeting<br>confirmed virologic withdrawal criteria; | Incidence of treatment-emergent genotypic and phenotypic resistance to DTG, LPV/RTV and other onstudy ART in subjects meeting confirmed virologic withdrawal criteria. |
| To evaluate the safety, tolerability,<br>and laboratory parameters of DTG<br>compared to LPV/RTV over time | <ul> <li>Incidence and severity of AEs and laboratory abnormalities;</li> <li>Absolute values and changes over time in laboratory parameters;</li> <li>The proportion of subjects who discontinue treatment due to AEs.</li> </ul> |
| To compare the effects of DTG and<br>LPV/RTV on fasting lipids over time | <ul> <li>Change from Baseline in fasting LDL cholesterol at Weeks 24 and 48;</li> <li>Change from Baseline in fasting TC/HDL ratio at Weeks 24 and 48;</li> <li>The incidence of maximum post-Baseline emergent Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Weeks 24 and 48;</li> </ul> |
| To compare the effects of DTG and<br>LPV/RTV on the occurrence of<br>gastrointestinal adverse events over<br>time | The incidence of maximum post-Baseline emergent<br>Grade 2 or greater drug-related diarrhoea by Weeks 24<br>and 48 |
| To compare the change in<br>gastrointestinal symptom rating score<br>for subjects treated with DTG and<br>LPV/RTV over time | Change from Baseline, using the Gastrointestinal<br>Symptom Rating Scale (GSRS), at Week 4, Week 24,<br>and Week 48 |
| To compare the satisfaction with | Change from Baseline in treatment satisfaction, using the |


| Objectives | Endpoints |
|---|---|
| treatment of patients with DTG compared to the LPV/RTV over time | HIV-Treatment Satisfaction Questionnaire (HIVTSQ), at Week 4, Week 24, and Week 48 |
| To compare patients' adherence with<br>DTG compared to LPV/RTV over time | Change from Baseline in adherence with treatment, using<br>the Morisky 8-Item Medication Adherence Scale (MMAS-8), at Week 4, Week 24, and Week 48. |
| To evaluate the effect of patient<br>demographics and baseline<br>characteristics (e.g. demographic<br>factors, HIV-1 subtype, baseline CD4+<br>cell count) on response to DTG<br>compared to LPV/RTV over time | Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Weeks 24 and 48 using the Snapshot algorithm |

## 2.3. Study Design



## **Overview of Study Design and Key Features**

An IDMC will be utilised in this study to ensure external objective medical and/or statistical review of safety and/or efficacy issues in order to protect the ethical and safety interests of subjects and to protect the scientific validity of the study. Planned stopping guidelines and schedule for interim analyses are provided in Section 8.3.4.2 of the Protocol.

## 2.4. Statistical Hypotheses

This study is designed to show that the antiviral effect of a regimen of DTG (administered once daily) + two NRTIs is non-inferior to LPV/RTV + two NRTIs.

If  $r_d$  is the response rate on DTG + two NRTIs and  $r_a$  is the response rate on LPV/RTV + two NRTIs then the hypotheses can be written as follows:

H1:  $r_d - r_a > -12\%$ .

H0: 
$$r_d - r_a \le -12\%$$

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

The main analysis will be conducted to evaluate the primary objective of the protocol when all subjects have completed their Week 52 visit.

#### 3.1.1. Week 24 data cut

An interim analysis will be conducted in order to provide an earlier assessment of efficacy to inform the Sponsor and clinicians after the following activities have been carried out:

- 1. All subjects have completed their Week 24 visit.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. Randomisation codes have been distributed according to RandAll NG procedures
- 4. All criteria for unblinding the randomisation codes have been met.

The analyses described in Section 7.1 and Section 8.1 will be performed with the sole difference being that the timepoint for these analyses will be Week 24 instead of Week 48.

No adjustment for multiplicity will be made for this analysis because the Week 24 endpoints represent secondary objectives for the study which are subordinate to the primary analysis at Week 48.

## 3.1.2. **IDMC interim analyses**

An IDMC has been instituted to provide independent review of the accumulating data, primarily to ensure subjects are not being sub-optimally treated in either arm.

Three formal interim analyses are planned for review by the IDMC (Table 1). Additional details are provided in the protocol and IDMC charter.

Table 1 Timing of Planned IDMC Interim Analyses and Stopping Guidelines

| Analysis | | | |
|---|---|---|---|
| #1 | Once 100 subjects (total)<br>have completed their Week<br>16 visit | Proportion of subjects with<br>HIV-1 RNA <50 c/mL<br>at Week 16<br>(Snapshot algorithm) | Inferiority <sup>a</sup> (one-sided p<0.01) |
| #2 | Once 300 subjects (total)<br>have completed their Week<br>24 visit | Proportion of subjects with<br>HIV-1 RNA <50 c/mL<br>at Week 24<br>(Snapshot algorithm) | Inferiority <sup>a</sup> (one-sided p<0.01) |
| <del>#3</del> | Once all subjects have completed their Week 24 visit | Proportion of subjects with<br>HIV-1 RNA <50 c/mL<br>at Week 48<br>(Snapshot algorithm) | <ul> <li>Inferiority<sup>a</sup> (one-sided p&lt;0.01)</li> <li>Superiority<sup>b</sup> (one-sided p&lt;0.0001)</li> </ul> |

At time of finalisation of Protocol Amendment 2, the IDMC had completed interim analyses #1 and #2. Prior to interim analysis #3, the IDMC conducted an ad hoc review of trial data and observed significant, clinically relevant differences between treatment arms in favour of DTG. The IDMC recommended to the sponsor that the LPV/RTV treatment arm be discontinued and subjects currently receiving LPV/RTV in the study be switched to a regimen with DTG as the third drug, if considered appropriate by the Investigator. Interim analysis #3 will no longer take place.

## 3.2. Primary Analyses

The planned primary analyses will be performed after:

- 1. All subjects have completed their Week 52 visit as defined in the protocol.
- 2. All required database cleaning activities have been completed and database release and database freeze has been declared by Data Management.

## 3.3. Final Analyses

A final End-of-Study analysis will be conducted when all subjects have completed the study as defined in Section 3.1 of the Protocol.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Screened | Comprised of all subjects screened for inclusion in the study. | Study Population |
| | Subjects may be re-screened once, for which they will receive a new subject number. | |
| | Only the latest re-screening data will be included in the screening population summaries/analyses but all screening data will be listed. | |
| Intent-to-Treat<br>Exposed (ITT-E) | Comprise of all randomised subjects who receive at least one dose of study medication. | <ul><li>Efficacy</li><li>Health Outcome</li></ul> |
| | Subjects will be assessed according to their randomised treatment, regardless of the treatment they receive | Study population |
| Safety | Comprise of all subjects who receive at least one dose of investigational product | Safety |
| | Subjects will be analyzed according to the actual treatments received. | |
| Intent-To-Treat | Comprise of all randomised subjects. | Sensitivity analyses |
| (ITT) | Subjects will be assessed according to their randomised treatment even if no study treatment was taken or the wrong treatment was received. | of the primary efficacy endpoint |
| Week 36 Intent-<br>to-Treat Exposed<br>(MITT-E-36) | Comprise all subjects in the ITT-E population randomised at least 36 weeks prior to 18 Jan 2017 (the last subject visit date for the Week 24 study report), excluding subjects still onstudy in the randomised phase that had yet to provide a Week 36 HIV-1 RNA result by the Week 24 study report cutoff date. | Week 36 snapshot<br>outcomes for Week<br>24 study report. |
| Week 48 Intent-<br>to-Treat Exposed<br>(MITT-E-48) | Comprise all subjects in the ITT-E population randomised at least 48 weeks prior to 18 Jan 2017 (the last subject visit date for the Week 24 study report), excluding subjects still onstudy in the randomised phase that had yet to provide a Week 48 HIV-1 RNA result by the Week 24 study report cutoff date. | Week 48 snapshot<br>outcomes for Week<br>24 study report. |
| Per-Protocol | Comprise of all subjects in the ITT-E population with the exception of major protocol violators, e.g. violations which could affect the | Sensitivity analyses<br>of the primary<br>efficacy endpoint |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | assessment of antiviral activity. | |
| | Protocol deviations that would exclude subjects from the PP population are defined in Section 4.1 (Protocol Deviations) and Appendix 1 (Protocol Deviation Management and Definition for Per-Protocol Population). | |
| | Only protocol deviations that occur duing the randomised phase and before the outcome of interest may lead to exclusion from the PP population. For example, a subject with a protocol deviation between Week 24 and Week 48 would not be excluded from the Week 24 PP Population, due to this deviation, but would be excluded from the Week 48 PP Population | |
| Viral Genotypic | Comprise of all subjects in the ITT-E population with available On-treatment genotypic resistance data at the time confirmed virologic withdrawal criterion is met | Genotypic |
| Viral Phenotypic | Comprise of all subjects in the ITT-E population with available On-treatment phenotypic resistance data at the time confirmed virologic withdrawal criterion is met | Phenotypic |

#### NOTES:

 Please refer to Appendix 18 List of Data Displays which details the population to be used for each displays being generated.

### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population)].
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - O Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the perprotocol analysis are captured and categorised on the protocol deviations dataset. This dataset will be the basis for the summaries and listings of protocol deviations.


200304

• A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

- There are planned examination of covariates and subgroups.
- There are no planned adjustments made for multiple centres in this study.
- There are no planned adjustments for multiple comparisons or multiplicity.
- There are no PK analyses planned in this study.

Table 2 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 2 Overview of Appendices

| Section | Component |
|---|---|
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| Section 11.2 | Appendix 2: Time & Events |
| Section 11.3 | Appendix 3: Assessment Windows |
| Section 11.4 | Appendix 4: Treatment States and Phases |
| Section 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 11.6 | Appendix 6: Derived and Transformed Data |
| Section 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| Section 11.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 11.9 | Appendix 9: Multicenter Studies |
| Section 11.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| Section 11.11 | Appendix 11: Handling of Multiple Comparisons & Multiplicity |
| Section 11.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Section 11.13 | Appendix 13: Snapshot |
| Section 11.14 | Appendix 14: Q2 Creatinine Assay Accuracy Issue |
| Section 11.15 | Appendix 15 Abbreviations & Trade Marks |
| Section 11.16 | Appendix 16: Example SAS code for Additional Estimand 2 |
| Section 11.17 | Appendix 17: End of Study Analysis |
| Section 11.18 | Appendix 18: List of Data Displays |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

All displays are for the randomised phase only, unless specified otherwise. This means that the analysis will not be "windowed" at Week 24 ie all data collected up to the point of Database Freeze for Week 24will be included in summary statistics, which could be past week 24 for subjects enrolled early in the study. However, in the Week 48 report, the analysis will be "windowed", ie summary statistics will include data up to Week 52 only for both arms.

Table 3 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 18 List of Data Displays.

 Table 3
 Overview of Planned Study Population Analyses

| Display Type | Data | Display's Gen | erated |
|---|---|---|---|
| | Figure | Table | Listing |
| Randomisation | | | |
| Randomisation | | | Υ[1] |
| Subject Disposition | | | |
| Study population <sup>[2]</sup> | | Υ | Υ [3] |
| Summary of Subjects Enrolled by Country and Investigator [2] | | Υ | Y |
| Study recruitment by age (EMA) | | Υ | |
| Reasons for Screening Failures [2] | | Υ | Υ |
| Subject Accountability by Phase (Overall, Randomised Phase, Continuation Phase) <sup>[4]</sup> | | Υ | |
| Reasons for Withdrawals by visit | | Υ | Υ |
| Study visit dates | | | Υ |
| Important Protocol Deviations | | Υ | Υ |
| Deviations Leading to Exclusions from PP Population | | Υ | Υ |
| Inclusion and Exclusion Criteria Deviations | | Υ | Υ |
| Drug Accountability | | | |
| Investigational Product Accountability <sup>[5]</sup> | | | Υ |
| Demography | | | |
| Demographics Characteristics <sup>[6]</sup> | | Υ | Υ |
| Race & Racial Combinations <sup>[7]</sup> | | Y x2 | Υ |
| CDC Classification of HIV Infection at Baseline | | Υ | Υ |
| Baseline Cardiovascular Risk Assessments | | Υ | Υ |

| Display Type | Data Display's Generated | | |
|---|---|---|---|
| | Figure | Table | Listing |
| Plasma HIV-1 RNA Results at Screening and Baseline | | Υ | |
| CD4+ Cell Count Results at Screening and Baseline | | Υ | |
| Hepatitis Status at Entry | | Υ | Y |
| History of Cardiac Therapeutic Procedures | | | Y |
| Medical Condition & Concomitant Medications | | | |
| Medical Conditions (Current/Past) | | Υ | <b>Y</b> [9] |
| Medical Conditions: sub-conditions (Current/Past) | | Υ | Y |
| Concomitant Medication (non ART) | | Yx3 <sup>[10]</sup> | Υ[11,9] |
| Prior Antiretroviral Therapy (including Duration) | | Yx4 | Y[11] |
| Baseline Background Antiretroviral Therapy (including conART) | | Υ | Y[11] |
| Lipid Modifying Agent Use (Starting Baseline/Post-Baseline) | | Υ | Υ |
| Virology | | • | |
| Summary of the Number of Baseline Major Mutations Associated with the Resistance to NRTI, NNRTI, and PI drug classes | | Yx2 <sup>[8]</sup> | |
| Proportion of subjects without at least 1 fully active NRTI | | Y | |
| Summary of Baseline Major NNRTI and NRTI<br>Mutations | | Y | |
| Summary of Stanford Baseline GSS to Background ART Regimen | | Υ | |
| Summary of Monogram Baseline GSS to Background ART Regimen | | Υ | |
| Summary of Baseline PSS to Background ART Regimen | | Υ | |
| Summary of Baseline OSS (Net Assessment) to Background Therapy | | Υ | |
| Summary of the Prevalence of HIV-1 Clades at Baseline by Frequency | | Υ | |
| Summary of First Line Regimen and Expected Second Line Regimen Using the WHO Algorithm <sup>[12]</sup> | | Υ | |
| Summary of Expected WHO Second Line vs. Background Regimen actually Taken <sup>[12]</sup> | | Y | |

#### NOTES:

- Y = Yes display generated, T = Tables, L = Listings, IP = Investigational Product.
- 1. One listing of subjects randomised but not treated, and one listing of planned and actual treatment strata
- 2. All subject screened population
- 3. Listing of subjects excluded from any population will be generated only.
- 4. Subjects who have not been recorded as either completing or withdrawing from the study will be categorised as "Ongoing at time of the analysis" for summary purposes.
- 5. Dispensation information (dates and number of tablets dispensed and returned)
- 6. Gender, age, ethnicity, weight and height collected at screening (Day 1 for height)
- 7. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- 8. Repeated for screening mutation for the Screen Failure population.
- 9. Repeated for Mexican subjects who experienced an adverse event at the End of Study SAC.
- 10. Three separate tables, summarised by Ingredient ATC Level 1, Ingredient combinations and Combination term ATC Level 1 (EG Includes single-ingredient medications with multi-ingredient medications labelled according to the sum of their ingredients, e.g., "TYLENOL Cold and Flu" would appear as "CHLORPHENAMINE MALEATE + DEXTROMETHORPHAN HYDROBROMIDE + PARACETAMOL + PSEUDOEPHEDRINE HYDROCHLORIDE" under the ATC headings for "Nervous System" and "Respiratory System" (the combination's ATC classifications).)
- One listing for concomitant non-ART medications, prior ART, background ART and one listing showing the relationship between verbatim text, ingredient and ATC Level 1.
- 12. WHO First and Second Line Regimens are defined in Appendix 6.

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Efficacy Analyses

## 7.1.1. Overview of Planned Efficacy Analyses

The primary efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Summaries will be presented by treatment group with no total column.

The primary estimand and additional estimands for the Week 48 deliverables is presented in Table 4 below. For all estimands, the population of interest (ITT-E population), variable (plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm), and summary measure (proportion of subjects with response) will be the same. All estimands will account for discontinuation (other than due to IDMC recommendation) and non-permitted changes in background ART, as per the snapshot algorithm.

Table 4 Primary and Additional Estimands for the Week 48 Deliverable

| Type of<br>Estimand | Post-baseline Intervention of interest |
|---|---|
| Primary | No additional post baseline interventions considered. |
| | Subjects will be analysed according to their original treatment assignment regardless of treatment switch. |
| Additional | Additional Estimand 1 |
| | In addition, accounting for subjects that switch from LPV/RTV to DTG or withdraw from the study due to the IDMC recommendation (and subsequent Protocol Amendment 2). HIV-1 RNA values collected after treatment switching or discontinuation will be excluded from the analyses. |
| Additional | Additional Estimand 2 |
| | In addition, for subjects that switch from LPV/RTV to DTG or withdraw from the study due to the IDMC recommendation (and subsequent Protocol Amendment 2), their subsequent HIV-1 RNA values will be replaced with imputed values. |

Table 5 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 18: List of Data Displays.

Table 5 Overview of Planned Efficacy Analyses

| Endpoint | S | tats Analysi | S | Summary | | Individual | |
|---|---|---|---|---|---|---|---|
| • | T | F | L | T | F | F | L |
| Proportion of<br>subjects with plasma<br>HIV-1 RNA <50 c/mL<br>at Week 48 using the | <b>Y</b> [1] | | | <b>Y</b> [2] | ΥŪ | | <b>Y</b> [2] |
| Snapshot algorithm | | | | | | | |
| Treatment Heterogeneity across randomisation strata | Y | | | | | | |
| Study Outcome<br>based on the<br>Snapshot | | | | Υ[4] | | | Y |
| Study Outcome based on the Snapshot by number of fully active background NRTIs | | | | Y | | | |
| Proportion <50 c/mL<br>at Week 48 by<br>subgroup <sup>[5]</sup> | | | | Y | Υ[6] | | |
| Summary of Study<br>Outcomes based on<br>the Snapshot at<br>Week 48 by<br>Subgroup | | | | Y | | | |
| Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm – Additional Estimand 1 <sup>[7]</sup> | <b>Y</b> [1] | | | <b>Y</b> [2] | | | |
| Study Outcome<br>based on the<br>Snapshot –<br>Additional Estimand | | | | Y[4] | | | |
| Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm – Additional Estimand 2 [7] | <b>Y</b> [1] | | | <b>Y</b> [2] | | | |
| Study Outcome | | | | <b>Y</b> [4] | | | Υ |

| Endpoint | Stats Analysis T F L | nt Stats Analysis Summary | | Individual | |
|---|---|---|---|---|---|
| • | | T | F | F | L |
| based on the<br>Snapshot –<br>Additional Estimand<br>2 <sup>[7]</sup> | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Statistical analysis displays will be generated using the 'Intent-to-Treat Exposed' (primary), 'Per-Protocol' and 'Intent-to-Treat' (sensitivity) populations.
- 2. Study outcomes (i.e., response below 50 c/mL, virologic failure or reason for no data in the window) based on the snapshot algorithm will be summarised and listed.
- 3. Line plots, with 95% confidence intervals, for the proportion of subjects below 50 c/mL by treatment group at each visit will be produced.
- 4. This summary will be produced for the week 24 study report.
- 5. Baseline demography (age, gender, race, country, CDC), HIV-1 subtype, Baseline CD4 and Baseline viral load, background ART (ABC+3TC vs not ABC+3TC).
- 6. Plot of 95% confidence intervals for the proportion of subjects below 50 c/mL by subgroup.
- 7. This summary will be produced for the week 48 study report.

## 7.1.2. Planned Efficacy Statistical Analyses

## **Primary Statistical Analyses**

## Endpoint(s)

 Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm (Missing, Switch or Discontinuation = Failure) for the ITT-E population

## **Snapshot Dataset**

- The Snapshot algorithm treats all subjects without HIV-1 RNA data at the visit of interest (due
  to missing data or discontinuation of IP prior to the visit window) as non-responders, as well as
  subjects who switch their concomitant ART prior to the visit of interest in certain
  scenarios(Section 11.13).
- Switch from 3TC to FTC (or vice versa) will not be considered a background NRTI change and will not incur a penalty as per the FDA's Snapshot algorithm.
- Otherwise, virologic success or failure will be determined by the last available HIV-1 RNA
  assessment while the subject is On-treatment within the visit of interest analysis window (see
  Section 11.4.2) Full details of the Snapshot algorithm are in Section 11.13.
- For subjects that switch from LPV/RTV to DTG, any subsequent HIV-1 RNA values will be left as is then virologic response or failure will be determined at Week 48 using snapshot algorithm, with subjects presented by their original randomised treatment..

#### •

### **Model Specification**

 The primary endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for Baseline plasma HIV-1 RNA (≤ vs. >100,000 c/mL)

## **Primary Statistical Analyses**

and number of fully active background NRTIs in the background regimen (<2 vs. 2) at Baseline.

- The CMH estimate of the adjusted treatment difference will be calculated as a weighted average of strata-specific estimates of the treatment difference calculated within each of the following four Baseline analysis strata:
  - o Plasma HIV-1 RNA ≤ 100,000 c/mL AND <2 fully active background NRTIs
  - Plasma HIV-1 RNA ≤ 100,000 c/mL AND 2 fully active background NRTIs
  - Plasma HIV-1 RNA > 100,000 c/mL AND <2 fully active background NRTIs</li>
  - Plasma HIV-1 RNA > 100,000 c/mL AND 2 fully active background NRTIs
- If n<sub>k</sub> is the number of DTG treated subjects, m<sub>k</sub> is the number of LPV/RTV treated subjects, and N<sub>k</sub> = n<sub>k</sub> + m<sub>k</sub> is the total number of subjects in the kth stratum, then the CMH estimate is given by

$$\hat{d}_{cmh} = \frac{\sum W_k \hat{d}_k}{\sum W_k}$$

• Where,

$$W_k = \frac{n_k m_k}{N_k}$$

are CMH weights and  $d_k$  are estimates of the differences in response proportions between the two treatment arms,  $r_d$ - $r_a$ , for the kth strata.

• The corresponding two-sided 95% CI will be calculated as

$$\hat{d}_{cmh} \pm 1.96 \times \sqrt{\hat{\text{var}}(\hat{d}_{cmh})}$$

using the variance estimator, var(d<sub>cmh</sub>), given by [Sato, 1989], which is consistent in both sparse data and large strata. The full equation for this variance estimate is provided in the Appendix 6 (Section 11.6.5).

For analysis purposes, fully active NRTI is defined at Baseline by the genotypic resistance
reports of the central laboratory (or a laboratory contracted by the central laboratory) showing
no evidence of full or of partial genotypic resistance for a given NRTI. If Baseline genotypic
results are not available, then activity of the background regimen will be based on genotypic
results at Screening.

#### **Model Results Presentation**

- Adjusted CMH estimate of the difference in the proportion of responders between each treatment group (DTG – LPV/RTV) and corresponding 95% confidence interval
- Non-inferiority will be concluded if the lower bound of the two-sided 95% confidence interval (CI) for the CMH adjusted difference in the proportion of patients who respond in the DTG group minus the proportion of patients who respond in the LPV/RTV group is greater than -

## **Primary Statistical Analyses**

12%.

## **Sensitivity and Supportive Statistical Analyses**

- Treatment Heterogeneity across randomisation strata:
  - Randomization strata will be re-derived using Baseline values (Section 11.10.1).
  - The weighted least squares chi-squared statistic [Fleiss, 1981] will be used to test for oneway homogeneity across the levels of each categorical variable of the randomisation strata, with each categorical variable considered separately.
  - Following Lui and Kelly [Lui, 2000], ½ will be added to each cell in any strata for which the stratum-specific rate estimates of either rd or ra are zero or one, and tests will be onesided.
  - Any heterogeneity found to be statistically significant will be explored and if necessary
    results will be reported for each level of the categorical variable. Investigation of
    heterogeneity will be confined to the primary endpoint at week 24/48. Tests of
    homogeneity will be assessed at the one-sided 10% level of significance.
- Per-protocol population analysis:
  - To assess the impact of major protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis. If both analyses show non-inferiority then the hypothesis that the antiviral effect of treatment with DTG + two NRTIs is superior to treatment with LPV/RTV + two NRTIs will be tested at the two-sided 5% level of significance. Superiority will be declared if the lower end of the confidence internal is above 0% for the ITT-E population analysis.
- Intent-to-Treat population analysis:
  - Statistical analysis will be repeated using the Intent-to-Treat population and compared for consistency with the results from the ITT-E and PP populations.
  - In this analysis, subjects randomised but not exposed to study treatment will be classified
    as non-responders, which therefore conservatively addresses any selection bias that may
    occur given the open-label study design.
- Exploration of Subgroups:
  - A simple analysis for all the subgroups listed in Section 11.10.1 will be performed. This will show the proportion of subjects with plasma HIV-1 RNA <50 c/mL at the time of analysis (Week 24/48) based on the Snapshot algorithm will be presented by treatment group.
  - Unadjusted difference in proportions between treatment groups and corresponding twosided 95% CI will also be presented by subgroup, and a 95% CI for the (unadjusted) treatment difference in each subgroup. These results will also be presented graphically.
  - If the basic summary suggests an interaction, then a corresponding summary of study outcomes (i.e., response below 50 c/mL, virologic failure or reason for no data in the window) by subgroup will be produced.

Note: These subgroup analyses will be exploratory and likely underpowered so that interpretation may therefore focus on point estimates as well as the lower bounds of 95% CIs for the treatment differences and response rates. Additionally, multiple comparisons are being

### **Sensitivity and Supportive Statistical Analyses**

made which inflates the risk of false positive findings. Therefore, if consistent findings across the multiple comparisons were observed then these analyses would still be suggestive of a generalizable finding of non-inferiority.

- Supportive analysis for the Week 48 deliverable:
  - Additional Estimand 1: Following the IDMC recommendation (and subsequent Protocol Amendment 2), subjects may switch from LPV/RTV to DTG or withdraw from the study. Therefore, prior to the application of the Snapshot algorithm for the Week 48 deliverable, the following step will be undertaken:
    - For subjects that switch from LPV/RTV to DTG, any subsequent HIV-1 RNA values will be set to missing before the Snapshot algorithm is applied.
    - Note: for subjects that withdraw, the Snapshot algorithm will be applied as usual.
  - The population of interest (ITT-E population), variable (plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm), and summary measure (proportion of subjects with response) will be the same as that used for the primary endpoint.
  - Additional Estimand 2: For subjects that switch from LPV/RTV to DTG or withdraw from the study due to the IDMC recommendation (and subsequent Protocol Amendment 2), their subsequent HIV-1 RNA values will be imputed prior to determination of virologic response or failure at Week 48 using snapshot algorithm. See below for more details.

## Additional Estimand 2 – Statistical Analyses

#### **Endpoint**

 Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm

### Covariates

- Baseline Plasma HIV-1 RNA (≤ vs. >100,000 c/mL)
- Baseline Number of Fully Active NRTIs in the Background Regimen (2 vs.<2)</li>

### Input Dataset, Imputation, and Statistical Analysis

- Select Log(HIV-1 RNA) samples and subset by treatment
- For the LPV/RTV arm:
  - For subjects that switch from LPV/RTV to DTG or withdraw from the study due to the IDMC recommendation, set any subsequent HIV-1 RNA values to missing
  - Using Markov Chain Monte Carlo methods, simulate 100 datasets replacing Below Limit of Quantification (BLQ) values with those from a Log(Uniform(0, BLQ) distribution. The BLQ value used for this step should be slightly below the actual BLQ cut-off so that response is correctly attributed when applying the snapshot algorithm later.
  - The statistical model used for the MI data generation will be the Markov Chain Monte Carlo (MCMC) method with for the data (covariates and Log HIV-1 RNA at Baseline, Week 4, Week 8, Week 16, Week 24, Week 36, Week 48, and Week 52) to produce a monotone pattern first, and then the imputation will continue using the Regression (REG) method for the monotone pattern with the same set of

## Additional Estimand 2 – Statistical Analyses

covariates.

- A seed of 200304 will be used in the SAS program.
- One imputation is required for each of the monotone and mean matching steps
- Since it is likely that subject discontinuation or switches treatment due to IDMC recommendation will be based on observed viral load counts, the missing at random (MAR) assumption is appropriate
- o For subjects that originally had missing HIV-1 RNA data within the Week 48 window but did not discontinue or switch from LPV/RTV to DTG arms due to the IDMC recommendation, replace the imputed data with their original data. Data related to these subjects will be used only for the imputation of data for those that switch from LPV/RTV to DTG or withdraw from the study due to the IDMC recommendation
- Log(HIV-1 RNA) data for subjects randomised to the DTG arm is merged back onto each imputed dataset.
- Using Snapshot Algorithm, derive virologic response or failure at Week 48 using snapshot algorithm, as per Section 11.13, for each imputed dataset.
- For each imputed dataset, the endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for Baseline plasma HIV-1 RNA ( ≤ vs. >100,000 c/mL) and number of fully active background NRTIs in the background regimen (<2 vs. 2) at Baseline. This will be the same model as used for the primary endpoint.
- Wilson-Hilferty transformation will be applied to normalise the CMH statistic
- PROC MIANALYZE in SAS will be used to combine the 1,000 estimated proportion of subjects with plasma HIV-1 RNA <50 c/mL and difference in proportions to produce one estimate with 95% CI and associated p-value for the adjusted difference between each treatment group at Week 48

See 11.16 for example SAS code.

## 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Efficacy Analyses

## 8.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

All displays are for the randomised phase only, unless specified otherwise. This means that the analysis other than "by-visit" summaries will not be windowed at Week 24 (CVW, time to suppression). In other words, all data collected up to the point of DBF will be included in summary statistics, which could be past week 24 for subjects enrolled early in the study. However, at the Week 48 analysis, summary statistics will include data up to Week 52 for both arms.

Table 6 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 18: List of Data Displays.

Table 6 Overview of Planned Efficacy Analyses

| Endpoints | S | tats Analysis | 3 | Summary | | Individual | |
|---|---|---|---|---|---|---|---|
| | T | F | L | T | F | F | L |
| <b>Proportion of Subjects</b> | with Plasm | a HIV-1 RN | A <50 copi | es/mL at We | eek 24- Snap | oshot | |
| Proportion of | Υ | | | Υ | Υ | | <b>Y</b> [2] |
| subjects with plasma | | | | | | | |
| HIV-1 RNA <50 c/mL | | | | | | | |
| at Week 24 using the | | | | | | | |
| Snapshot | | | | | | | |
| algorithm <sup>[1]</sup> | | | | | | | |
| Treatment | Υ | | | | | | |
| Heterogeneity across | | | | | | | |
| randomization strata | | | | | | | |
| Study Outcome | | | | Y | | | |
| based on the | | | | | | | |
| Snapshot by number | | | | | | | |
| of fully active | | | | | | | |
| background NRTIs | | | | | | | |
| Proportion <50 c/mL | | | | Υ | Υ | | |
| at Week 24 by | | | | | | | |
| subgroup <sup>[3]</sup> | | | | | | | |
| Proportion of Subjects | | | | Y | | | |
| with Plasma HIV-1 | | | | | | | |
| RNA <50 c/mL by Visit | | | | | | | |
| and Subgroup - | | | | | | | |
| Snapshot | | | | | 1 00/10 0 | | |
| Proportion of Subjects | | a HIV-1 RN | A <50 copi | es/mL at We | eek 36/48- S | napshot, at | time of |
| Week 24 interim analys | SIS <sup>[7,0]</sup> | | | | | <u> </u> | 1 |
| Proportion of | | | | | | | |

| Endpoints | St | ats Analysis | 3 | Summary | | Individual | |
|---|---|---|---|---|---|---|---|
| | T | F | L | Т | F | F | L |
| subjects with plasma | | | | | | | |
| HIV-1 RNA <50 c/mL | | | | | | | |
| at Week 36/48 using | | | | | | | |
| the Snapshot | | | | | | | |
| algorithm[1][9] | | | | | | | |
| <b>Proportion of Subjects</b> | with Plasma | a HIV-1 RN | <b>4 &lt;400 &amp; &lt;</b> | <50 copies/m | L - Snapsho | ot | |
| <50 c/mL by Visit | | | | Υ | | | |
| <400 c/mL at | | | | Υ | | | Υ |
| analysis timepoint | | | | | | | |
| (Week 24/48) | | | | | | | |
| outcome | | | | | | | |
| <400 c/mL by Visit | | | | Υ | Υ | | |
| Virologic Failure endpo | oints | | | | | | |
| Proportion of | Yx2 | | | Yx2 | Yx2 | | Yx2 |
| subjects without | | | | | | | |
| virologic or | | | | | | | |
| tolerability failure by | | | | | | | |
| analysis timepoint | | | | | | | |
| (Week 24/48) [4] | | | | | | | |
| Proportion of | Υ | | | Υ | Υ | | Υ |
| subjects without | | | | | | | |
| virologic or | | | | | | | |
| tolerability failure by | | | | | | | |
| analysis timepoint | | | | | | | |
| (Week 36/48) [5] | | | | | | | |
| Confirmed Virologic | | | | Yx2 <sup>[6]</sup> | | | Υ |
| Withdrawal Criteria | | | | | | | |
| by Visit | | | | | | | |
| Viral load for | | | | Υ | | | |
| Confirmed Virologic | | | | | | | |
| Withdrawal Criteria | | | | | | | |
| Time to viral | Υ | Υ | | Υ | | | |
| suppression (HIV-1 | | | | | | | |
| RNA <50 c/mL) | | | | | | | |
| Proportion of Subjects | | | | Yx2 <sup>[7]</sup> | | <u> </u> | |
| With Detectable Viral | | | | | | | |
| Load Below the Limit | | | | | | | |
| of Quantification at | | | | | | | |
| Week 24/48 | | | | | | | |
| Disease Progression | | | | Υ | | | Υ |
| HIV Conditions | | | | T | | | ľ |
| including Recurrences | | | | | | | |
| HIV Conditions | | | | Y | | | |
| excluding Recurrences | | | | | | | |
| HIV Disease | | | | Υ | | | |
| Progressions | | | | | | | |

| Endpoints | S | tats Analysi | S | Sum | mary | Individual | |
|---|---|---|---|---|---|---|---|
| • | Т | F | L | Т | F | F | L |
| <b>Exploratory Analysis</b> | | | | | | | |
| Proportion of<br>subjects with plasma<br>HIV-1 RNA <50 c/mL<br>at Week 48 using the<br>Snapshot algorithm –<br>Projected estimate | <b>Y</b> [8] | | | <b>Y</b> [2] | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. See full description in Section 11.13.
- 2. Study outcomes (i.e., response below 50 c/mL, virologic failure or reason for no data in the window) based on the snapshot algorithm will be summarised and listed.
- 3. Baseline demography (age, gender, race, country, CDC), HIV-1 subtype, Baseline CD4+ and Baseline viral load, background ART (ABC+3TC vs not ABC+3TC).
- 4. Outputs will be produced for TRD=F and ERD=F.
- 5. Outputs will be produced for TRD=F only using the MITT-E-36 & MITT-E-48 populations
- 6. The proportion of subjects with Confirmed Virologic Withdrawal Criteria will be summarised by visit, and also cumulatively by visit in terms of virologic non-response, virologic rebound and overall (see Appendix 6.)
- 7. Repeat by Baseline Viral Load
- 8. This summary will be produced for the week 24 study report
- 9. Based on the MITT-E-36 and MITT-E-48 populations

| Endpoint | Absolute | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual |
| | T F L | Т | F | F | Г | Т | F | L | Т | F | F | L |
| Immunologic | | | | | | | | | | | | |
| CD4+ cell counts | | | N | | | Υ | | | | Υ | Υ | |
| Plasma HIV-1 RNA Over Time | | | | | | | | | | | | |
| Observed | | | N | | Υ | Yx | | | | Υ | | |
| | | | | | | 4[1] | | | | | | |
| | | | | | | [2] | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - 1. Include the interpretation of whether the virus is detected or not ('Detected' or 'Not Detected') by the assay.
  - A Separate listing for Subjects with Virologic Failure (during randomised phase and separately during the
    continuation phase) or Last On-treatment VL >400 c/mL. Another listing of HIV-1 RNA and CD4 at baseline
    versus suspected and confirmed virologic failure.

## 8.1.2. Planned Efficacy Statistical Analyses

| Statistical Analyses |
|----------------------|
| Endpoint(s) |

## **Statistical Analyses**

 Proportion of subjects without virologic (ERDF) or virological and tolerability (TRDF) failure by analysis timepoint (Week 24/48)

## Model Specification/Analysis Methodology

- Estimated using the Kaplan-Meier nonparametric method based on the time to Confirmed Virologic Withdrawal Criteria (CVWC) or treatment related/efficacy related discontinuation (i.e., drug-related AE, protocol defined safety stopping criteria, or lack of efficacy)
- Subjects who have not met CVW criteria and are ongoing in the study, or who have discontinued for reasons other than those related to treatment, or switch from LPV/RTV to DTG, will be censored.
- The estimate of the standard error used to derive confidence intervals for the difference in proportions between treatment groups will be based on Greenwood's formula [Kalbfleisch, 1980].
- Quartiles of time to viral failure (including median) will be summarised by treatment group.
   Cls will estimated using the Brookmeyer Crowley Method.
- Cox proportional hazards model will also be used to estimate the hazard ratio (DTG vs. LPV/RTV) and 95% confidence interval.
- The estimated proportion of subjects without confirmed virologic withdrawal criteria and not discontinued due to treatment related/efficacy related reasons at the time of analysis (Week 24/48) will be presented by treatment group, along with estimated difference in proportions between treatment groups and its associated two-sided 95% CI.

0

#### **Model Results Presentation**

- Kaplan-Meier Plots for Time to Failure will be provided. The statistical analysis table will present:
  - Number and percentage of subjects with event or censored at week 24/36/48
  - Kaplan-Meier point estimate and 95% confidence intervals at week 24/36/48
  - Kaplan-Meier point estimate and 95% confidence interval of difference between groups at week 24/48

#### **Statistical Analyses**

### Endpoint(s)

The time to viral suppression (i.e. first viral load value <50 copies/mL)</li>

## Model Specification/Analysis Methodology

- Culmulative incidence curves estimated using the Kaplan-Meier method
  - Subjects who withdraw for any reason or switch from LPV/RTV to DTG without having suppressed prior to the analysis will be censored
  - Quartiles of time to viral suppression (including median) will be summarised by treatment group. Cls will estimated using the Brookmeyer Crowley Method.
  - Proportion of subjects with suppression at week 24/48 presented by treatment group.
- The generalised Wilcoxon procedure will be used to estimate a p-value for detecting a difference in cumulative incidence curves between treatment groups.
  - Note: In general, the logrank test tends to be sensitive to distributional differences which are most evident late in time. In comparison, the generalised Wilcoxon test tends to be more powerful in detecting differences early in time (when the proportional hazard assumption are not met).

## Statistical Analyses

- Cox proportional hazards model will also be used to estimate the hazard ratio (DTG vs. LPV/RTV) and 95% confidence interval.
- Kaplan-Meier Plots for time to viral suppression will be provided

#### **Model Results Presentation**

- Kaplan-Meier Plots for Time to Viral Suppression will be provided.
  - The statistical analysis table will present:
    - Number and percentage of subjects with event or censored at week 24/48
    - Quartiles of time to viral suppression (including median) and 95% confidence intervals
    - Proportion of subjects with suppression at week 24/48
- Hazard ratio for viral suppression (DTG vs. LPV/RTV) and 95% confidence interval

## **Exploratory Statistical Analyses**

The proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm will be estimated using the data collected at time of the Week 24 interim analysis. The purpose of this exploratory analysis is to explore the application of multiple imputation in predicting Week 48 response which may be useful for IDMC and futility analyses purposes in future. Subject data within the database at time of the Week 24 analysis should be considered into 3 groups:

- [1] Subjects completed the study at Week 52
- [2] Subjects withdrawn from the study prior to the Week 24 data cut-off
- [3] Subjects ongoing within the study at time of the Week 24 data cut-off
- Data for subjects in group 3 will be imputed using the methodology proposed below using all subject data from groups 1-3.

#### Endpoint(s)

 Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm – Projected Estimate

#### Covariates

Baseline Plasma HIV-1 RNA (≤ vs. >100,000 c/mL)
 Baseline Number of Fully Active NRTIs in the Background Regimen (2 vs.<2)</li>

#### Model Specification/Analysis Methodology

- Select Log(HIV-1 RNA) samples
  - Using Markov Chain Monte Carlo methods, simulate 100 datasets replacing BLQ with values with those from a Log(Uniform(0, BLQ) distribution. The BLQ value used for this step should be slightly below the actual BLQ cut-off so that response is correctly attributed when applying the snapshot algorithm later.
  - The statistical model used for the MI data generation will be the Markov Chain Monte Carlo (MCMC) method with for the data (covariates, randomised treatment group, and Log HIV-1 RNA at Baseline, Week 4, Week 8, Week 16, Week 24, Week 36, and Week 48) to produce a monotone pattern first, and then the imputation will continue using the Regression with Predictive Mean Matching (REGPMM) method for the monotone pattern with the same set of covariates.
    - A seed of 200304 will be used in the SAS program.
    - One imputation is required for each of the monotone and mean matching steps

#### Statistical Analyses

- For subjects that discontinued from the study prior to Week 24 data cut off, replace the imputed data with their original data. Data related to these subjects will be used only for the imputation of data for those that were ongoing at time of the Week 24 data cut off.
- Week 52 HIV-1 RNA data for subjects that completed the study will not be included in the multiple imputation. Instead, the Week 52 data will be merged back onto the imputed datasets prior to the application of the snapshot algorithm.
- Using Snapshot Algorithm, derive virologic response or failure at Week 48 using snapshot algorithm, as per Section 11.13, for each imputed dataset.
- For each imputed dataset, the endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for Baseline plasma HIV-1 RNA ( ≤ vs. >100,000 c/mL) and number of fully active background NRTIs in the background regimen (<2 vs. 2) at Baseline. This will be the same model as used for the primary endpoint.
- Wilson-Hilferty transformation will be applied to normalise the CMH statistic
- PROC MIANALYZE in SAS will be used to combine the 1,000 estimated proportion of subjects with plasma HIV-1 RNA <50 c/mL and difference in proportions to produce one estimate with 95% CI and associated p-value for the adjusted difference between each treatment group at Week 48

#### **Model Results Presentation**

Adjusted CMH estimate of the difference in the proportion of responders between each treatment group (DTG – LPV/RTV) and corresponding 95% confidence interval

## 8.2. Safety Analyses

## 8.2.1. Overview of Planned Analyses

The safety analyses will be based on the Safety population, presented by treatment group with a total column and included in all reporting efforts unless otherwise specified.

The observed case (OC) dataset will be used, which contains the data that is available at a particular timepoint, with no imputation for missing values, unless otherwise stated. All displays are for the randomised phase only, unless specified otherwise. This means that the analysis other than "by-visit" summaries will not be windowed at Week 24 (AEs, maximum post-baseline toxicities). In other words, all data collected up to the point of DBF will be included in summary statistics, which could be past week 24 for subjects enrolled early in the study. However, at the Week 48 analysis, summary statistics will include data up to Week 52 for both arms.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 18: List of Data Displays.

For the purposes of summarising AE data, unless stated otherwise, the summaries will include post-baseline data from the Randomised Phase of the study. AEs are considered post-baseline if the onset date is on or after IP start date and before entering continuation phase. AE onset during the Continuation Phase will not be included in the Randomised Phase summaries unless it is specified in the title ie Randomised and Continuation Phase.

Following the IDMC recommendation to switch subjects on the LPV/RTV treatment arm to a regimen with DTG as the third drug, in the Week 48 analysis, the summaries of AE and laboratory data will only include AEs/laboratory data prior to switch, and AEs/labs post switch will just be listed

An issue was identified with the creatinine testing at the central laboratory. Sensitivity analyses will be conducted excluding any suspect creatinine samples from laboratory summaries including creatinine see Appendix 14.

Table 7 Overview of Planned Safety Analyses

| Endpoint | | | | Abso | olute | | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|--|
| | Stats<br>Analysis | | | Summary | | | vidual | Stats<br>Analysis | | | Summary | | Individual | | |
| | T | F | L | Т | F | F | L | T | F | L | Т | F | F | L | |
| Exposure Extent of Exposure | | Ι | I | 1010-34 | 1 | I | Υ[10] | | I | | | | 1 | 1 | |
| Extent of Exposure Adverse Events [19] | | | | Yx2 <sup>[9]</sup> | | | Y[10] | | | | | | | <u> </u> | |
| | Υ | | | | | | | | | | | | | | |
| Grade 2 or greater<br>Drug-Related<br>Diarrhoea | | | | | | | | | | | | | | | |
| All AEs by SOC [1] | | | | Y | | | Y (x3) | | | | | | | | |
| All AEs by SOC by Toxicity Grade [12] | | | | Y | | | | | | | | | | | |
| Common AEs by frequency <sup>[13]</sup> | | | | Y | Y<br>[15] | | | | | | | | | | |
| Common grade 2-4<br>AEs by frequency [13] | | | | Y | | | | | | | | | | | |
| All Grade 2-4 AEs by SOC | | | | Y | | | | | | | | | | | |
| All Drug-Related AEs<br>by SOC and toxicities<br>[12] | | | | Y | | | | | | | | | | | |
| All Drug-Related AEs by SOC <sup>[12</sup> ] | | | | Y | | | | | | | | | | | |
| Common Grade 2-4<br>Drug-Related AEs by<br>frequency [13] | | | | Y | | | | | | | | | | | |
| All Grade 2-4 Drug-<br>Related AEs by SOC | | | | Y | | | | | | | | | | | |
| Serious AEs | | | | Y[10] | | | Y | | | | | | | | |
| Reason for<br>Considering as a<br>Serious Adverse<br>Event (FDA) | | | | | | | Y | | | | | | | | |
| Drug-Related Serious<br>AEs | | | | Y | | | | | | | | | | | |
| Fatal AEs | | | | | | | Υ | | | | | | | | |
| Non-Fatal Serious<br>AEs | | | | Y | | | Υ | | | | | | | | |
| AEs leading to withdrawal | | | | Y | | | Y | | | | | | | | |
| Common non-<br>serious AEs | | | | Y | | | | | | | | | | | |
| Endpoint | | | | Abso | lute | | | | ( | Char | nge from | Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Stats | | Sumn | nary | Indi | vidual | | tats<br>alysi | | Summ | | | ridual |
| | T | F | L | Т | F | F | L | T | F | L | Т | F | F | L |
| (FDAAA) | | | | | | | | | | | | | | |
| Number of<br>occurrences on Non-<br>serious AEs by SOC<br>(EudraCT) | | | | Y | | | | | | | | | | |
| Number of<br>occurrences of SAEs,<br>Drug-related SAEs,<br>Fatal AEs, and Drug-<br>related SAEs<br>(EudraCT) | | | | Y | | | | | | | | | | |
| Non-serious AEs and SAE of Mexican Subjects <sup>[8]</sup> | | | | | | | Y | | | | | | | |
| SAEs of non-Mexican subjects (include drug-related as a column) [8] | | | | | | | Y | | | | | | | |
| CV events | | | | | | | Υ | | | | | | | |
| PSRAE | | | | | | | Υ | | | | | | | |
| Summary of<br>Cumulative Adverse<br>Events | | | | Y | | | | | | | | | | |
| Laboratory Values | | | | | | | ı | | | | I | ı | | |
| Fasting LDL<br>Cholesterol | | | | | | | | Yx3 | Υ | | | | | |
| Fasting TC/HDL ratio | | | | | | | | Yx3 | Υ | | | | | |
| Fasting LDL Cholesterol Treatment Emergent Abnormalities of Grade 2 or Greater <sup>[7]</sup> | | | | | | | | <b>Y</b> [7] | | | | | | |
| Clinical Chemistry | | | | | | | <b>Y</b> [3] | | | | Yx3 <sup>[2,3]</sup> | | | |
| Hematology | | | | | | | Yx2 <sup>[4]</sup> | | | | Yx2 <sup>[2]</sup> | | | |
| Urinalysis (Dipstick) | | | | | | | Y | | | | | | | |
| Liver chemistries <sup>[7][6]</sup> | | | | | | | | | | | | Y | Υ | |
| NCEP shifts in lipids [21][7] | | | | | | | | | | | Yx4 | Yx4 | | |
| ECGs <sup>[5]</sup> | | | | | | | | | | | | | | |

| Endpoint | | | | Abso | lute | | | | ( | Chan | ge from | Basel | Baseline | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 5 | Stats | ; | Sumn | nary | Indi | vidual | Stats | | | Summary | | Indiv | Individual |
| | Ar | alys | is | _ | | <u>.</u> | | Analysis | | | | | | |
| | Т | F | L | T | F | F | L | Т | F | L | T | F | F | L |
| ECG Findings | | | | | | | Y | | | | | | | |
| Vital Signs | • | • | | | | • | | • | | | | | • | • |
| Vitals Values | | | | | | | Υ | | | | Υ | | | |
| Other | | | | | | • | | • | | | | | | • |
| Abacavir HSR | | | | | | | Υ [16] | | | | | | | |
| Liver Assessment | | | | | | | Υ [17] | | | | | | | |
| Hepatobiliary<br>Abnormality criteria –<br>post baseline<br>emergent | | | | Y | | | Y | | | | | | | |
| Columbia suicidality | | | | Y | | | Υ [18] | | | | | | | |
| Subjects who became<br>Pregnant | | | | | | | Y | | | | | | | |
| Patient profiles | | | | | | | Yx2<br>[20] | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Listings will include subject's numbers for individual AE's & AE system organ classes, preferred terms and verbatim text.
- Chemistry & haematology summaries will include both changes from baseline & maximum post baseline emergent toxicities. Change from Baseline chemistry summaries will be repeated for Lipids and Glucose in Conventional Units.
- 3. Clinical chemistry summaries will be re-run excluding subjects with suspect creatinine samples.
- 4. Listing of Chemistry, haematology data for subjects with abnormalities of PCI will be listed.
- 5. Only measured as part of CV assessment
- 6. Scatter Plot of Maximum vs. Baseline for ALT, Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin
- 7. Maximum Post-baseline
- 8. Includes Continuation Phase and is only for the End of Study reporting effort.
- 9. One for Randomisation Phase and one including the Continuation Phase.
- 10. Repeated for Mexican subjects. Outputs for Mexican subjects include Continuation Phase and are only needed for the end of study reporting effort.
- 11. One listing of all AEs including verbatim text and preferred term, one showing the relationship between verbatim text, preferred term and SOC and another giving subject numbers for individual all treatment emergent AEs.
- 12. For AEs reported more than once by a subject, the most severe intensity will be included.
- 13. Common AEs are those with >5% incidence in either treatment group summarised by frequency.
- 14. Common AE by frequency graph description
- 15. Plots of incidence rates and relative risk for DTG vs. LPV/RTV.
- 16. Separate listings for exposure to abacavir, history of drug allergies, family conditions, skin rash, symptoms, vital signs, individual symptoms and diagnostic category assignment.
- 17. Separate listings for time of event from trt, RUCAM score, biopsy, imaging, past/ current conditions & FU
- 18. Listing but classed as a Table. Includes Baseline and lists all visits for a subject who reports any ideation or behaviour at any visit..
- 19. Adverse events will be coded using the MedDRA coding dictionary to give a preferred term and a system organ class. Summaries include only Post-baseline AEs with onset date up to cut-off date for reporting effort, listings

- include all AEs including those with onset pre- or post-treatment.
- 20. Patient profiles for subjects meeting protocol defined liver stopping criteria and for patients with virological failures. Patient profiles can also be provided for any other subjects, as necessary for medical review.
- 21. One output will be created for each lipid parameter. Bar chart for LDL, HDL, TC, Trig and HDL/TC ratio

## 8.2.2. Planned Safety Statistical Analyses

## Statistical Analyses

## **Endpoints**

- Change from Baseline in fasting LDL cholesterol at Weeks 24 and 48
- Change from Baseline in fasting TC/HDL ratio at Weeks 24 and 48

## **Lipids Last Observation Carried Forward (LOCF) Dataset**

• See Appendix 7

## **Covariates**

- Baseline Plasma HIV-1 RNA (≤ vs. >100,000 c/mL)
- Baseline Number of Fully Active NRTIs in the Background Regimen (2 vs.<2)</li>
  - Age (<35, 35-<50, ≥50)

## **Data Handling**

- If a subject is on lipid-lowering therapy from Baseline, they will be excluded from the analysis.
- If a subject initiates lipid-lowering therapy during the study, all visits after that date will be set to missing.
- All other data remains as is (observed or missing).
- A multiple imputation technique will be used to deal with the missing data.

## **Model Specification**

- Multiple imputations will be drawn from a multivariate normal model for the data (Fasted LDL, cholesterol and fasted TC/HDL measurements at Baseline, Week 16, Week 24 and Week 48 (including covariates) with a Markov Chain Monte Carlo (MCMC) approach used to estimate posterior distributions. A seed of 200304 will be used in the SAS program. Where a subject has a monotone or non-monotone pattern of missingness, all of their missing observations can be imputed under this approach. The absolute value will be imputed before the change value is calculatedImputations will be drawn separately for subsets of subjects according to their treatment group, i.e., based on means and variance-covariances from the same treatment group (Missing At Random (MAR) approach) conditioning on observed covariates listed above. This will be known as the MAR method.
- The imputations will be carried out 1,000 times. An ANOVA will be performed on each datasets produced adjusting for treatment, baseline value and the categorical covariates, regardless of their significance. PROC MIANALYZE in SAS will be used to combine the 1,000 estimated means and difference to produce one estimated mean with 95% CI and associated p-value for the adjusted mean difference between each treatment group at Week 24/48.
- Interactions between treatment and each of the covariates will not be assessed.

## **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

## **Model Results Presentation**

 Adjusted means and corresponding standard error of means (SEs) will be presented for each treatment, together with estimated treatment difference (DTG – LPV/RTV) and corresponding

## **Statistical Analyses**

95% confidence interval and p-value.

• Plots of LS means and 95% confidence intervals from the model will be generated for each treatment by time.

## Sensitivity Analyses

Sensitivity analyses will be performed as follows:

- using the standard Observed Case (OC) dataset, with no adjustment or imputation for withdrawing, initiating lipid-lowering agents or other missing data. An analysis of covariance (ANCOVA) model will be used with covariates (listed above), and baseline value as a covariate.
- using the Lipid LOCF dataset, but also carrying forward the last observation to any missing
  visits, an ANCOVA model will be used with treatment, covariates (listed above), and baseline
  value as a covariate.

## **Statistical Analyses**

## **Endpoints**

- The incidence of maximum post-Baseline emergent Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Weeks 24 and 48
- The incidence of maximum post-Baseline emergent Grade 2 or greater drug-related diarrhoea by Weeks 24 and 48

## **Dataset**

• The observed case (OC) dataset uses only the data that is available at a particular timepoint, with no imputation for missing values.

# Model Specification/Analysis Methodology

 Endpoints will be statistically analysed for the comparison between DTG and LPV/RTV by Fisher's exact test using the Safety Population

## **Model Results Presentation**

 Incidence for each treatment group and a p-value for the difference in incidence between treatment groups.

# 9. OTHER STATISTICAL ANALYSES

# 9.1. Health Outcomes Analyses

# 9.1.1. Overview of Planned Analyses

The Health Outcomes (HO) analyses will be based on the Intent-to-treat Exposed population, presented by treatment group with a total column and included in all reporting efforts unless otherwise specified.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 18: List of Data Displays.

Following the IDMC recommendation to switch subjects on the LPV/RTV treatment arm to a regimen with DTG as the third drug, the Week 48 summaries and analyses of HO data will only include HO data prior to switch, and HO post switch will just be listed.

Table 8 Overview of Planned Health Outcome Analyses

| Endpoint | | | F | bsolu | ite | | | | Ch | ange | from | Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | | idual | | s Anal | ysis | Sum | mary | | ridual |
| | Т | F | L | Τ | F | F | L | T | F | L | T | F | F | L |
| HIVTSQs | | | | • | | | | | 1 | 1 | • | • | • | |
| Individual Item | | | | Υ | | | Υ | | | | Υ | | | |
| Scores | | | | | | | | | | | | | | |
| Treatment | | | | Υ | | | Υ | Yx2 | | | Υ | | | |
| Satisfaction Score | | | | | | | | | | | | | | |
| HIVTSQc | | | | | | • | • | , | | | , | | , | |
| Individual Item | <b>Y</b> [1] | | | Υ | | | Υ | | | | | | | |
| Scores (Change) | | | | | | | | | | | | | | |
| Treatment | Υ | | | Υ | | | Υ | | | | | | | |
| Satisfaction | | | | | | | | | | | | | | |
| (Change) | | | | | | | | | | | | | | • |
| MMAS-8 | | | | | | | | | | | | | | |
| Total Score | | | | Υ | | | Υ | | | | | | | |
| Adherence Level | Υ | | | Υ | | | Υ | | | | | | | |
| Gastrointestinal Sym | ptom | Rati | ng S | cale ( | GSRS | 3) | | | | | | | | |
| Individual Item | | | | Υ | | | Υ | | | | | | | |
| Scores | | | | | | | | | | | | | | |
| Diarrhoea Syndrome | | | | Υ | | | Υ | Υ | | | Υ | | | |
| Score | | | | | | | | | | | | | | |
| Indigestion | | | | Υ | | | Υ | Υ | | | Υ | | | |
| Syndrome Score | | | | | | | | | | | | | | |
| Constipation Score | | | | Υ | | | Υ | Υ | | | Υ | | | |
| Abdominal Score | | | | Υ | | | Υ | Υ | | | Υ | | | |
| Reflux Score | | | | Υ | | | Υ | Υ | | | Υ | | | |

| Endpoint | Absolute | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | is Summary Individual | | | idual | Stats | Anal | ysis | Summary | | Individual | |
| | Т | F | L | Τ | F | F | L | Т | F | L | Т | F | F | L |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- HIVTSQ questionnaire included in Section 11.6.6
   Individual = Represents FL related to any displays of individual subject observed raw data

## 9.1.2. Planned Health Outcomes Statistical Analyses

## Statistical Analyses

#### **HIVTSQs**

- Change from Baseline at Week 4, Week 24, and Week 48:
  - Treatment Satisfaction Score

## **Model Specification**

- The MMRM will adjust for visit, Baseline Plasma HIV-1 RNA (≤ vs. >100,000 c/mL) and Baseline Number of Fully Active NRTIs in the Background Regimen (2 vs.<2).
- The model will make no further assumptions about the correlations between a subject's score (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between
  visits (ie. a treatment\*visit interaction will be included in the model), and separates estimates
  and 95% confidence intervals will be produced at each visit. The model will also assume that
  the effect of baseline score can vary between visits (ie. baseline score\*visit interactions will be
  included in the model).
- Interactions between treatment and each of the covariates will not be assessed unless the exploratory subgroup analyses described in Section 7.1.2 on the primary endpoint highlights significant interactions. In this situation, the interaction(s) of interest will be assessed and, if necessary, results will be reported in the clinical study report. Interactions between treatment and the baseline score will be investigated but not included in the model. If interactions are found to be significant, results might have to be presented separately by subgroup.

## **Dataset**

• The observed case (OC) dataset uses only the data that is available at a particular timepoint, with no imputation for missing values in addition to the ones described in Section 11.6.7.

## **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

## **Model Results Presentation**

- The summaries will include the adjusted mean change from baseline and confidence interval for each treatment group across visits.
- The interaction between treatment and the baseline score will be included in a footnote.

## **Statistical Analyses**

## **HIVTSQc**

Treatment Satisfaction Score (Change) at Week 48

## Model Specification

# Statistical Analyses

•

 An analysis of covariance (ANCOVA) model will be used with covariates: treatment, Baseline Plasma HIV-1 RNA (≤ vs. >100,000 c/mL) and Baseline Number of Fully Active NRTIs in the Background Regimen (2 vs.<2).</li>

## Dataset

• The observed case (OC) dataset uses only the data that is available at a particular timepoint, with no imputation for missing values in addition to the ones described in Section 11.6.7.

## **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 Adjusted means and corresponding standard error of means (SEs) will be presented for each treatment, together with estimated treatment difference (DTG – LPV/RTV) and corresponding 95% confidence interval and p-value.

## **Statistical Analyses**

#### MMAS-8

Adherence level

# Model Specification/Analysis Methodology

• Endpoints will be statistically analyzed for the comparison between DTG and LPV/RTV by Fisher's exact test using the ITT(e) Population

#### **Dataset**

• The observed case (OC) dataset uses only the data that is available at a particular timepoint, with no imputation for missing values in addition to the ones described in Section 11.6.7.

## **Model Results Presentation**

• Incidence for each treatment group and a p-value for the difference in incidence between treatment groups.

## Statistical Analyses

## Gastrointestinal Symptom Rating Scale (GSRS)

- Change from Baseline at Week 4, Week 24, and Week 48:
  - Diarrhoea Syndrome Score
  - Indigestion Syndrome Score
  - Constipation Score
  - Abdominal Score
  - Reflux Score

## **Model Specification**

•

 A Wilcoxon rank sum test will be used to compare the change in gastrointestinal symptom rating score sub-items for subjects treated with DTG and LPV/RTV at each visit

| Statistical Analyses |
|---|
| Dataset |
| • The observed case (OC) dataset uses only the data that is available at a particular timepoint, with no imputation for missing values in addition to the ones described in Section 11.6.7. |
| Model Checking & Diagnostics |
| Model Results Presentation |
| • |

# 9.2. Virology Analyses

## 9.2.1. **Overview of Planned Analyses**

The virology analyses will be based on the Viral Genotypic or Viral Phenotypic population, unless otherwise specified.

Phenotype data may not be available for all subjects in China at the time of the Week 24 analyses. The China subjects may also have genotype data from Q2 and/or Monogram. In the event that subjects have both Q2 and Monogram data at a timepoint, the Monogram data will be used. Footnotes will be included in summaries indicating which subjects have Q2 data only or Q2 and Monogram.

Table 9 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 15 List of Data Displays.

Table 9 Overview of Planned Virology Analyses

| Endpoint | S | tats Analysi | S | Sum | mary | Indiv | ridual |
|---|---|---|---|---|---|---|---|
| • | Τ | F | L | Т | F | F | L |
| Incidence of treatment | Incidence of treatment-emergent genotypic and phenotypic resistance to DTG, LPV/RTV and other | | | | | | |
| on-study ART in subject | cts meeting | confirmed | virologic w | ithdrawal c | riteria | | |
| Genotype | | | | | | | |
| Summary of | | | | Υ | | | |
| Genotypes Available | | | | | | | |
| Treatment Emergent | | | | Y | | | |
| Major Mutations of | | | | | | | |
| NRTI, NNRTI and PI | | | | | | | |
| Classes | | | | | | | |
| Pre-specified | | | | Υ | | | |
| Treatment Emergent | | | | | | | |
| IN Substitutions at | | | | | | | |
| Time of Confirmed | | | | | | | |
| Virologic Withdrawal | | | | | | | |

| Endpoint | S | tats Analysis | 3 | Sum | mary | Indiv | ridual |
|---|---|---|---|---|---|---|---|
| | T | F | L | T | F | F | L |
| Changes in Genotypic<br>Susceptibility (GSS)<br>to Background ART<br>Therapy at Time of<br>Confirmed Virologic<br>Withdrawal | | | | Y | | | |
| All Genotypic Data | | | | | | | Y |
| Phenotype | | | | | | | |
| Summary of Phenotypes Available | | | | Y | | | |
| Fold Change to DTG<br>and LPV/RTV at<br>Baseline and Time of<br>Confirmed Virologic<br>Withdrawal | | | | Y | | | |
| Changes in Phenotypic Resistance (PSS <sub>f</sub> ) to Background ART Regimen at Time of Confirmed Virologic Withdrawal | | | | Y | | | |
| All Phenotypic Data | | | | | | | Yx2 <sup>[2]</sup> |
| Net Assessment for Ov | erall Susce | ptibility Sco | ore | | | | |
| Overall Susceptibility Score (OSS) | | | | <b>Y</b> [3] | | | |
| Other | | | | | | | |
| Key Virologic Data | | | | | | | Yx4 <sup>[1]</sup> |
| Virology Data at<br>Confirmed Virologic<br>Withdrawal | | | | Y | | | |

## NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. A Separate listing for Subjects with Virologic Failure (during randomisation phase and separately during the continuation phase) or Last On-treatment VL >400 c/mL.
- 2. Include a separate listing for screening results from Quest.
- 3. Produce for CVW resistance populations.
- 4. This is a listing of subject data to be included as a Table.

## 10. REFERENCES

Fleiss J.L. Statistical Methods for Rates and Proportions. 2<sup>nd</sup> ed. New York:John Wiley; 1981.

GlaxoSmithKline Document No.: 2013N172672\_01A Phase 3b, randomised, open-label study of the antiviral activity and safety of dolutegravir compared to lopinavir/ritonavir both administered with dual nucleoside reverse transcriptase inhibitor therapy in HIV-1 infected adult subjects with treatment failure on first line therapy Effective 30-Apr-14

Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). *JAMA*. 2001;285 (19):2486-2497.

HIVTSQ user guidelines

Kalbfleisch J.D., Prentice R.L. The Statistical Analysis of Failure Time Data. 1<sup>st</sup> ed. New York: John Wiley & Sons; 1980.

Liu TF, Shafer RW. Web Resources for HIV type 1 Genotypic-Resistance Test Interpretation. *Clin Infect Dis.* 2006;42 (11):1608-1618.

Lui K.J., Kelly C. A Revisit on Tests for Homogeneity of the Risk Difference, *Biometrics*, 2000;56:309-315.

Ralph B. D'Agostino, Ramachandran S. Vasan, Michael J. Pencina, Philip A. Wolf, Mark Cobain, Joseph M. Massaro, William B. Kannel. 2008. General Cardiovascular Risk Profile for Use in Primary Care (The Framingham Heart Study). Circulation 2008; 117: 743-753.

Sato T. On the variance estimator for the Mantel-Haenszel risk difference. *Biometrics*. 1989;42:311-323.

Wensing AM, Calvez V, Günthard HF et al. 2014 Update of Drug Resistance Mutations in HIV-1. *Topics in Antiviral Medicine* 2014; 22(3): 642-650.

# 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | Analysis Populations |
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 11.2 | Appendix 2: Time and Events |
| Section 11.3 | Appendix 3: Assessment Windows |
| Section 11.4 | Appendix 4: Treatment States & Phases |
| Section 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | • Efficacy |
| | Virology |
| Section 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| 0 11 11 0 | Handling of Missing Data |
| Section 11.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 11.9 | Appendix 9: Multicentre Studies |
| Section 11.10 | Appendix 10: Examination of Covariates and Subgroups |
| Section 11.11 | Appendix 11: Handling of Multiple Comparisons & Multiplicity |
| Section 11.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | |
| Section 11.13 | Appendix 13: Snapshot |
| Section 11.14 | Appendix 14: Q2 Creatinine Assay Accuracy Issue |
| Section 11.15 | Appendix 15 Abbreviations & Trade Marks |
| Section 11.16 | Appendix 16: Example SAS code for Additional Estimand 2 |
| Section 11.17 | Appendix 17: End of Study Analysis |
| Section 11.18 | Appendix 18 : List of Data Displays |

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 11.1.1. Exclusions from Per Protocol Population

Protocol deviations leading to exclusion from PP population are those deviations which

- may directly impact the efficacy endpoint of HIV-1 RNA; or
- lead to permanent discontinuation of IP/withdrawal and hence indirectly impact the efficacy endpoint by causing data to be missing.

The following criteria define the protocol deviations which, if they occur prior to an analysis timepoint of interest, will lead to exclusion of a subject from the Per-Protocol population for that analysis. Potential protocol deviations leading to exclusion from PP population will be reviewed by the study team to confirm that they meet these criteria. This review will occur before the clinical database has been frozen for analysis.

A subject meeting any of the following criteria prior to the timepoint of interest (eg week 24 or 48) will be excluded from the Per Protocol population for the week 24 interim or week 48 respectively:

| <b>Exclusion Description</b> |
|---|
| Subject deviates from any inclusion or exclusion criteria, as recorded in the eCRF |
| Prohibited medications. |
| There are several sub-categories for prohibited medication use: |
| <ul> <li>a) Subject receiving prohibited non-ART medications (See<br/>protocol) or receiving non-ART medication that would<br/>potentially impact exposure or response to therapy.<br/>Duration of &gt;2 consecutive weeks will be considered<br/>prohibited.</li> </ul> |
| <ul> <li>HIV immunotherapeutic vaccines</li> <li>Other experimental agents</li> <li>Antiretroviral drugs not otherwise specified in the protocol</li> <li>Cytotoxic chemotherapy</li> <li>Radiation therapy</li> <li>Immunomodulators: <ul> <li>Calcineurin Inhibitors</li> <li>Cyclosporine A, Pimecrolimus, Tacrolimus</li> <li>Fluorouracil (including topical)</li> <li>Interferon (rectal and transdermal routes are permitted)</li> </ul> </li> </ul> |

| Number | <b>Exclusion Description</b> |
|---|---|
| | <ul> <li>Everolimus, Sirolimus</li> <li>Methotrexate</li> <li>Purine Analogues <ul> <li>Azathioprine, 6-Mercaptopurine</li> </ul> </li> <li>Targeted Immune Modulators (Biological Response Modifiers) <ul> <li>Abatacept, Adalimumab, Alefacept, Anakinra, Certolizumab, Efalizumab, Etanercept, Golimumab, Infliximab, Natalizumab, Rituximab, Tocilizumab, Ustekinumab</li> </ul> </li> <li>HCV therapy sofosbuvir (Sovaldi, Virunon),ledipasvir/sofosbuvir (Harvoni), paritaprevir/ritonavir/ombitasvir + dasabuvir (Viekira Pak),paritaprevir/ritonavir/ombitasvir (Viekirax), dasabuvir (Exviera), simeprevir (Olysio), telaprevir (Incivek, Incivo), boceprevir (Victrelis), peginterferon alfa (e.g. Pegasys), interferon alfa (e.g. Intron A,</li> </ul> |
| | <ul> <li>Roferon-A), ribavirin (Copegus, Rebetol)</li> <li>b) Chronic use (&gt;30 days) of systemic glucocorticoids</li> <li>oral &amp; iv routes are not permitted</li> <li>topical &amp; nasal routes are permitted</li> <li>c) Treatment dependent prohibited medications. Any duration is considered prohibited</li> </ul> |
| | For subjects randomised to DTG: |
| | <ul> <li>For subjects randomised to LPV/RTV:</li> <li>Alfuzosin</li> <li>Amiodarone</li> <li>Antihistamines (astemizole, terfenadine)</li> <li>Cisapride</li> <li>Ergot alkaloids (dihydroergotamine, ergonovine, ergotamine, methylergonovine)</li> <li>Fusidic acid (in dermatological infections)</li> <li>HMG Co-A reductase inhibitors (specifically lovastatin, simvastatin)</li> </ul> |

| Number | Exclusion Description |
|---|---|
| | <ul> <li>Pimozide</li> <li>Rifampicin</li> <li>Sildenafil (when used for the treatment of pulmonary arterial hypertension)</li> <li>Vardenafil</li> <li>Avanafil</li> <li>Midazolam (oral)</li> <li>Triazolam</li> <li>St John's wort (Hypericum perforatum)</li> </ul> |
| | As these deviations are treatment dependent it will not be possible to identify if they are deviations until treatment details are known post unblinding. d) Prohibited ART Medication Use Receiving ART medication other than that prescribed/allowed by the |
| | study for any duration |
| 03 | Non-permitted switch of background ART, specifically: On-treatment changes of background ART post the Week 4 visit window that • Are made for reasons other than toxicity or tolerability management, or • Introduce new agents which are not within class substitutions, or Result in a background regimen that consists of more than 2 NRTIs (or 3 NRTIs in the case of subjects receiving 3TC/FTC for treatment of hepatitis B. If a subject does not take an NRTI or a fully active NRTI this will be considered a protocol deviation and lead to exclusion from the PP Population. This will be considered as a non-permitted switch of background ART. |
| 04 | Subject took/received incorrect IP, i.e., other than the one to which they were randomised for greater than 10% of the total time On-treatment. It will not be possible to identify whether subjects received a different treatment to the one they were randomised to until post unblinding. |
| 05 | Interruption of IP for greater than 10% of the total time On-treatment, for reasons other than treatment-related adverse events/laboratory abnormalities, based on eCRF IP exposure forms. This is mentioned in the PDMP but it is not listed as a PD category. |
| 06 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF). This is stated in the PDMP but it is not listed as a PD category as the PD will be classified under one of the other PD categories. |

# 11.2. Appendix 2: Time & Events

# 11.2.1. **Protocol Defined Time & Events**

| Procedures | | | | | Ra | ndomise | d Phase | | | | tinuation | Withdrawal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening* | Baseline<br>(Day 1) | | | Day 1 to | Week 48 | 3 | | 4-week<br>Treatment<br>Extension | F | haseb | | upe |
| | | | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | Week<br>36 | Week<br>48 | Week 52 | Week<br>60 | Every 12<br>weeks<br>thereafter | | |
| Clinical and Other | r Assessmen | ta | | | | | | | | | | | |
| Written informed<br>consent | X | | | | | | | | | | | | |
| Indusion/Exclusion<br>criterias | X | | | | | | | | | | | | |
| Subject<br>demography | X | | | | | | | | | | | | |
| Medical history* | X | | | | | | | | | | | | |
| Prior ART history | X | | | | | | | | | | | | |
| CDC HIV-1<br>dessification | X | X | | | | | | | | | | | |
| Limited physical<br>examination/ | X | X | X | Х | Х | X | Х | Х | X | X | X | X | X |
| Body weight and<br>height | | X | | | | | | | | | | | |
| Current medical<br>conditions | | X | | | | | | | | | | | |
| CV risk<br>assessment# | | X | | | | | | | | | | | |
| Concomitant<br>medication | X | X | X | X | Х | Х | X | X | Х | X | X | X | X |

| Procedures | | | Randomised Phase | | | | | | | Continuation | | Withdrawal | Follow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening* B | | · [ | | | | | 4-week Phaseb<br>Treatment<br>Extension | | up <sup>c</sup> | | | |
| | | | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | Week<br>36 | Week<br>48 | Week 52 | Week<br>60 | Every 12<br>weeks<br>thereafter | | |
| HIV associated<br>conditions | | | Х | X | Х | Х | Х | Х | X | Х | X | х | |
| Columbia<br>Suicidality Seventy<br>Rating Scale | | χ'n | X | X | X | X | X | X | X | X | X | X | |
| Adverse events | | X | X | X | X | X | Х | X | X | X | X | Х | X |
| SAE <sub>5</sub> | χı | X | X | X | X | X | Х | X | Х | X | X | Х | X |
| GSRS | | X | X | | | X | | X | | | | X | |
| HIVT9Qs | | X | X | | | X | | X | | | | X | |
| HIVTSQc | | | | | | | | Х | | | | X | |
| MMAS-8 | | X | X | | | X | | X | | | | X | |
| Laboratory Asses | sments | | | | | | | | | | | | |
| Ouantitative<br>plasma HIV-1 RNA<br>PCR | X | X | X | X | Х | X | X | X | х | X | X | X | |
| Lymphocyte subset | X | X | X | X | Х | X | Х | X | Х | X | X | X | |
| Plasma for HIV<br>genotyping | х | | | | | | | | | | | | |
| Plasma for<br>storage <sup>k</sup> | X | X | Х | X | X | Х | X | X | X | X | X | Х | |
| HLA-B* 5701<br>testing | X | | | | | | | | | | | | |
| Clinical chemistry | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Haematology | X | X | X | X | Х | X | Х | Х | X | X | X | Х | X |
| PT/INR | X | | | | | | | | | | | | |
| Fasting lipids and<br>glucose <sup>n</sup> | | Х | | | X | X | | X | | | | | |
| Pregnancy tests | S | U | S | S | S | S | S | S | S | S | S | S | S |

| Procedures | | | | | Ra | ndomise | d Phase | | | | tinuation | Withdrawal | Follow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening* | Baseline<br>(Day 1) | | Day 1 to Week 48 4-week<br>Treatme<br>Extensio | | | | | | | | | mbe |
| | | | Week<br>4 | Week<br>8 | Week<br>16 | Week<br>24 | Week<br>36 | Week<br>48 | Week 52 | Week<br>60 | Every 12<br>weeks<br>thereafter | | |
| HBsAg, anti-HBc<br>and anti-HCV <sup>a</sup> | X | | | | | | | | | | | | |
| HBV DNAP | | X | | | | | | | | | | | |
| Pharmacogenetic<br>samples | | X | | | | | | | | | | | |
| PBMCs <sup>r</sup> | | X | | | | | | | | | | | |
| Investigational pr | oduct | | | | | | | | | | | | |
| MRS | X | X | X | Х | X | Х | X | X | X | X | X | X | X |
| Dispense IP | | X | X | X | X | X | X | X | Χs | X | X | | |
| IP accountability<br>(pill counts) | | | Х | Х | X | Х | Х | Х | Х | Х | X | Х | |

- The 28-day Screening period may be extended to 42 days. Randomisation may occur as soon as all Screening results are available.
- For subjects who completed rendomised DTG through Week 52 and entered into the DTG Continuation Phase: subjects completing the DTG Continuation Phase must return to the clinic when transitioning to commercial supplies. Conduct study assessments, with the exception of dispensing IP, as specified for all Continuation Phase visits at this end of Continuation Phase visit.
- c. A follow-up visit will be conducted 4 weeks after the last dose of study provided IP and is required only if a subject has ongoing AEs or laboratory abnormalities at the last on-study visit. The assessments performed should reflect what is considered medically necessary to assess the event(s).
- d. Inclusion/exclusion criteria will be fully assessed at the Screening visit. Changes between the screening visit and the Day 1 visit should be assessed to ensure eligibility, including additional assessments performed at Day 1.
- e. Full medical history will be collected. Targeted Medical History assessments will include cardiovascular, gastrointestinal (e.g. Gl bleeding, PUD, etc), metabolic (e.g. Type I or II DM), psychiatric (e.g. depression), renal (e.g. nephrolithiasis, nephropathy, renal failure) and neurological disorders.

  f. Limited physical examination to include blood pressure at Baseline (recorded in eCRF) for Framingham score assessment. Blood pressure to be measured after resting in a semi-
- supine position for at least 5 minutes.
- Assessment for cardiovascular risk will include height, weight, blood pressure, smoking history, medical conditions, and family history of premature cardiovascular disease. On Day 1, the Columbia Suicidality Severity Rating Scale is to be administered prior to randomisation.
- Only SAEs related to study participation or to a concomitantly administered GSK/ViV product will be collected between obtaining informed consent and administration of IP at Day
- At Week 52, repeat HIV-1 RNA testing will only be performed for subjects with HIV-1 RNA ≥50 o'mL at Week 48.
- k. Plasma samples for storage will be collected at each visit for possible future analyses (including but not limited to HIV-1 RNA genotypic and phenotypic analyses, HIV-1 RNA levels, and immunological parameters). These samples will be used when needed such as when samples are lost or arrive at the laboratory unevaluable. Additionally, for genotypic and phenotypic resistance analyses Baseline samples from all subjects will be used and later samples in cases of confirmed virologic withdrawal criteria met (for paired baseline and endpoint genotypes).
- Subjects starting ABC as one of the NRTIs should have been screened and be negative for the HLA-8\*5701 allele.
- m. An overnight fast is preferred, however a minimum of a 6 hour fast is acceptable.
- n. Pregnancy testing will be conducted (women of child bearing potential only) on serum (S) samples with the exception of Day 1, which must be a urine (U) test to confirm status prior to administration of IP.
- o. Subjects who are hepatitis B surface antigen (HBsAg) positive require appropriate HBV therapy based on local guidelines (see Section 6.2.3 for details).
- Suppose minor in repense a parience arrange in reading possive require appropriate now merepy based on local guidelines (see Section 8.2.3 for details).
   HBV DNA testing will be performed on Day 1 for subjects with negative HBsAg and positive hepatitis B core antibody (anti-HBs) results at Screening. Subjects with positive anti-HBs and positive HBV DNA results require appropriate HBV therapy based on local guidelines (see Section 6.2.3 for details).
   Informed consent for optional pharmacogenetics (PGx) research must be obtained before collecting a sample. Collection of the PGx sample at Day 1 is preferred; however, this sample are not provided at least time of the sample and the collection of the PGx.
- sample may be collected at any time during the study.
- Whole blood collection (please refer to the SPM).
  For subjects receiving DTG during the Continuation Phase only.

# 11.3. Appendix 3: Assessment Windows

Laboratory data, vital signs, health outcomes assessments, and genotypic and phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database. The CVW algorithm will be derived using nominal CRF visit rather than using the assessment window defined below.

A window around a target Study Day will typically include all days from the midpoints between it and the target Study Days of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w)+1.

Based on the Study Day (see Section 11.6.1), assessments are assigned as shown in Section 11.3.1.

## 11.3.1. **Definitions of Assessment Windows for Analyses**

| Analysis Set / | Parameter | Target | Analysis | Analysis | |
|---|---|---|---|---|---|
| Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| Efficacy | Snapshot<br>(MSDF)<br>endpoints | -28 | ≤-4 | ≤-4 | Screen |
| | | 1 | -3 | 1 | Day 1 |
| | | 29 | 2 | 42 | Week 4 |
| | | 57 | 43 | 84 | Week 8 |
| | | 113 | 85 | 126 | Week 16 |
| | | 169 | 127 | 210 | Week 24 |
| | | 253 | 211 | 294 | Week 36 |
| | | 337 | 295 | 378 | Week 48 |
| | | 421 | 379 | 462 | Week 60 |
| | | 7*w + 1 | (7*w – 41) | (7*w + 42) | Week w<br>w = 72, 84,<br>96, |
| | | Study Day of last dose<br>+ 28 | > (Study<br>Day of last<br>dose + 1) | > (Study<br>Day of last<br>dose + 1) | Follow-up |
| Safety/Virology<br>/Health<br>Outcome | | -28 | <u>≤-4</u> | <u>≤-4</u> | Screen |
| | | 1 | -3 | 1 | Day 1 |
| | | 29 | 2 | 42 | Week 4 |
| | | 57 | 43 | 84 | Week 8 |
| | | 113 | 85 | 126 | Week 16 |
| | | 169 | 127 | 210 | Week 24 |
| | | 253 | 211 | 294 | Week 36 |

| Analysis Set / | Parameter | Target | Analysis | Analysis | |
|---|---|---|---|---|---|
| Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| | | 337 | 295 | 350 | Week 48 |
| | | 365 | 351 | 392 | Week 52 |
| | | 421 | 393 | 462 | Week 60 |
| | | 7*w + 1 | (7*w – 41) | (7*w + 42) | Week w<br>w = 72, 84,<br>96, |
| | | Study Day of last dose<br>+ 28 | > (Study<br>Day of last<br>dose + 1) | > (Study<br>Day of last<br>dose + 1) | Follow-up |

#### NOTES:

- For key timepoints at Week 24 and Week 48, the efficacy windows have been defined to cover ± 6 weeks, regardless of the midpoint between adjacent target Study Days. The windows for the adjacent periods are adjusted accordingly.
- For parameters that are not scheduled to be assessed at particular visits, the all-inclusive windows defined above will still be used; however, data summaries will only report scheduled visits. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g. snapshot).
- See Section 11.6.1 for how to handle multiple assessments within a time window.

# 11.4. Appendix 4: Treatment States and Phases

# 11.4.1. Study Phases

All displays are for the randomised phase only, unless specified otherwise. This means that the analysis other than "by-visit" summaries will not be windowed at Week 24 (AEs, maximum post-baseline toxicities). In other words, all data collected up to the point of DBF will be included in summary statistics, which could be past week 24 for subjects enrolled early in the study. However, at the Week 48 analysis, summary statistics for the randomised phase will only include data up to Week 52 for both arms.

For subjects entering the continuation phase, which phase an assessment or an event occurred in will be determined by comparing the event date with the week 52 visit date.

The study phases are defined as follows:

| Phase | Start | End |
|---|---|---|
| Randomised Phase | IP start date | Week 52 DOV, IP end date or<br>Withdrawal date if on or before Week<br>52 DOV |
| Continuation Phase | Week 52 DOV | IP end date or Withdrawal date if post Week 52 DOV |

## 11.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

# 11.4.2.1. Treatment States for HIV-1 RNA Data, Laboratory Data, HIV Associated Conditions, Vital Signs, , Health Outcomes assessments, and Genotypic and Phenotypic Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date +1 |
| Post-Treatment | Date > Study Treatment Stop Date +1 |

## NOTES:

If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 11.4.2.2. Treatment States for AE Data

For adverse events, a partial AE start date uses imputation as described in Section 11.7.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date – Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date – Treatment Start Date +1 Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing]. |

#### NOTES:

- In the case of a completely missing start date, the event will be considered to have started On-treatment unless
  an end date for the AE is provided which is before start of investigational product; in such a case the AE is
  assigned as Pre-treatment.
- If the IP Stop Date is missing, then any event with a start date on or after IP Start Date will be considered to be On-treatment. If the start date of the AE is after IP Stop Date but has been recorded as potentially related to IP, then it will be classified as On-treatment.

## 11.4.2.3. Treatment States for Prior/Concomitant/Post-Therapy Medications Data

- Prior medications are those taken (i.e., started) before the start date of investigational product.
- Concomitant medications are those taken (i.e., started or continued) at any time between the start date and stop date of IP, inclusive. Prior medications that were continued during this period are also considered as concomitant medications.
- Post-treatment medications are those started after the stop date of IP. Concomitant medications that were continued during this period are also considered as post-treatment medications.

It will be assumed that medication has been taken on the date in which it is reported as started or stopped. Also, for any medication starting on the same date as IP, it will be assumed that the medication was taken after the subject started taking IP.

ART medications will also be classified as prior, concomitant and/or post-treatment according with the following modifications:

- ART starting on study treatment stop date will be considered as only posttreatment and not concomitant. It is expected that after discontinuation of study treatment, a subject may immediately begin taking another ART. (Note: this is different to concomitant medications which are considered concomitant and posttreatment if they start on the IP stop date).
- ART stopping on study treatment start date will only be considered as prior and not concomitant. (Note: this is different to concomitant medications which are

considered concomitant and post-treatment if they start on the IP stop date). Any ART entered on the Prior ART eCRF with partial end date will be assumed to have finished before Screening.

Table 10 Concomitant, and Post-treatment Classification of Medications

| | Pre-<br>treatment | | On-treatment | | Ро | Post-treatment | | Conco-<br>mitant | Post |
|---|---|---|---|---|---|---|---|---|---|
| (a) | хх | | | | | | Υ | N | N |
| (b) | X | | ———х | | | | Υ | Υ | N |
| (c) | x | | | | | ———х | Υ | Υ | Υ |
| (d) | _ | | хх | | | | N | Υ | N |
| (e) | | e. | X | e. | + | ———х | N | Υ | Υ |
| (f) | | IP Start Date | | IP Stop Date | IP Stop Date+1 | xx | N | N | Υ |
| (g) | ?——x | art | | do | р D | | Υ | N | N |
| (h) | ? | St | ———х | St | Sto | | Υ* | Υ | N |
| (i) | ? | <u> </u> | | 4 | П | ———Х | Y* | Y* | Y |
| (j) | X | | | | | ? | Υ | Y** | Y** |
| (k) | _ | | X | | | ? | N | Υ | Y** |
| (l) | | | | | | x? | N | N | Υ |
| (m) | ? | | | | | ? | Y*** | Y*** | Y*** |
| (n) | X | Х | | | | | Υ | Y | N |
| (o) | ? | Х | | | | | Y* | Υ | N |
| (p) | | Х | ———х | | | | N | Υ | N |
| (q) | | Х | | Х | | | N | Υ | N |
| (r) | | | | Х | | ———х | N | Υ | Υ |
| (s) | | | | Х | | ? | N | Υ | Y** |
| (t) | | | | | Χ | x | N | N | Υ |
| (u) | | | | | Χ | ? | N | N | Υ |
| (v) | | | х | | Х | | N | Y | Υ |

x = start/stop date of medication

<sup>? =</sup> missing start/stop date of medication

<sup>\*</sup> If a medication is stopped On-treatment or Post-treatment and no start date is recorded it will be assumed that the medication was ongoing from the Pre-treatment phase

<sup>\*\*</sup> If a medication is started Pre-treatment or On-treatment and no stop date is recorded then usage will be assumed to be ongoing for the remainder of the study

<sup>\*\*\*</sup> If a medication has no start or stop date it will be assumed that the medication was ongoing from the Pretreatment phase to the Post-treatment phase

## 11.4.3. Post-treatment Assessments and Phases

On-treatment and Post-treatment assessments and events will be classified as occurring during the Randomised Phase or the Continuation Phase of the study as follows:

- If a subject did not enter the Continuation Phase, then any Post-treatment data will be assigned to the Randomised Phase.
- For subjects who did enter the Continuation Phase, any Post-treatment data will be assigned to the Continuation Phase.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

## 11.5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order [1] |
| Α | Dolutegravir 50mg once daily | DTG | 1 |
| В | Lopinavir/ritonavir 800mg/200mg once daily or 400mg/100mg twice daily | LPV/RTV | 2 |

#### NOTES:

#### 11.5.2. **Baseline Definition & Derivations**

#### 11.5.2.1. Baseline Definitions

For all endpoints (unless stated otherwise) the baseline value will be the latest pre-dose assessment. This is generally expected to be from the Day 1 visit, although such values may be missing or unscheduled assessments may be performed before treatment start.

In the scenario where the treatment start date is more than 2 weeks after randomisation date, the randomisation date will be used as baseline for change from baseline. Therefore, for example, the week 12 visit data would be included in the week 12 visit summary rather than the week 8 visit summary. All analyses will use this rule, except for resistance analyses; as the resistance test at or just before treatment start is more representative of a patient "baseline" rather than the randomisation date, since patients would have stayed on a failing regiment for longer than they should have.

## Example:

A subject was randomised on 26Feb2016 but did not start IP until 18Mar2016. Baseline will be 26Feb2016 for everything apart from resistance analyses where baseline will be 18Mar2016.

## 11.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| | = Calculate the change from baseline at each given timepoint |
| Maximum Change from Baseline | |
| | and determine the maximum change |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

## 11.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | Software |
| The currently support to the currently su | The currently supported versions of SAS software and TSCG will be used. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : \ARPROD\GSK1349572\200304 |
| QC Spreadsheet | : \ARPROD\GSK1349572\200304\(Week24, Week48 or Final)\Documents |
| <b>Analysis Datasets</b> | |
| <ul> <li>Analysis datasets will be created according to according to CDISC standards (SDTM IG<br/>Version 3.1.3 &amp; AdaM IG Version 1.0.</li> </ul> | |
| <ul> <li>For creation of AdaM datasets (ADCM/ADAE), the same version of dictionary datasets will be<br/>implemented for conversion from SI to SDTM.</li> </ul> | |

## **Generation of RTF Files**

RTF files will be generated for every reporting effort.

## **Reporting Standards**

### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

## **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Actual time relative to dosing will be used in figures, summaries, statistical analyses and

## **Reporting Standards**

calculation of any derived parameters, unless otherwise stated.

- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

## **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section 11.3.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the T&E table).
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

## **Invalid Laboratory Assessments**

 Certain laboratory endpoints are required to be collected in a fasting state, i.e., glucose and lipids (triglycerides, total cholesterol, HDL, LDL). If these endpoints are collected in a nonfasting state, then the results will be excluded from summaries; such results will be included in data listings with the fasting status noted.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7 01 to 7 13 | |

# 11.6. Appendix 6: Derived and Transformed Data

## 11.6.1. Week 24 cut off date

For the week 24 interim it is necessary to define a cut-off for the purposes of defining prohibited medications and also for the calculation of total time on treatment during the Week 24 time period.

To be considered prohibited the medication has to be taken before the date of Week 24 viral load. If the date of the Week 24 viral load is before the prohibited medication was taken then this does not impact the snapshot algorithm. If the Week 24 viral load date is missing then the cut off date is defined as follows:

- For subjects who have a Week 24 visit: use Week 24 date from Visit dataset (SV).
- For subjects who have withdrawn (or last IP end date) before Week 24:visit use the minimum of: withdrawal date, disposition date, last visit date, last drug exposure date (while taking into account study drug interruptions) and last laboratory date.
- For subjects who have not withdrawn but no IP stop date or week24 visit date yet: Cut-off= IP start date + week24studyday 1

where week24studyday could be 169 (the target date of wk24 window) or 210 (upper bound of wk24 window).

The last exposure data should use both EXSTDTC and EXENDTC in case the IP was interrupted and re-started.

This cut-off date also applies for the calculation of total on treatment during Week 24.

A similar approach will be used for the Week 48 cut-off.

#### 11.6.2. **General**

## Multiple Measurements at One Time Point

- If after window assignment (see Section 11.3), there are multiple valid assessments of a
  parameter within the same window, then the following hierarchy will be used to determine the
  value to be used for summary statistics of observed values:
  - the assessment closest to the window target Study Day;
  - if there are multiple assessments equidistant from the target Study Day, then the
    mean of these values will be used. For HIV-1 RNA, the geometric mean of the
    number of copies will be used as opposed to the arithmetic mean
- Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings. Also, such valid assessments will be used when determining values of

## Multiple Measurements at One Time Point

potential clinical concern for the 'any time On-treatment' time point, and for any algorithm that has specific rules for which observation to use (e.g., MSDF or LOCF).

- In the event of laboratory re-tests being performed the last re-test in the visit window will be used. For example:
  - If a subject had a week 24 viral load and then two re-tests (ie three viral loads labeled as week 24, unscheduled 1 unscheduled 2). and the first two viral loads were within the upper bound of the week 24 visit (Day 210) but the last re-test was slotted to week 36 then the last re-test would not be used for the week 24 snapshot.
  - If a subject had a week 24 viral load but the re-test was performed on Day 220 (week 36) then the re-test viral load would not be used for the week 24 snapshot.

## Study Day

- Calculated as the number of days from the initial treatment start date :
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Treatment Start Date → Study Day = Ref Date Treatment Start Date
  - Ref Data ≥ Treatment Start Date → Study Day = Ref Date (Treatment Start Date) + 1

Note that Treatment Start Date is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

## Post-baseline

 Post-baseline refers to the combined time periods of On-treatment and Post-treatment (Section 11.4.2). Post-baseline may be further specified according to phase of the study: Randomised or Continuation (Section 11.4.1).

# 11.6.3. Study Population

## **Demographics**

## Age

- Age, in whole years, will be calculated with respect to the subject's Screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied.
   Consequently, the age of the subject will not be calculated and will remain missing.

## **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

# **Background ART**

 For purposes of calculating susceptibility scores (Section 11.6.6), a subject's baseline background ART regimen is defined as the last full regimen received at the end of the Week 4

## **Demographics**

visit window. This allows time to accommodate any early, protocol-permitted changes in background ART or for short, unexpected delays in implementing the chosen background NRTI regimen

## WHO First Line and Second Line Regimen

## First line combination regimen is defined as follows:

```
TDF + 3TC + EFV
TDF + FTC + EFV
AZT + 3TC + EFV
AZT + FTC + EFV
D4T + 3TC + EFV
D4T + FTC + EFV
AZT + 3TC + NPV
AZT + FTC + NPV
D4T + 3TC + NPV
D4T + FTC + NPV
TDF + 3TC + NVP
TDF + FTC + NVP
```

## Second line combination regimen is defined as follows:

```
AZT + 3TC + LPV/r
TDF + 3TC + LPV/r
TDF + FTC + LPV/r
```

## Framingham Risk Equation

The predicted probability,  $\hat{p}$ , of having a cardiovascular disease (CVD) within the next 10-years according to the Framingham formula [D'Agostino, 2008] is

```
for females:
```

```
\vec{p}_F = 1 - S_0(t) \exp\{2.32888 \times \log(\text{age}) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 2.76157 \times \log(SBPu) + 2.82263 \times \log(SBPt) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 2.76157 \times \log(SBPu) + 2.82263 \times \log(SBPt) + 1.20904 \times \log(TC) + 1.20904 \times 
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                 0.52873 \times I_s + 0.69154 \times I_d - 26.1931
```

## for males:

```
\vec{p}_{M} = 1 - S_{0}(t) \exp\{3.06117 \times \log(\text{age}) + 1.12370 \times \log(TC) - 0.93263 \times \log(HDL) + 1.93303 \times \log(SBPu) + 1.99881 \times \log(SBPt) +
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                   0.65451 \times I_{s} + 0.57367 \times I_{d} - 23.9802
```

#### where

```
S_0(t) = \begin{cases} 0.95012, \text{ females} \end{cases}
            l 0.88936, males
```

TC = total serum cholesterol (mg/dL),

HDL = serum HDL cholesterol (mg/dL),

SBPu = systolic blood pressure (mmHg) if subject is not treated for high blood pressure (note that if a subject is treated for high blood pressure then log(SBPu) = 0)

SBPt = systolic blood pressure (mmHg) if subject is treated for high blood pressure (note that if a subject is not treated for high blood pressure then log(SBPt) = 0)

## **Demographics**

$$I_{s} = \begin{cases} 1, \ current \ smo \ ker \\ 0, \ otherwise \end{cases}$$

$$I_{d} = \begin{cases} 1, \ diabetic \\ 0, \ otherwise \end{cases}$$

- A subject will be considered as treated for high blood pressure if during screening it has specified that is suffering from hypertension.
- A subject is classified as diabetic if current or past is indicated in the medical conditions eCRF for Type 1 or Type 2 diabetes mellitus, or if baseline fasting glucose ≥7.00 mmol/L (126 mg/dL).
- Smoking status is collected in the eCRF on Day 1. A current smoker is defined as currently smoking/using tobacco or has smoked/used tobacco within the previous 6 months; a former smoker is defined as previously smoked/used tobacco products and has not smoked/used tobacco products within the previous 6 months.
- This calculation will not be performed for subjects who have indicated current or past
  myocardial infarction conditions on the eCRF. These subjects will not be included in
  summary statistics of risk, but will be counted in the highest category of risk in the summary
  by category.

# 11.6.4. **Safety**

# **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Subjects who were randomised but did not report a treatment start date will be categorised as having zero days of exposure.
- Missing Treatment Stop Date will be imputed, for purposes of calculating exposure, as the date of last visit or the recorded date of withdrawal/completion, whichever is earlier.
- An alternative calculation of exposure will be performed where the duration of any dosing interruptions based on eCRF data will be subtracted from the result above
  - The ratio (percentage) of the actual exposure to the overall exposure (i.e. study treatment stop date study treatment start date+1) will be used to define protocol deviation leading to exclusion from PP Population due to study treatment interruption (i.e. >10%).

#### **ECG Parameters**

Not applicable as not routinely collected.

## **Adverse Events**

# **AE Severity – DAIDS Grading**

- The DAIDS grading for severity of clinical adverse events will be performed.
- See protocol for DAIDS grading criteria.

## **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

## Lab Toxicities – DAIDS Grading

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, as specified in the protocol.
- Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a particular parameter.
- When summarising toxicity grades for such parameters, they will be categorised according to whether they are above or below the midpoint of normal range.

| Parameter | Below Midpoint | Above Midpoint |
|----------------|----------------|----------------|
| Fasted glucose | Hypoglycaemia | Hyperglycaemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |

## National Cholesterol Education Program (NCEP) Lipid Categories

• In addition to DAIDS toxicity scales (see protocol), lipid values will be categorised according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001].

| Parameter | Value Range (mmol/L) | Value Range (mg/dL) | Category |
|---|---|---|---|
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |
| | 5.18 to <6.21 | 200 to <240 | Borderline High |
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |
| | 1.04 to <1.56 | 40 to <60 | Normal |
| | ≥1.56 | ≥60 | High |
| LDL Cholesterol | <2.59 | <100 | Optimal |
| | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | 4.14 to <4.92 | 160 to <190 | High |
| | ≥4.92 | ≥190 | Very High |

## Total Cholesterol / HDL Cholesterol Ratio

 When both total cholesterol and HDL cholesterol results are available from the same date for a subject, then the ratio will be calculated by dividing the total cholesterol result by the HDL cholesterol result.

## **Hepatitis Status**

- Hepatitis C status will be determined using antibody (anti-HCV) assessments performed during screening.
- A subject will be considered chronically infected with hepatitis B virus (HBV) if they test HbsAg
  positive OR anti-HBc positive with HBV DNA present (HBV DNA is determined at Baseline for
  subjects who are tested HbsAg negative and anti-HBc positive at Screening).

## **Other Safety Endpoints**

## **Columbia Suicide Severity Rating Scale (C-SSRS)**

- Missing data will not have any imputation performed.
- Incomplete calls:
  - when no complete call is databased on the same day, the incomplete data will be used
  - when a complete call is databased on the same day, the data from the complete call will be used in the summaries.
- Duplicate calls:
  - If they occur on the same day, the latest entry will be used.
  - If they occur on different days, take the entry closest to the target visit date.

## 11.6.5. **Efficacy**

## **Efficacy**

## **Snapshot (Missing, Switch or Discontinuation=Failure)**

- The FDA's "snapshot" algorithm is also known as the MSDF algorithm. It is intended to be
  primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy.
- Virologic Success (e.g., <50 c/mL) or Virologic Failure within an analysis window (see Section 11.3) is typically determined by the last available HIV-1 RNA measurement in that window while the subject is On-treatment.
- When no HIV-1 RNA data is available within a window, a subject cannot be a Virologic Success. Depending on the reason for lack of data, the subject will be classified as a Virologic Failure or reported as 'No Virologic Data at Week X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a subject withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Week X'. Should a subject withdraw for reasons other than AE and was not suppressed at the time, they will be a Virologic Failure.
- A subject may also be considered a Virologic Failure if they make changes to their background regimen. This includes:
  - background ART substitutions not permitted per protocol;
  - background ART substitutions permitted per protocol unless the decision to switch is documented as being before or at the first On-treatment visit where HIV-1 RNA is assessed.
- For each scheduled assessment time, the MSDF (also known as snapshot) response rate for a given threshold (e.g., <50 c/mL) is defined as:</li>

## **Efficacy**

Number of responders in that analysis window Snapshot Rate = Number of subjects in the analysis population

Full details of the algorithm, including the handling of special cases, are included in Section 11.13.

## Treatment and Efficacy Related Discontinuation = Failure (TRDF and ERDF)

- The analysis of time to confirmed virologic withdrawal criteria (CVWC) or discontinuation due to treatment related reasons (i.e., drug-related AE, protocol defined safety stopping criteria, or lack of efficacy) will censor subjects who have not met CVW criteria and are ongoing in the study, or who have discontinued for reasons other than those related to treatment. This will be the Treatment Related Discontinuation = Failure (TRDF) data.
- Subjects who have not met CVW criteria and are ongoing in the study, or who have discontinued for reasons other than lack of efficacy, will be censored in the analysis of the Efficacy Related Discontinuation = Failure (ERDF) data.

## Plasma HIV-1 RNA

- For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used
- HIV-1 RNA results may be provided as censored values, such as <40 or >9.999.999 c/mL. For the purposes of summary statistics, such values will be replaced by the next value beyond the limit of detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data listings will show the censored values as provided.

## Variance Estimator of Cochran Mantel-Haenszel Risk Difference

$$\hat{\text{var}}(\hat{d}_{cmh}) = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum n_k m_k / N_k\right)^2} = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum W_k\right)^2}$$

where

$$P_{k} = \frac{n_{k}^{2} y_{k} - m_{k}^{2} x_{k} + n_{k} m_{k} (m_{k} - n_{k})/2}{N_{k}^{2}}$$

$$Q_{k} = \frac{x_{k} (m_{k} - y_{k})/N_{k} + y_{k} (n_{k} - x_{k})/N_{k}}{2}$$

$$Q_k = \frac{x_k (m_k - y_k) / N_k + y_k (n_k - x_k) / N_k}{2}$$

## **CVW** Derivation

There are 3 parts to the derivation of CVW. All parts of the derivation need to use nominal visits (i.e. VISIT and VISITNUM).

## Virologic Non-response (Parts 1 &2)

- A decrease in plasma HIV-1 RNA of less than 1 log<sub>10</sub> c/mL by Week 16, with subsequent confirmation, unless plasma HIV-1 RNA is <400 c/mL.</li>
- Confirmed plasma HIV-1 RNA levels ≥400 c/mL on or after Week 24.

## **Virologic Rebound (Part 3)**

 Confirmed rebound in plasma HIV-1 RNA levels to ≥400 c/mL after prior confirmed suppression to <400 c/mL.</li>

A patient can only be classified as CVW for the analyses if the patient is on-treatment at the time of the HIV-RNA value.

# Part 1. A decrease in Plasma HIV-1 RNA of less than 1 log10 c/mL by week 16, with subsequent confirmation, unless Plasma HIV-1 RNA is <400 c/mL

- This applies to Week 16 data only (where INT(VISITNUM)=80)
- If there is a decrease < 1 log10 from Baseline at Week 16 and LBORRESN>=400, then -> suspected virologic withdrawal
- If there is a confirmatory sample, then check if there is a decrease <1 log10 from Baseline and the LBORRESN>=400 then confirmed virologic withdrawal
- The protocol states that the confirmatory sample needs to be taken within 1-4 weeks of initial sample, unless one of the extenuating circumstances outlined below apply:

The following guidelines will be followed for scheduling confirmatory HIV-1 RNA testing in an effort to avoid false-positive results:

- Confirmatory testing should be scheduled 2 to 4 weeks following resolution of any intercurrent illness, during which time the subject should receive full dose of all IP.
- Confirmatory testing should be scheduled at least 4 weeks following any immunisation, during which time the subject should receive full dose of IP.
- If therapy is interrupted due to toxicity management, non-compliance, or other reasons, confirmatory testing should be scheduled 2 to 4 weeks following resumption of full dose of IP.
- The subject should have received full doses of IP for at least 2 weeks at the time confirmatory plasma HIV-1 RNA is done.

Example: subject PPD

| subject | nominal<br>visit | visit date | c/mL | log10<br>c/mL | log10<br>decrease<br>from BL | CV<br>outcome | comments |
|---|---|---|---|---|---|---|---|
| PPD | Baseline | PPD | 3398 | 3.53 | | | |
| | Week 4 | | 39 | 1.59 | 1.94 | | |
| | Week 8 | | 2354 | 3.37 | 0.16 | | |
| PPD | Week 16 | PPD | 368742 | 5.56 | -2.03 | Suspected virologic withdrawal | <1 log 10<br>decrease<br>from<br>baseline,<br>and value<br>>400 c/mL |
| PPD | Week 16 | PPD | 17293 | 4.24 | -0.71 | Confirmed virologic withdrawal | <1 log 10<br>decrease<br>from<br>baseline,<br>and value<br>>400 c/mL |

Example subject PPD

| subj | | nominal<br>visit | visit date | c/mL | log10<br>c/mL | log10<br>decrease<br>from BL | CV outcome | comments |
|---|---|---|---|---|---|---|---|---|
| _ | PPD | Baseline | PPD | 38286 | 4.58 | | | |
| | | Week 4 | | 332 | 2.52 | 2.06 | | |
| | | Week 8 | | 66 | 1.82 | 2.76 | | |
| | | Week 16 | | <50 | <1.70 | 2.99 | | |
| | | Week 24 | | 87394 | 4.94 | -0.36 | suspected<br>virologic<br>withdrawal | value >400<br>on/after weel<br>24 |
| F | PPD | Week 24 | PPD | 413 | 2.62 | 1.97 | confirmed<br>virologic<br>withdrawal | Consecutive value >400 on/after weel 24 |

## Part 2: Confirmed Plasma HIV-1 RNA levels >=400 c/mL on or after Week 24

- If patient is not already a confirmed VF due to the rules in Part 1, we can then continue to check the results from Week 24 onwards
- Use nominal visits i.e. int(visitnum)>=100
- If a patient has a sample on/after Week 24 and the result is >=400 then -> suspected virologic withdrawal.
- If a patient then has a 2nd consecutive sample >=400 then -> confirmed virologic withdrawal.

# Part 3: Confirmed rebound in plasma HIV-1 RNA levels to >=400 c/mL after prior confirmed suppression to <400 c/mL

- Virologic rebound can happen at any visit.
- Patient must have 2 consecutive values <400, followed by 2 consecutive values >=400.
- Once a patient has 2 consecutive values <400, if the next value is >=400 this is a suspected rebound
- If a patient then has a 2nd consecutive sample >=400 then this is a confirmed rebound
- Subject PPD (above) is classified as virologic rebound, as they have values <400 at Weeks 4, 8, and 16, then continues to have 2 consecutive values >=400. On subject is a 'confirmed rebound'. Also see subject PPD below:

Note that there is greater than 1-4 weeks (PPD from suspected sample to confirmed sample, hence this rule has not been applied

| subject | nominal<br>visit | visit date | c/mL | log10<br>c/mL | log10<br>decrease<br>from BL | CV<br>outcome | comments |
|---|---|---|---|---|---|---|---|
| PPD | Baseline | PPD | 303007 | | | | |
| | Week 4 | | 270 | 2.43 | 3.05 | | |
| | Week 8 | | 140 | 2.15 | 3.33 | | |
| PPD | Week 16 | PPD | 29153 | 4.46 | 1.02 | Suspected rebound | 2 consecutive<br>values <400,<br>followed by an<br>initial value<br>>=400 |
| PPD | week 16 | PPD | 454 | 2.66 | 2.82 | Confirmed rebound | 2 consecutive<br>values <400,<br>followed by 2<br>consecutive<br>values >=400 |
| | Withdrawal | | <40 | 1.59 | 3.89 | TODOUTIU | Tuluco - 100 |

## 11.6.6. **Virology**

## Genotype

## Amino Acid Changes

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may
  not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the
  number of mutated amino acids, only one mutation is considered to be present at the codon of
  interest

| Representation of Amino Acid Changes | |
|---|---|
| Mutations | Amino acid change |
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' (vendor |
| | reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

 Treatment-emergent genotypic mutations are defined as mutations that appear between baseline and an On-treatment assessment (e.g., at time of confirmed virologic withdrawal criteria).

#### Resistance Associated Mutations

Known INI mutations associated with the development of resistance to RAL, EVG or DTG:

| HIV Integrase for | H51Y, <b>T66A/I/K</b> , L74M, <b>E92Q/V</b> /G, Q95K, T97A, G118R, F121Y, E138A/K/D, G140A/C/S, <b>Y143C/H/R/K/S/G/A, P145S, Q146P, S147G, Q148H/K/R</b> , |
|---|---|
| Analysis | V151I/L/A, S153F/Y, N155H/S/T, E157Q, G163R/K, S230R, R263K, |
| | L68V/I*, L74I*, E138T*, V151I*, G193E* |

#### NOTES:

- Draft listing; may be modified in case of additional substantive data availability.
- INI mutations listed taken from Stanford HIV Resistance Database (https://hivdb.stanford.edu/hivdb/by-mutations/http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INI cited PPD and accessed on PPD
- Each INI mutation listed had a score of ≥15. INI substitutions listed above in bold had a score of =60.
- \* Denotes additional INI mutations added as they were identified during in vitro passage of DTG or seen in a previous DTG study in INI-experienced subjects (ING112574).
- Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis.
| Class | Mutations |
|---|---|
| NRTIs | M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, F116Y, Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, |
| | Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L, |
| Pis | D30N,V32I, M46I/L, I47A/V, G48V, I50V/L, I54M/L, Q58E, T74P, L76V, |
| | V82A/T/F/L/S, N83D, I84V, N88S,L90M |

Note: List generated from Wensing, 2014

#### Susceptibility Scores

#### Stanford Genotypic Susceptibility Score (GSS)

- To establish genotypic susceptibility to background treatment, a genotypic sensitivity score will be calculated.
- Genotypic sensitivity to each drug will be assessed using the HIVdb, the Integrated Genotypic Resistance Interpretation System [Liu, 2006].
- In the HIVdb system, each HIV-1 drug resistance mutation is assigned a drug penalty score.
   The penalty scores for each drug resistance mutation are available at

NNRTI: https://hivdb.stanford.edu/dr-summary/mut-scores/NNRTI/

NRTI: https://hivdb.stanford.edu/dr-summary/mut-scores/NRTI/

PI: https://hivdb.stanford.edu/dr-summary/mut-scores/PI/

INSTI: https://hivdb.stanford.edu/dr-summary/mut-scores/INSTI/. Scores for particular patterns of INSTIs are also available at https://hivdb.stanford.edu/dr-summary/pattern-scores/INSTI/

The drug resistance estimate is obtained by adding together the penalty scores from all
mutations associated with resistance to that drug and then a numeric score (S-GSS) is applied
for each drug as shown below. The sum scores are titrated to fall within the following ranges:
susceptible, potential low-level resistance, low-level resistance, intermediate resistance, and
high-level resistance (see table below).

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

 For a drug which is not assessed by HIVdb (e.g., enfuvirtide), this drug will be assigned a numeric score of 0 if ccl

and 1 if ccl (see Table 11). Maraviroc will be assigned a score of 0 if and

1 if CCI

The HIVdb GSS will then be calculated for each subject defined as the sum of the resistance

scores for each of their background drugs.

#### Monogram Genotypic Susceptibility Score (GSS)

 Genotypic sensitivity to each drug will be assessed using the Monogram resistance score for each background drug provided in the database.



 The Monogram GSS will then be calculated for each subject defined as the sum of the resistance scores for each of their background drugs.

#### Phenotypic Susceptibility Score (PSS)

To establish susceptibility to background treatment, a phenotypic sensitivity score will be
calculated. Phenotypic susceptibility to each drug in a subject's background regimen will be
determined by applying drug-associated cutoffs as defined by the PhenoSense algorithm to the
phenotypic fold resistance to that drug at a certain timepoint (e.g., Screening or Baseline). A
numeric score will be assigned to each background drug using two different methods: one with
full sensitivity only (PSSf; Table 11) and one with partial sensitivity included (PSSp; Table 12).

#### Table 11 PSS with Full Sensitivity Only (PSSf)

| Fold Change | Score | Interpretation |
|--------------------------------------------|-------|----------------|
| > clinical lower cutoff or biologic cutoff | CCI | |
| ≤ clinical lower cutoff or biologic cutoff | | |

#### Table 12 PSS with Partial Sensitivity Included (PSSp)

| Fold Change | Score | Interpretation |
|---|---|---|
| > clinical higher cutoff | CCI | |
| ≤ clinical higher cutoff and > clinical lower cutoff | | |
| ≤ clinical lower cutoff | | |

- If only a biological cutoff is available, the algorithm for PSSf will be applied. Maraviroc will be assigned a score of 0 if the column , and 1 if the column .
- Both PSSf and PSSp will be calculated separately for each subjected defined as the sum of the resistance scores for each background drug.

| Drug | Abbreviation | Class | PhenoSense cutoff |
|---------------|--------------|-------|--------------------------|
| Abacavir | ABC | NRTI | (4.5 − 6.5) <sup>a</sup> |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |

| Tenofovir | TDF | NRTI | (1.4 – 4) a |
|-----------------|-------|-------|----------------------|
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivarine | RPV | NNRTI | 2 |
| Fosamprenavir/r | FPV/r | Pl | (4-11) a |
| Atazanavir/r | ATV/r | PI | 5.2 a |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) a |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
| Tipranavir/r | TPV/r | PI | (2 – 8) <sup>a</sup> |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |

a. clinical cutoff (lower cutoff – higher cutoff)

#### Net Assessment for Optimised Susceptibility Scoring

#### Resistance Data from China

At the time of the Week 24 analysis not all of the phenotype data may be available from Monogram for subjects in China. The genotype data may be a mixture of Q2 and Monogram data, and in the event that both Q2 and Monogram are available at the same timepoint the Monogram data will be used.

Day 1 genotypic and phenotypic resistance data for RT and PRO is provided for all subjects by Monogram and will be used in the analysis. Subjects with CVW criteria will also have resistance testing performed by Monogram at SVW timepoints. PSS is only provided by Monogram. The screening genotype from QUEST may be used if Monogram genotype is missing.

#### Definition of TAMS

TAMS are thymidine analogue mutations and are a combination of the thymidine analogues AZT (ZDV) mutations and d4T mutations in RT (reverse transcripitase). They can be found at the Stanford database, details are included in the following table:

| | Thymidine Analog Mutations (TAMs) | | | | | |
|---|---|---|---|---|---|---|
| Amino acid position in RT | 41 67 70 210 215 219 | | | | | |
| Wild type | M | D | K | L | T | K |
| Muations | L | N | R | W | FY | QE |

#### 11.6.7. **Health Outcomes**





#### MMAS-8

#### **Total Score**

- Derived as the summation of the following scores:
  - Items 1,2,3,4, 6, and 7 are each scored as 1 if answered as as and 0 if answered as as a local.
  - Item 5 is scored as 1 if answered as [100] and 0 if answered as [100] (i.e., reversing the code response in a positive direction);

- Item 8 is scored as the value reported (0-4) divided by 4 (i.e., standardizing the 5-point Likert Scale for this item). For the purposes of summarising the n (%) of subjects with each score the standardized score will be rounded up in 0.5 will be rounded to 1.
- This results in a Total Score with a possible range of 0 to 8.0.
- 75% completion is necessary to calculate the score (ie 6 out of 8 questions need to be answered).
- If 1 or 2 items are missing, the median values of the other 7 or 8 items would be substituted for the missing item.





#### **Constipation Syndrome Score**

Mean value for items 10 (CCI ), 13 (CCI ), 15 (CCI )

This domain score can be computed if at least 2 out of 3 items are available (i.e. less than 50% of the item scores within a dimension are missing); in which case, the missing items will be imputed using the mean score of the non-missing item scores.

#### Abdominal Pain Syndrome Score

- Mean value for items 1 (CCI), 4 (CCI)

  ), 5 (CCI)

  )
- This domain score can be computed if at least 2 out of 3 items are available (i.e. less than 50% of the item scores within a dimension are missing); in which case, the missing items will be imputed using the mean score of the non-missing item scores.

#### Reflux Syndrome Score

- Mean value for items 2 (CCI), 3 (CCI)
- This domain score can be computed if at least 1 out of 2 items are available (i.e. less than 50% of the item scores within a dimension are missing); in which case, the missing items will be imputed using the mean score of the non-missing item scores.

# 11.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

## 11.7.1. **Premature Withdrawals**

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as: <ul> <li>Randomised to LPV/RTV + two NRTIs and completed the Randomised Phase including the Week 52 study visit;</li> <li>Randomised to DTG + two NRTIs, completed the Randomised Phase including the Week 52 study visit, and did not enter the Continuation Phase;</li> <li>Randomised to DTG + two NRTIs, completed the Randomised Phase, including the Week 52 study visit, entered and completed the Continuation Phase (defined as remaining on study until commercial supplies of DTG become locally available to patients [e.g. through public health services]).</li> </ul> </li> <li>Withdrawn subjects were not replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed.</li> </ul> |

# 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument :</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded</li> </ul> |
| | from the table. o Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Health<br>Outcome | See Section 11.6.7. |

# 11.7.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Section 11.4.</li> <li>Missing Stop Day: Last day of the month will be used ( '28/29/30/31' dependent on the month and year), unless this is after the stop date of study treatment; in the per scale the study treatment stop date will be used.</li> </ul> </li> </ul> |
| | <ul> <li>Completely missing start or end dates will remain missing, with no<br/>imputation applied. Consequently, time to onset and duration of such<br/>events will be missing.</li> </ul> |
| Prior/Concomitant<br>Medications | <ul> <li>Partial dates for any prior/concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>For medications recorded in the eCRF as prior ART, the earlier of this imputed date or the day before IP start will be used.</li> <li>The recorded partial date will be displayed in listings.</li> <li>Handling of completely missing start or end dates is discussed in Appendix 4: Treatment States and Phases.</li> </ul> |

# 11.7.2.2. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Snapshot<br>(MSDF) | <ul> <li>In the Snapshot dataset, subjects without HIV-1 RNA data in the assessment window for the visit of interest (due to missing data or discontinuation of IP prior to the visit window) are classified as non-responders in the derivation of the proportion of subjects with HIV-1 RNA &lt; 50 c/mL (or &lt;400 c/mL). The nature of this missing data will be further classified in Snapshot summaries as either 'Virologic Failure' or 'No Virologic Data at Week X'. Full details of the Snapshot algorithm are in Section 11.13.</li> <li>For the Week 48 deliverable, there will be 3 versions of the Snapshot dataset relative to the Primary Estimand and Additional Estimands 1 &amp; 2. For the Week 24 deliverable, there will only be one version of the dataset.</li> </ul> |
| LOCF | In the LOCF dataset, missing values will be carried forward from the previous, non-missing available on-treatment assessment. |
| НО | <ul> <li>Missing data in the Health Outcome questionnaires are described in Section<br/>11.6.7.</li> </ul> |
| Lipids LOCF | <ul> <li>If subjects initiate serum lipid-lowering agents Post-baseline, then the last available fasted On-treatment lipid values prior to the initiation will be used in place of future, observed On-treatment values.</li> <li>Imputation will continue even if the subject discontinues the lipid-lowering agent.</li> <li>Missing baseline assessments will not be imputed. Subjects on lipid-lowering agents at baseline will be excluded from this dataset.</li> <li>This dataset will be used for all summaries and analyses of lipids data</li> </ul> |

# 11.8. Appendix 8: Values of Potential Clinical Importance

| Element | Reporting Detail |
|---|---|
| Laboratory<br>Values and<br>Adverse | The DAIDS grading for severity of laboratory toxicities and clinical adverse events is included in the protocol. The part of the protocol. |
| Events | <ul> <li>The central laboratory will flag lab parameter toxicities directly in the provided<br/>datasets.</li> </ul> |

# 11.9. Appendix 9: Multicenter Studies

# 11.9.1. **Methods for Handling Centres**

Data will be summarised for all centres combined. Country will be treated as an exploratory subgroup for analyses of the primary efficacy endpoint as described in Section 7.1.2.

# 11.10. Appendix 10: Examination of Covariates, Subgroups & Other Strata

#### 11.10.1. Handling of Covariates, Subgroups & Other Strata

- The following is a list of covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses (See Section 7.1.2 and Section 9.1 for further details).
- Additional covariates of clinical interest may also be considered.
- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Category | Covariates and / or Subgroups |
|---|---|
| Randomization Strata using Baseline Values | <ul> <li>Baseline plasma HIV-1 RNA (≤ vs. &gt;100,000 c/mL);</li> <li>Number of fully active background NRTIs (&lt;2 vs. 2) based on GSS at Baseline.</li> </ul> |
| | For analysis purposes, randomization strata will be re-derived using Baseline values. In particular, fully active is defined at Baseline by the genotypic resistance reports of the central laboratory (or a laboratory contracted by the central laboratory) showing no evidence of full or of partial genotypic resistance for a given NRTI. If Baseline genotypic results are not available, then activity of the background regimen will be based on genotypic results at Screening. |
| | All statistical analyses will adjust for the above baseline randomization strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis Section 7.1 (primary endpoint) and Section 8.1 (secondary endpoint analyses) and Section 9.1 (health outcomes analyses). |
| Background Regimen and Resistance Subgroups | <ul> <li>WHO recommended public-heath approach second-line NRTI background regimen (yes vs. No ) (use definition in 11.6.3)</li> <li>Baseline PSS to background regimen: (&lt;2 vs. 2)</li> <li>Baseline GSS to background regimen: (&lt;2 vs. 2)</li> <li>ABC+3TC vs not ABC+3TC</li> </ul> |
| Demographic and Baseline<br>Characteristic Subgroups | <ul> <li>Age: &lt;35, 35-&lt;50, ≥50</li> <li>Race: <ul> <li>White; Non-White</li> <li>African American/African Heritage; Non-African</li> </ul> </li> </ul> |

| Category | Covariates and / or Subgroups |
|---|---|
| Category | American/African Heritage Sex: Female Male Country Baseline plasma HIV-1 RNA: <1000; 1000 to <10,000; 10,000 to <50,000; 50,000 to 100,000; >100,000 c/mL. <100,000; >100,000 c/mL. ≤100,000, >100,000 c/mL HIV-1 subtype: Subtype is found as part of the Monogram phenotype assay output. It is also known as clade eg, clade B = subtype B. Baseline CD4+ cell count: ≤Y cells/mm3 or >Y cells/mm3 (Y=cutoff closest to median); <200, 200-<350, ≥350 cells/mm3 Baseline Centers for Disease Control and Prevention (CDC) category: CDC Category A, |

# 11.11. Appendix 11: Handling of Multiple Comparisons & Multiplicity

A pre-specified fixed sequence testing procedure is used to control for multiplicity: if the primary comparison is significant for NI at the 5% two-sided alpha level then testing for superiority will proceed at the 5% two-sided alpha level; otherwise testing of superiority will not be performed.

The interim analysis schedule does not require an adjustment for multiplicity since the IDMC analyses do not inflate the type I error rate to any measurable degree (see protocol Section 8.3.4.2), and the Week 24 interim analysis is supportive to the primary Week 48 analysis and will not be used to make definitive claims of a positive finding.

# 11.12. Appendix 12: Model Checking and Diagnostics for Statistical Analyses

#### 11.12.1. Statistical Analysis Assumptions

# Endpoint(s) Change from Baseline in fasting LDL cholesterol at Weeks 24 and 48 Change from Baseline in fasting TC/HDL ratio at Weeks 24 and 48 HIV-Treatment Satisfaction Questionnaire (treatment satisfaction score) Gastrointestinal Symptom Rating Scale (Individual scores) Analysis

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### 11.13. Appendix 13: Snapshot

- Consider an arbitrary visit window, Week X (see Section 11.3).
- A subject's response (i.e., 'Virologic Success', 'Virologic Failure', or 'No Virologic Data at Week X') in that window is determined as indicated below, in the order stated.
- If non-permitted change in background ART prior to Week X: <u>Subject = Virologic Failure</u>.
- If permitted change in background ART prior to Week X AND decision to make this change is after the first On-treatment HIV-1 RNA result AND the latest On-treatment HIV-1 RNA result prior to the date of decision to switch is ≥ 50 c/mL: <u>Subject = Virologic Failure</u>.
- If non-permitted change in background ART during Week X

OR

if permitted change in background ART **during** Week X AND decision to make this change is *after* the first On-treatment HIV-1 RNA result AND the latest On-treatment HIV-1 RNA result prior to the date of decision to switch is >=50 c/mL

#### AND:

- no HIV-1 RNA result is available during Week X prior to change: <u>Subject = Virologic</u>
   Failure;
- there is at least one HIV-1 RNA result available during Week X prior to the change, then consider the latest such result:
  - If < 50 c/mL: Subject = Virologic Success</li>
  - If ≥ 50 c/mL: Subject = Virologic Failure.
- 4. If there is no change in background ART prior or during Week X

OR

a permitted change **prior or during** Week X is decided on *before* the first On-treatment HIV-1 RNA result,

OR

a permitted change **prior or during** Week X is decided on *after* the first On-treatment RNA result AND the latest On-treatment HIV-1 RNA result prior to the decision to switch is <50 c/mL,

AND

at least one HIV-1 RNA result is available during Week X, then consider the latest such result:

- If < 50 c/mL: Subject = Virologic Success;</li>
- If ≥ 50 c/mL: Subject = Virologic Failure.
- 5. If there is no change in background ART **prior or during** Week X

OR

a permitted change **prior or during** Week X is decided on *before* the first On-treatment HIV-1 RNA result

#### OR

a permitted change **prior or during** Week X is decided on *after* the first On-treatment RNA result AND the latest On-treatment HIV-1 RNA result prior to the decision to switch is <50 c/mL.

#### AND

no HIV-1 RNA results are available during Week X:

- If the subject has not withdrawn from the study prior to or during Week X: <u>Subject = No Virologic Data at Week X</u>, with a reason of 'Missing data during window but on study';
- If the subject was withdrawn from the study prior to or during Week X due to AE or death: <u>Subject = No Virologic Data at Week X</u>, with a reason of 'Discontinued due to AE or Death';
- Otherwise, consider the subject's last available On-treatment HIV-1 RNA result:
  - If <50 c/mL or no result is available: <u>Subject = No Virologic Data at Week X</u>, with a reason of 'Discontinued for Other Reasons';
  - If ≥ 50 c/mL: <u>Subject = Virologic Failure</u>.

#### **Examples from FDA guidance**

#### Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

 HIV-RNA = 580 copies/mL at Day 336, HIV-RNA below 50 copies/mL on Day 350. This should be categorized as HIV-RNA below 50 copies/mL.

#### No Data in Window

Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be
  classified as *Discontinued due to AE or Death* (as appropriate), regardless of the HIV-RNA
  result, even if the HIV-RNA is below 50 copies/mL at the time of discontinuation.
- However, if a patient has an HIV-RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response. This is the Virology First hierarchy:
  - a. HIV-RNA below 50 copies/mL at Day 336 and discontinues because of AE or even dies on Day 360 — this person is categorized as having HIV-RNA below 50 copies/mL.
  - b. HIV-RNA is 552 copies/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as having HIV-RNA greater than or equal to 50 copies/mL.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as Discontinued for Other Reasons.
- If a patient discontinues the study before the time window because of *lack of efficacy* then

- the patient should be included in the HIV-RNA greater than or equal to 50 row and not in the Discontinued for Other Reasons row.
- If a patient discontinues because of subject withdrew consent and his or her HIV-1 RNA
  result at the time of discontinuation was equal to or above 50 copies/mL, then he or she
  should be categorized as HIV-RNA greater than or equal to 50 and NOT as Discontinued
  for Other Reasons.
- If a patient discontinued because of *Lost to Follow-Up* and the last HIV-RNA result was 49 copies/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment not permitted by protocol— they should be considered an efficacy failure and captured in the HIV-RNA greater than or equal to 50 copies/mL row.

#### On study but missing data in window:

- If there are no data during Days 294 to 377, but there is an HIV-RNA below 50 copies/mL on Day 380, this patient should be considered *On Study but Missing Data in Window.*
- If there are no data during Days 294 to 377, but there is an HIV-RNA equal to or above 50 copies/mL on Day 280, this patient also should be classified as *On Study but Missing Data in Window.*

#### Optimized Background Therapy Substitutions After Randomisation

 OBT substitutions (in-class or cross-class) permitted per protocol for documented toxicity reasons can be permitted on or before the first trial visit without penalty.

If OBT substitutions for toxicity reasons occur after the first trial visit, then patients should be categorized as having HIV-RNA greater than or equal to 50 copies/mL if they have HIV-RNA above 50 copies/mL at the time of switch.

# 11.14. Appendix 14 – Q2 Creatinine Assay Accuracy Issue

## 11.14.1. Sensitivity Analyses

The machine at the central laboratory had debris in the system which led to suspect samples for creatinine. The impacted samples are indicated in the spreadsheet below.

Sensitivity analyses will be conducted excluding the suspect creatinine samples from any laboratory summaries. The details of the samples to be excluded are in the excel spreadsheet Suspect Creatinine Samples Study 200304 (Reference: RAP-Amend1-200304-Appendix 14.xls).

# 11.15. Appendix 15 – Abbreviations & Trade Marks

# 11.15.1. Abbreviations

| Abbreviation | Description |
|---|---|
| A&R | Analysis and Reporting |
| ABC | Abacavir |
| AdaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| ALT | Alanine aminotransferase |
| ART | Antiretroviral Treatment |
| ATC | Anatomical Therapeutic Chemical |
| ATV | Atazanavir |
| c/ml | Copies per milliliter |
| CD4+ | Helper-inducer T-lymphocyte having surface antigen CD4 (cluster of |
| | differentiation 4) |
| CDC | Centers for Disease Control and Prevention |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CMH | Cochran-Mantel-Haenszel |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTR | Clinical Trial Register |
| CV | Cardiovascular |
| CVWC | Confirmed Virologic Withdrawal Criteria |
| DAIDS | Division of AIDS |
| DBF | Database Freeze |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| ERDF | Efficacy Related Discontinuation = Failure |
| FC | Fold change |
| FDA | Food and Drug Agency |
| FDC | Fixed Dose Combination |
| FTC | Emtricitabine |
| FU | Follow-up |
| GFR | Glomerular Filtration Rate |
| GSK | GlaxoSmithKline |
| GSK | GlaxoSmithKline |
| GSRS | Gastrointestinal Symptom Rating Scale |
| GSS | Genotypic Susceptibility Score |
| GUI | Guidance |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| HDL | High density lipoprotein |
| HIV(-1) | Human immunodeficiency virus (type 1) |
| HIVTSQ | HIV Treatment Satisfaction Questionnaire |
| HSR | Hypersensitivity reaction |
| IA | Interim Analysis |
| IAS-USA | International Antiviral Society-USA |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | |
| | International Modules Management System |
| IN(I) | Integrase (Inhibitor) |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| ITT(e) | Intent-To-Treat Exposed |
| LDL | Low density lipoprotein |
| LOCF | Last Observation Carries Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMAS-8 | Morisky 8-Item Medication Adherence Scale |
| MMRM | Mixed Model Repeated Measures |
| NCEP | National Cholesterol Education Program |
| NNRTI | Non-nucleoside Reverse Transcript Inhibitor |
| NRTI | Nucleoside Reverse Transcript Inhibitor |
| OC | Observed Case |
| OSS | Optimised Susceptibility Scoring |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PI | Protease Inhibitor |
| PP | Per Protocol |
| PSRAE | Possibly suicidality related Adverse Event |
| PSS | Phenotypic Susceptibility Score |
| QC | Quality Control |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAMOS | Randomization & Medication Ordering System |
| RAP | Reporting & Analysis Plan |
| RNA | Ribonucleic acid |
| RTV | Ritonavir |
| RUCAM | Roussel Uclaf Causality Assessment Method |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis Software |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| | Sjotem Organ Class |

| Abbreviation | Description |
|--------------|---------------------------------------------|
| SOP | Standard Operation Procedure |
| SVW | Suspected Virologic Withdrawal |
| TA | Therapeutic Area |
| TC | Total Cholesterol |
| TDF/FTC | Tenofovir/emtricitabine |
| TFL | Tables, Figures & Listings |
| TRDF | Treatment Related Discontinuation = Failure |
| VF | Virologic Failure |
| WHO | World Health Organisation |

# 11.15.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| DOLUTEGRAVIR |
| EPZICOM/KIVEXA |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Monogram Biosciences |
| Norvir |
| Quest Diagnostics |
| Reyataz |
| SAS |
| Truvada |
| TSCG |
| TYLENOL |

## 11.16. Appendix 16 – Example SAS code for Additional Estimand 2

```
*Presented below are excerpts of code that can be used for the multiple
imputation steps for the Additional Estimand 2 methodology for the
Primary Efficacy Endpoint at Week 48;
*The code has not been extensively QC'ed therefore care must be taken
when implementing;
*Programming Steps:
[1] Select LOG HIV-1 RNA data from ADLB
[2] Subset data by Treatment group
[3] Multiple Imputation on the Continuous scale
[3a] For LPV/RTV arm: run a simulation replacing BLQ with values from
U(0,BLQ) distribution;
* 100 simulated datasets;
data step3a ;
 set step3a ;
 do i=1 to 100;
   if substr(LBSTRESC,1,1)="<" then aval2 = rand('uniform')*1.59;
                   *i.e. 1.59 is slightly below log(50) hence BLQ;
   else aval2=aval;
      imputation = i;
     output;
 end;
 drop i;
run;
*Programming steps continued:
[3b] Transpose datasets LPV/RTV & DTG datasets ready for MI
[3c] For LPV/RTV subjects, PROC MI to create Monotone structure;
*** Note: AVAL1 = Week 1 (baseline), to AVAL52 (Week 52);
*** Programming Note: add stratification factors;
proc mi data=step3c out=DATAIN MONO nimpute=1 seed=200304;
   by imputation;
     var AVAL1 AVAL4 AVAL8 AVAL16 AVAL24 AVAL36 AVAL48 AVAL52;
     mcmc impute=monotone;
run;
*Programming steps continued:
[3d] Impute the remaining monotone missing values
*** Assumption: MAR;
data DATAIN MONO (rename=( Imputation =Imputation));
 set DATAIN MONO ;
run;
*** Programming Note: add stratification factors;
proc mi data= DATAIN MONO out= DATAIN REG nimpute=1 seed=200304;
     by Imputation;
     var AVAL1 AVAL4 AVAL8 AVAL16 AVAL24 AVAL36 AVAL48 AVAL52;
     monotone regression;
run:
```

```
data DATAIN REG;
 set DATAIN REG;
 rename Imputation = impute ;
run;
*Programming steps continued:
[4] Merge DTG to LPV/RTV imputed dataset. For DTG dataset, create
duplicate rows (=number of imputed datasets)
data step4dtg;
 set step4dtg;
  impute =1;
  do _impute_= 1 to 100;
 output;
 end;
run;
*Programming steps continued:
[5a] Remove non-IDMC affected subjects from LPV/RTV imputed dataset.
[5b] Merge original data of non-IDMC LPV/RTV subjects LPV/RTV imputed,
replacing imputed data for these subjects with original observations.
Do so by creating duplicate rows (=number of imputed datasets)
[6] apply Snapshot algorithm
[7a] Perform CMH test & obtain Mantel-Haenszel estimate of the common
odds ratio & P-value;
*programming note: need to add stratification factors;
*take care when specifying tables statement;
proc freq data=step7;
 tables trt01p * snapresp /cmh riskdiff measures;
 by impute ;
 ODS OUTPUT CMH=cmh COMMONRELRISKS=comrrout CrossTabFreqs = Freqout
measures=measures est riskdiffcol1=riskdiff est;
RUN:
data Prop (keep= p SEp TREAT impute );
 set riskdiff est ;
 p=1-risk;
 SEp=ase;
  if Row in("Row 1", "Row 2");
      if Row="Row 1" then TREAT="DTG
  else if Row="Row 2" then TREAT="LPV/RTV";
run;
proc sort data=PROP;
 by TREAT ;
run;
*Programming steps continued:
[7b] Combine results;
PROC MIANALYZE DATA=prop ;
 modeleffects p ;
  stderr SEp;
 by TREAT ;
RUN;
```

```
*Programming steps continued:
[7c] for the P-value, apply Wilson-Hilferty transformation to the CMH
statistic and standardize the resulting normal variable;
DATA cmh wh;
 SET cmh(WHERE=(AltHypothesis="General Association"));
  cmh value wh=((VALUE/DF)**(1/3) - (1-2/(9*DF)))/SQRT(2/(9*DF));
  cmh sterr wh = 1.0;
RUN;
*Programming steps continued:
[7d] Combine results;
PROC MIANALYZE DATA=cmh wh;
 ODS OUTPUT PARAMETERESTIMATES=mian cmh wh;
 MODELEFFECTS cmh value wh;
 STDERR cmh sterr wh;
RUN;
*Programming steps continued:
[7e] Compute one-sided p-value;
DATA mian_cmh_wh_p;
 SET mian cmh wh;
 IF tValue > 0 THEN Probt upper = Probt/2;
 ELSE Probt upper = 1-Probt/2;
RUN;
```

## 11.17. Appendix 17 – End of Study Analysis

This appendix will provide the details of planned analyses and data displays for MID200304 End of Study (EoS) reporting. These analyses may be included for disclosure purposes.

#### 11.17.1. General considerations for data analyses

This section is written specifically for the EoS analysis. Since the primary analyses have been completed, the present section is written to cover only analyses included in the final EoS reporting. Only those definitions and derivations that have changed since the previous interim analyses will be included in this section, i.e., for the derivation of analysis windowing, how to deal with missing dates, definition of concomitant medications, etc. refer to the previous corresponding RAP sections. The current section summarises only the key endpoints of interest for the final analysis and explains any deviations from the previous analysis.

The details of the final EoS reporting and analysis are described below:

- The analyses for which the data have not been changed since the primary (Week 48/52) analysis will not be reported again to avoid redundancy. This includes the analyses of demographic, baseline characteristics and health outcomes.
- 2) No subgroup analysis, hypotheses testing, or statistical analyses will be performed.
- All required disclosure outputs following the FDAAA and EudraCT guidelines will be produced.

#### 11.17.1.1. Study Phases

In the previous analysis (primary Week 48 reporting), data were summarised for the Randomised Phase of the study. However, when data from the Continuation Phase were available, certain displays were repeated for the combined period of Randomised plus Continuation Phases. For the EoS reporting, data from both study phases (Randomised Phase plus Continuation Phase) will be tabulated in one summary table, unless specified otherwise, and this will be noted in the title of the output. Listings will contain all the data with a new column added to specify the phase of the study for each record. Randomised and Continuation Phases are defined as below:

| Phase | Start | End |
|---|---|---|
| Randomised Phase | IP start date | Non-switch participants: Week 52 DOV, IP end date or Withdrawal date if on or before Week 52 DOV; Switch participants: last LTV/RPV treatment date. |
| Continuation Phase | Non-switch participants: | IP end date or Withdrawal |

| Phase | Start | End |
|-------|---------------------------|--------------------------|
| | Week 52 DOV+1 day; | date if post Week 52 DOV |
| | Switch participants: last | |
| | LTV/RPV treatment date+1 | |
| | day. | |

Note: Switch participants are participants that switched from LPV/RTV to DTG treatment between Week 48 and Week 52 visits (Please see Section 11.17.1.3).

Note: A participant enters the Continuation Phase if they have at least one exposure to the Investigational Product after the end of Randomisation Phase.

# 11.17.1.2. Analysis Population for the Continuation Phase

In addition to the populations defined in Section 4 of the RAP amendment 2, the following populations were defined for the End of Study Analysis:

| Population | Definition/ Criteria. | Analysis Evaluated |
|---|---|---|
| Safety Continuation | Comprises all participants in the Safety Population who receive at least one dose of Investigational Product after entering the Continuation Phase. | • Safety |
| Intent-to-Treat Exposed (ITT-E) Continuation | Comprises all participants in the ITT-E Population who continue into the Continuation Phase. | <ul><li>Efficacy</li><li>Study Population</li></ul> |
| Viral Genotypic | Comprises all participants in the ITT-E Population with available ontreatment genotypic resistance data. | Genotypic |
| Viral Genotypic Continuation | Comprises all participants in the ITT-E- Continuation Population with available on-treatment genotypic resistance data in the Continuation Phase. | Genotypic |
| Viral Phenotypic | Comprises all participants in the ITT-E Population with available ontreatment phenotypic resistance data. | Phenotypic |
| Viral Phenotypic Continuation | Comprises all participants in the ITT-E- Continuation Population with available on-treatment phenotypic resistance data in the Continuation Phase. | Phenotypic |

# 11.17.1.3. Participants that Switched from LPV/RTV to DTG Treatment ("Switch participants")

Following the IDMC's recommendation and as per Protocol Amendment No. 2, there are two instances where participants continue to have access to DTG in the Continuation Phase. One is that participants randomised to receive DTG who successfully complete 52 weeks of treatment, the other is that participants originally randomised to receive LPV/RTV but switched to DTG prior to or at Week 52. Treatment arm "Switch from LPV/RTV to DTG" is added for switch treatment participants in the Continuation Phase.

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Data Displays for F | | Data Displays for Reporti | porting |
| Code | Description | Description | Order [1] |
| Α | Dolutegravir 50mg once daily | DTG | 1 |
| В | Lopinavir/ritonavir 800mg/200mg<br>once daily or 400mg/100mg twice<br>daily | LPV/RTV | 2 |
| B/A | Lopinavir/ritonavir 800mg/200mg<br>once daily or 400mg/100mg twice<br>daily / Dolutegravir 50mg once daily | Switch from LPV/RTV to DTG | 3 |

#### NOTES:

Order represents treatments being presented in TFL, as appropriate.

For EoS reporting, detailed information for both DTG and switch participants are included in the corresponding listings. Summary statistics are done according to below:

Two treatment arms are to be reported for summary tables that cover both Randomization Phase and Continuation Phase, one for DTG and the other for LPV/RTV. For Safety summary tables, only data before the switch date are to be included for the switch participants in the LPV/RTV arm. A footnote, "Data on or after the switch date are not included for participants who switched from LPV/RTV to DTG", will be added for these tables. For Efficacy or Study Population summary tables, all data for the LPV/RTV arm will be included for the table, no matter whether the participants switched treatment to DTG or not.

For summary tables that only cover Continuation Phase, the switch participants are included in the table as a separate arm. Data are summarised for DTG treatment group, Switch treatment group and Total.

#### 11.17.1.4. Decision tree for Monogram resistance data analyses

#### **Decision tree for Monogram resistance data analyses**

- We might have resistance data that come from mixed datasets: PSGT, PSIN, GSIN (primary assays)
   vs PSGT+IN (secondary assay)
- If one of the primary assay does not work for a specific timepoint, we might report the secondary assay if data is available. If all primary assays for a specific timepoint work then we report primary. For example, for baseline if the same assay section (PSGT, PSIN, GSIN) worked then we report. If at least one of PSGT or PSIN or GSIN didn't work then we report secondary PSGT+IN.
- Secondary assay testing results might not always be available.
- For examples please refer to decision tree below.

#### **Background:**

- PSGT provides both geno and pheno data for PRO/RT (NRTI and NNRTI) only
- PSIN Provides pheno data on Integrase only
- GSIN Provides geno data on Integrase only
- PSGT+IN Secondary assay used if PSGT or GSIN assay fails; it provides both geno and pheno data on PRO, RT and Integrase

#### **Table Symbol Key:**

y = assay test successful n = assay test failure 2<sup>nd</sup> = back up test performed **bold** = assay to use for analysis

#### How to make decisions:

<u>Scenario 1</u>: if primary PSGT, PSIN and GSIN assays all work) for both baseline and CVW samples, then PSGT+IN assay will not be performed, no PSGT+IN data should be generated.

| Assays | Baseline | CVW |
|--------|----------|-----|
| PSGT | у | у |
| PSIN | у | у |
| GSIN | у | у |

Scenario 2: If PSGT works for baseline, but PSIN and GSIN fail, then secondary PSGT+IN assay will be performed on baseline sample; similarly, if PSGT works for CVW sample but PSIN and GSIN fail to work, in this scenario, use data generated from PSGT+IN assay on both Baseline and CVW sample for analyses, regardless of obtained PSGT assay data.

| Assays Baseline CVW |
|---------------------|
|---------------------|

| PSGT | у | у |
|-------------------------|---|---|
| PSIN | n | n |
| GSIN | n | n |
| 2 <sup>nd</sup> PSGT+IN | Υ | Υ |

Scenario 3: If PSGT, PSIN and GSIN all work for baseline samples; PSGT works for CVW but PSIN and GSIN fail, while PSGT+IN on CVW sample works, then use CVW PSGT+IN (PR, RT and INSTI) to do comparison with PSGT, PSIN and GSIN baseline data (do not use PSGT at CVW data vs. PSGT at Baseline)

| Assays | Baseline | CVW |
|-------------------------|----------|-----|
| PSGT | у | у |
| PSIN | у | n |
| GSIN | у | n |
| 2 <sup>nd</sup> PSGT+IN | - | Υ |

Scenario 4: If PSGT works but GSIN and PSIN both fail on baseline sample, then secondary PSGT+IN assay might be performed. And if PSGT, PSIN and GSIN all work for CVW sample, then use Baseline PSGT+IN data to do comparison with CVW Primary assay data, regardless of PSGT Baseline data. In other words, don't use PSGT Baseline to do comparison of PSGT part of PSGT+IN assay data for CVW sample

| Assays | Baseline | CVW |
|-------------------------|----------|-----|
| PSGT | у | у |
| PSIN | n | У |
| GSIN | n | у |
| 2 <sup>nd</sup> PSGT+IN | Υ | - |

#### 11.17.2. Study Population

The study population summaries and data listings will be based on the ITT-E or ITT-E Continuation Population, unless otherwise specified. Demographic and baseline characteristics will not be reported in EoS. Participant accountability summary will be produced for the overall study and separately for the Continuation Phase.

Overview of the key planned study population endpoints:

- Study Populations
- Participant Accountability
- Concomitant and Antiretroviral Medications.
- Protocol deviation.

Full details of the data displays are given in Section 11.17.7.1.

#### 11.17.3. Efficacy Analysis

The study efficacy summaries and data listings will be based on the ITT-E Population except for Table 2.16. Table 2.16 summarises plasma HIV-1 RNA results for participants meeting CVW criteria during the Continuation Phase and is based on the ITT-E Continuation Population.

Overview of the key planned efficacy endpoints:

- Proportion of Participants with Plasma HIV-1 RNA < 50 c/ mL Observed Data
- Proportion of Participants with Confirmed Virologic Withdrawal (observed data)
- Change from baseline CD4+ cell count over time
- Incidence of disease progression and HIV-associated conditions

Full details of data displays are given in Section 11.17.7.2.

#### 11.17.4. Safety Analysis

All safety displays will be based on the Safety Population or the Safety Continuation Population.

The core adverse event displays for the final report have been identified based on the IDSL library required tables. For the purposes of summarising the AE data, unless stated otherwise, the summaries will include only those AEs that occurred during the Continuation Phase. Common AEs are those with 2% (without rounding) incidence for any treatment.

Summaries of AEs required for the FDAAA and EudraCT will be generated in this report. These summaries will include participants from both the Randomised and Continuation Phases. Common and/or serious AEs will be summarized for the Continuation Phase. SAEs and non-SAEs will be listed for Mexican participants only.

Summaries of Maximum Post-Baseline Grade 3 or 4 Emergent Clinical Toxicities and Hepatobiliary Abnormality criteria will be reported only for the events that occurred during the Continuation Phase.

A new figure of cumulative exposure showing the number of participants exposed to DTG and LPV/RTV over time will be added for EoS reporting. Missing Treatment stop date will be imputed as the last day of month or year if partial dates, the date of last visit or the recorded date of withdrawal/completion, whichever is earlier.

Overview of the key planned safety endpoints:

- Extent of Exposure
- Adverse Events
- Maximum Post-Baseline Emergent Clinical Chemistry/ Haematology Toxicities

- Hepatobiliary Laboratory Abnormality Criteria
- Liver Events Assessment
- Columbia Suicide Severity Rating Scale (C-SSRS)

Full details of data displays are given in Section 11.17.7.3.

#### 11.17.5. Virology analysis

The virology summaries will be based on the Viral Genotypic and Viral Phenotypic Continuation Populations, unless otherwise specified. Data listings will be presented for the ITT-E Population, unless otherwise specified.

Virology summaries will focus on the Continuation Phase and be tabulated only for participants in the Viral Genotypic or Genotypic Continuation Population except table 4.2 and 4.3. Table 4.2 and 4.3 summarises emergent major mutations during Randomised Phase and is based on Viral Genotypic Population. Emergent Major Mutations of NRTI, NNRTI and PI Classes and Emergent Prespecified INSTI mutations are summarised both for the Randomised and the Continuation Phases in separate Tables.

Prespecified lists of integrase substitutions have been modified since the previous interim analysis, hence an updated list of known INSTI mutations has been added in **** and IAS-USA major r esistance associated mutations (RAMs) to other classes (i.e., NRTI, NNRTI, PI) are listed in **** 

Table 13 Known INSTI mutations associated with the development of resistance to RAL, EVG or DTG

| Amino Acids | H51Y, <u>T66A/I/K</u> , L74M, <u>E92Q/V</u> /G, Q95K, T97A, G118R, |
|---|---|
| in HIV | <b>F121Y</b> , E138A/K, G140A/C/S, <b>Y143C/H/R/K/S/G/A</b> , <b>P145S</b> , |
| Integrase for | Q146P, S147G, Q148N/H/K/R, V151I/L/A, S153F/Y, |
| Analysis | N155H/S/T, E157Q, G163R/K, S230R, R263K, L68V/I*, L74I*, |
| | E138T*, G193E* |

#### NOTES:

- Current listing includes INSTI mutations identified via the Stanford HIV Resistance database, or identified during in vitro passage of DTG, or as seen in a previous DTG studies in INSTI-experienced participants (i.e. ING112574) and may be modified in case of additional substantive data availability.
- INSTI mutations in bold have the maximum score of 60 and are for any INSTI drug in the Stanford database v8.9 (http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INSTI last updated on 25 OCT 2019 and accessed on 17 FEB 2020); the rest have a maximum score <60.
- The INSTI mutations listed are historically identified via the Stanford HIV Resistance database, and also include mutations identified during in vitro passage of DTG, or as seen in a previous DTG study in INI-experienced participants (ING112574).
- This table is updated only by Virologists.

Table 14 Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA).

| Class | Mutations |
|---|---|
| NRTIs | M41L, K65R/E/N, D67N, 69 insert, K70E/R, L74V, Y115F, M184V/I, L210W, T215Y/F, K219Q/E; [A62V, V75I, F77L, F116Y, Q151M] |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138A/G/K/Q/R, V179L,Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L |
| Pls | D30N,V32I , M46I/L, I47A/V, G48V, I50V/L, I54V/M/L, Q58E, T74P, L76V, V82A/T/F/L/S, N83D, I84V, N88S, L90M |

#### NOTES:

- Updated to "2019 Resistance Mutations Update Volume 27 Issue 3, July/August 2019
- The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis.
- Q151M Complex: Q151M usually occurs in combination with two or more of the following four accessory NRTI mutations A62V, V75I, F77L, and F116Y However if any one of these mutations occur alone, they shall be considered as major mutation for the NRTI class.

Clinical and Biological Cut-off Values for the PhenoSense HIV Drug Resistance Assay have changed since the previous interim analysis, hence for EoS phenotypic susceptibility will be categorised according to Fold Change as shown in Table 15 (based on Monogram PhenoSense assay).

Table 15 Clinical and Biological Cutoff Values for the PhenoSense HIV Drug Resistance Assay

| Drug | Abbreviation | Class | PhenoSense |
|-----------------|--------------|-------|-----------------------|
| | | | Cutoff |
| Abacavir | ABC | NRTI | $(4.5 - 6.5)^a$ |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 <sup>a</sup> |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF | NRTI | $(1.4-4)^a$ |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivirine | RPV | NNRTI | 2.5 |
| Fosamprenavir | FPV | PI | 2 a,c |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir | ATV | PI | 2.2 a, |
| Atazanavir/r | ATV/r | PI | 5.2 a,c |
| Indinavir/r | IDV/r | PI | 10 <sup>a</sup> |
| Lopinavir/r | LPV/r | PI | (9 – 55) <sup>a</sup> |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir | SQV | PI | 1.7 a,c |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 <sup>b</sup> |
| Raltegravir | RAL | INSTI | 1.5 |
| Elvitegravir | EVG | INSTI | 2.5 |
| Dolutegravir | DTG | INSTI | (4-13) a |

a: clinical cutoff (lower cutoff – higher cutoff)

#### Overview of the key planned virology endpoints:

- Genotypic and Phenotypic Accountability
- INSTI mutations
- Major NRTI, NNRTI, PI mutations
- Fold Change to DTG

b: standard cut-off used by Monogram Inc. until clinical or biological cutoff have been determined

c: Only the boosted cutoff shall be used to compute the PhenoSense sensitivity for Atazanavir, Fosamprenavir and Saquinavir except stated otherwise.

Full details of data displays are given in Section 2.7.4.

#### 11.17.6. **COVID - 19 analysis**

This study started in 2014 and continued during the COVID -19 pandemic. The information regarding the number of participants affected by COVID-19 and its symptoms will be reported according to GSK core standards. The visits impacted due to the pandemic outbreak will be reported. Protocol deviations or adverse events related to COVID-19 if any, will also be reported according to GSK core standards.
# 11.17.7. **Data Displays for End of Study Final Report**

• Outputs that were not reported at Week 48 reporting are identified in Programming Notes as 'New output'

## 11.17.7.1. Study Population

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Table | 1.1 | All Participants Screened | Summary of Study Populations | |
| Table | 1.2 | ITT-E | Summary of Number of Participants by Study Visit | New output (refer to the template provided) |
| Table | 1.5 | ITT-E | Summary of Participant Accountability: Study<br>Conclusion Record by Relationship to COVID-19<br>Pandemic | FDAAA, EudraCT<br>Have an overall and then split by<br>COVID-19 relationship |
| Table | 1.7 | ITT-E Continuation | Summary of Participant Accountability: Continuation Phase Conclusion Record by Relationship to COVID-19 Pandemic | Have an overall and then split by COVID-19 relationship |
| Table | 1.10 | ITT-E | Summary of Important Protocol Deviations by Relationship to COVID-19 Pandemic | Have an overall and then split by COVID-19 relationship |
| Table | 1.26 | ITT-E | Summary of Concomitant Medication by ATC Level 1 and Ingredient | Only non-ART medications |
| Listing - ICH | 4 | ITT-E | Listing of Study Conclusions Reasons for Study Withdrawal | |

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Listing - ICH | 8 | ITT-E | Listing of Important Protocol Deviations | |
| Listing - Other | 29 | All Participants Screened | Listing of Study Populations | |
| Listing - Other | 31 | ITT-E | Listing of Visit Dates | |
| Listing - Other | 38 | ITT-E | Listing of Concomitant Medications | |
| Listing - Other | 39 | ITT-E | Listing of Relationship Between ATC Level 1, Ingredient and Verbatim Text | |
| Listing - Other | 41 | ITT-E | Listing of Concomitant and Post-treatment<br>Antiretroviral Therapy | |
| Listing - Other | 43 | ITT-E | Listing of Relationship Between ATC Level 4, Ingredient and Verbatim Text for ART | |
| Listing - Other | 79 | ITT-E | All Non-Important COVID-19 Related Protocol Deviations | New output (refer to Sailing EoS L.41) |

No figures for the Study Population.

# 11.17.7.2. Efficacy

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Table | 2.8 | ITT-E | Summary of Proportion of Participants with Plasma<br>HIV-1 RNA <50 c/mL by Visit -Observed Data | Observed data calculates proportions using denominator of subjects with HIV RNA readings at visit week |
| Table | 2.15 | ITT-E | Proportion of Participants Meeting CVW Criteria by Visit by Type of Virologic Failure -Observed Data | Proportion instead of 'Cumulative Proportion' comparing to w48 RE. Observed data calculates proportions using denominator of subjects with HIV RNA readings at visit week |
| Table | 2.16 | ITT-E Continuation | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Virologic Withdrawal Criteria for Participants with CVW During the Continuation Phase | |
| Table | 2.19 | ITT-E | Summary of Post-Baseline HIV-1 Associated Conditions Including Recurrences | |
| Table | 2.20 | ITT-E | Summary of Post-Baseline HIV-1 Associated Conditions Excluding Recurrences | |
| Table | 2.21 | ITT-E | Summary of Post-Baseline HIV-1 Disease Progressions | |

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Table | 2.22 | ITT-E | Summary of Change from Baseline in CD4+ Cell Count (cells/mm^3) by Visit | |
| Table | 2.23 | ITT-E | Summary of Change from Baseline in Plasma HIV-1 RNA (log10 c/mL) by Visit | |
| Listing - ICH | 12 | ITT-E | Listing of Quantitative Plasma HIV-1 RNA Data | |
| Listing - Other | 44 | ITT-E | Listing of CD4+ Cell Count Data | |
| Listing - Other | 45 | ITT-E | Listing of HIV-1 Associated Conditions | |
| Listing - Other | 47 | ITT-E | Listing of Viral Load over time for Participants with CVW Criteria | W48 RE only reported participants with CVW during continuation phase. Here please report all participants with CVW and group by phase. |
| Figure | 2.8 | ITT-E | Individual Plasma HIV-1 RNA and CD4+ Profiles by Visit for Participants with at least One Suspected Virologic Withdrawal Criteria Met | Please use title and shell from F2.3 gsk3515864/mid204861/primary_15 |

# 11.17.7.3. Safety

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Table | 3.1 | Safety Continuation | Summary of Extent of Exposure to Investigational Product for Participants who Entered Continuation Phase | |
| Table | 3.2 | Safety | Summary of Extent of Exposure to Investigational Product for All Participants in Randomised and Continuation Phase | |
| Table | 3.5 | Safety Continuation | Summary of All Adverse Events by System Organ Class, Preferred Term and Maximum Toxicity - Continuation Phase | |
| Table | 3.6 | Safety Continuation | Summary of Common (>=2%) Adverse Events by Preferred Term and Overall Frequency - Continuation Phase | Common adverse events are those with >=2% (with rounding) incidence for any treatment. |
| Table | 3.7 | Safety Continuation | Summary of Common (>=2%) Grade 2-4 Adverse<br>Events by Preferred Term and Overall Frequency -<br>Continuation Phase | Common adverse events are those with >=2% (with rounding) incidence for any treatment. |
| Table | 3.9 | Safety Continuation | Summary of All Drug-related Adverse Events by<br>System Organ Class, Preferred Term and Maximum<br>Toxicity - Continuation Phase | |

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Table | 3.11 | Safety Continuation | Summary of Common (>=2%) Drug-related Grade 2-4<br>Adverse Events by Overall Frequency - Continuation<br>Phase | Common adverse events are those with >=2% (with rounding) incidence for any treatment. |
| Table | 3.13 | Safety Continuation | Summary of Serious Adverse Events by System Organ Class and Preferred Term - Continuation Phase | |
| Table | 3.18 | Safety Continuation | Summary of Adverse Events Leading to<br>Withdrawal/Permanent Discontinuation of Study<br>Treatment by System Organ Class and Preferred<br>Term - Continuation Phase | |
| Table | 3.20 | Safety | Summary of Participants and Number of Occurrences of Common (>= 2%) Non-Serious Adverse Events by System Organ Class and Preferred Term - Randomised and Continuation Phases | FDAAA, EudraCT Common adverse events are those with >=2% (without rounding) incidence for any treatment. |
| Table | 3.21 | Safety | Summary of Participants and Number of Occurrences of Serious Adverse Events by System Organ Class and Preferred Term - Randomised and Continuation Phases | FDAAA, EudraCT |
| Table | 3.22 | Safety | Summary of COVID-19 Assessment for Participants with COVID-19 Adverse Events | New output. Please refer to Sailing<br>EoS T8.26 |

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Table | 3.23 | Safety | Summary of COVID-19 Symptoms for Participants with COVID-19 Adverse Events | New output. Please refer to Sailing EoS T8.27 |
| Table | 3.36 | Safety Continuation | Summary of Maximum Post-Baseline Emergent<br>Clinical Chemistry Toxicities - Continuation Phase | |
| Table | 3.38 | Safety Continuation | Summary of Maximum Post-Baseline Emergent<br>Hematology Toxicities - Continuation Phase | |
| Table | 3.45 | Safety Continuation | Summary of Participants Meeting Hepatobiliary<br>Laboratory Abnormality Criteria - Post-Baseline<br>Emergent - Continuation Phase | Abbreviated (see template provided) |
| Table | 3.48 | Safety | Summary of Participants with C-SSRS Suicidal Ideation or Behaviour during Treatment | |
| Listing - ICH | 15 | Safety | Listing of Investigational Product Exposure Data | Star * Switch participant and add footnote |
| Listing - ICH | 18 | Safety | Listing of All Adverse Events | Star * Switch participant and add footnote |
| Listing - ICH | 21 | Safety | Listing of Fatal Serious Adverse Events | |
| Listing - ICH | 22 | Safety | Listing of Non-Fatal Serious Adverse Events | |

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Listing - ICH | 23 | Safety | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Study Treatment | |
| Listing - ICH | 24 | Safety | Listing of Relationship of Adverse Event System<br>Organ Class, Preferred Terms and Verbatim Text | |
| Listing - Other | 25 | Safety | Listing of Non-Serious AEs of Mexican Participants | New output |
| Listing - Other | 26 | Safety | Listing of SAEs of Mexican Participants | New output |
| Listing - Other | 27 | Safety | Listing of SAEs of Non-Mexican Participants | New output |
| Listing-Other | 28 | Safety | Listing of COVID-19 Assessments and Symptoms | New output |
| Listing - Other | 53 | Safety | Listing of Participants Who Became Pregnant During the Study | |
| Listing - Other | 56 | Safety | Listing of Laboratory Data for Participants with Grade 3 or 4 Post-Baseline Emergent Toxicities | |
| Listing - Other | 57 | Safety Continuation | Listing of Post Baseline Maximum ALT and Maximum Bilirubin – Continuation Phase | New output (Please refer to Sailing EoS L.30) |
| Listing - Other | 58 | Safety Continuation | Listing of Participants Meeting Hepatobiliary<br>Laboratory Criteria -Continuation Phase | |

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Listing - Other | 59 | Safety | Listing of Liver Monitoring/Stopping Event Reporting | |
| Listing - Other | 86 | Safety | Listing of Start and Stop Dates in the<br>Continuation Phase | New output. Please refer to Listing 86 in Aria |
| Listing - Other | 93 | Safety | Listing of C-SSRS Suicidal Ideation and<br>Behaviour Data | |
| Figure | 3.5 | Safety Continuation | Scatter Plot of Maximum Post-Baseline ALT vs. Maximum Post-Baseline Total Bilirubin - Continuation Phase | |
| Figure | 3.6 | Safety | Plot of Cumulative Exposure to Investigational Product | Please refer to Sailing EoS F8.27 For switch subjects, only data before the switch date will be plotted |

# Virology

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Table | 4.1 | Viral Genotypic<br>Continuation | Summary of Participant Accountability: Genotypes<br>Available - Continuation phase | |
| Table | 4.2 | Viral Genotypic | Summary of Emergent Major Mutations of NRTI,<br>NNRTI and PI Classes for Participants with CVW -<br>Randomised Phase | |
| Table | 4.201 | Viral Genotypic<br>Continuation | Summary of Emergent Major Mutations of NRTI,<br>NNRTI and PI Classes for Participants with CVW -<br>Continuation phase | |
| Table | 4.3 | Viral Genotypic | Summary of Pre-specified Treatment Emergent INSTI<br>Substitutions at Time of Confirmed<br>Virologic Withdrawal - Randomised Phase | |
| Table | 4.301 | Viral Genotypic<br>Continuation | Summary of Pre-specified Treatment Emergent INSTI Substitutions at Time of Confirmed Virologic Withdrawal - Continuation Phase | |
| Table | 4.5 | Viral Phenotypic<br>Continuation | Summary of Participant Accountability: Phenotype Available - Continuation phase | |
| Table | 4.8 | Viral Phenotypic<br>Continuation | Summary of Fold Change to DTG at Baseline and Time of CVW - Continuation Phase | |
| Listing Other | 77 | ITT-E | Listing of All Genotypic Data | |

| Туре | Display<br>Number | Population | Display Title | Programming Notes |
|---|---|---|---|---|
| Listing Other | 78 | ITT-E | Listing of All Phenotypic Data | |
| Listing Other | 80 | ITT-E | Listing of Virology Data for Participants with CVW | Please follow SAILING EoS L.37 format |
| Listing Other | 82 | ITT-E | Listing of Virology Data for Participants with On-<br>Treatment Virology Results at Non-CVW timepoints | Please follow SAILING EoS L.38 format |
| Listing Other | 83 | ITT-E | Participant Level Summary of Key Virologic Data of Background Regimens for Participants with On-Treatment Virology Results at CVW timepoints | |
| Listing Other | 84 | ITT-E | Participant Level Summary of Key Virologic Data of Background Regimens for Participants with On-Treatment Virology Results at Non-CVW timepoints | New output, same format as L.83 |

No figures for Virological Analysis

## 11.17.8. Abbreviations and Trademarks

## 11.17.8.1. Abbreviations

| ALT | Alanine aminotransferase |
|---|---|
| ART | Antiretroviral Therapy |
| BID | Twice Daily |
| DTG | Dolutegravir |
| EoS | End of Study |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials Database |
| FDAAA | Food and Drug Administration Amendment Act (2007) |
| FI | Fusion Inhibitor |
| GSS | Genotypic susceptibility score |
| IAS-USA | International Antiviral Society-USA |
| INSTI | Integrase Strand Transfer Inhibitor |
| ITT-E | Intent-to-Treat-Exposed |
| mITT-E | Modified Intent-to-Treat-Exposed |
| NRTI | Nucleoside reverse transcriptase inhibitor |
| NNRTI | Non-nucleoside reverse transcriptase inhibitor |
| CVW | Confirmed Virologic Withdrawal |
| PI | Protease Inhibitor |
| QD | Once daily |
| LPV/RTV | Lopinavir/Ritonavir |
| RAP | Reporting and analysis plan |
| RAM | Resistance Associated Mutations |
| TAM | Thymidine Analogue-Associated Mutations |

## Example Mock Shells for Data Displays

Table 2.15 Proportion of Participants Meeting CVW Criteria by Visit by Type of Virologic Failure

Protocol: 200304 

Population: Intent-To-Treat Exposed

Table 2.15
Proportion of Participants Meeting CVW Criteria by Visit by Type of Virologic Failure

| Virologic Failure Type | DTG<br>(N=31 | 2) | LPV/F<br>(N=31 | |
|------------------------|--------------|-------|----------------|-------|
| Any time | <br>296 | | 298 | |
| CVW | 27 | (X%) | 31 | (X%) |
| Virologic non-response | 4 | (1%) | 14 | (5%) |
| Rebound | 23 | (8%) | 17 | (6%) |
| Week 16 | 290 | | 296 | |
| CVW | X | (X%) | X | (X%) |
| Virologic non-response | 1 | (<1%) | 0 | |
| Rebound | 0 | | 1 | (<1%) |
| Week 24 | 293 | | 287 | , |
| CVW | XX | (X%) | XX | (X%) |
| Virologic non-response | 3 | (1%) | 11 | (4%) |
| Rebound | 2 | (<1응) | 6 | (2%) |
| • • | | | | |
| • • | | | | |
| Week 216 | | | | |

Note: The denominator for the proportion is the number of subjects with viral load data at visit week.

Note: Subjects who switched treatment from LPV/RTV to DTG by Week 52 are included in their original treatment group, and all data from before and after switch dates are included in this summary table.

Table 3.13 Summary of Serious Adverse Events by System Organ Class and Preferred Term - Continuation Phase

| System Organ Class | DTG | Switch from LPV/RTV to DTG | Total |
|---|---|---|---|
| Preferred term | N=(XX) | (N=12) | (N=XX) |
| Any Event | xx (xx%) | xx (xx%) | xx (xx%) |
| Infections and infestations | xx (xx%) | xx (xx%) | xx (xx%) |
| Any event | xx (xx%) | xx (xx%) | xx (xx%) |
| Nasopharyngitis | xx (xx%) | xx (xx%) | xx (xx%) |

### Table 4.1 Viral Genotypic Continuation Summary of Participant Accountability: Genotypes Available - Continuation phase

Reference: Sailing Table 12.1


Population: Viral Genotypic Continuation

Table 4.1

Summary of Participant Accountability: Genotypes Available - Continuation phase

| Genotype Assessment | DTG<br>( <b>N=XX</b> ) | |
|----------------------------------------|------------------------|---|
| Assessment | (N-AA) | _ |
| Integrase | | |
| Screening Sample | XX (<1%) | |
| Baseline Sample | XX (XX%) | |
| On-Treatment CVW Sample | XX (XX%) | |
| On-Treatment Non-CVW Sample | XX (<1%) | |
| Baseline & On-Treatment CVW Sample | XX (XX%) | |
| Baseline & On-Treatment Non-CVW Sample | XX (<1%) | |
| Protease | | |

Reverse Transcriptase

....

Note: 'On-treatment CVW' is at the time of confirmed virologic withdrawal.

Note: Decision tree for Monogram resistance data has been used.

Note: Baseline is set to latest pre-treatment assessment. If Day 1 sample is not available,

screening sample will be used as baseline.

200304

Table 4.2 Viral Genotypic

Summary of Emergent Major Mutations of NRTI, NNRTI and PI Classes for Participants with CVW - Randomised Phase

Table 4.201 Viral Genotypic Continuation

Summary of Emergent Major Mutations of NRTI, NNRTI and PI Classes for Participants with CVW - Continuation phase Reference Sailing 12.1


Population: Viral Genotypic

Table 4.2

Summary of Emergent Major Mutations of NRTI, NNRTI and PI Classes for Participants with CVW - Randomised

-

T DIT (DMIT

Phase

Region: NRTI

| Codon | Mutation | DTG<br>(N=11) | LPV/RTV<br>(N=30) |
|-------|--------------|---------------|-------------------|
| Any | Any Mutation | 1 (9%) | 3 (10%) |
| D67 | Any Mutation | 1 (9%) | 0 |
| | Any D67N | 1 (9%) | 0 |
| | D67N | 1 (9%) | 0 |
| K70 | Any Mutation | 0 | 2 (7%) |
| | Any K70R | 0 | 2 (7%) |
| | K70K/Q/R | 0 | 1 (3%) |
| | K70K/R | 0 | 1 (3%) |

Region: NNRTI Region: PI

Note: Decision tree for Monogram resistance data has been used

Note: Subject PPD was randomised to LPV/RTV but actually received DTG treatment and included

in the LPV/RTV treatment group.

Viral Genotypic : ITTE + after baseline PF data,

Viral Genotypic Continuation : Viral Genotypic + continuation phase PF data.

# Table 4.3 Viral Genotypic Pre-specified Treatment Emergent INSTI Substitutions at Time of Confirmed Virologic Withdrawal - Randomised Phase

# Table 4.301 Viral Genotypic Continuation Pre-specified Treatment Emergent INSTI Substitutions at Time of Confirmed Virologic Withdrawal - Continuation Phase

Protocol: 200304 

Population: Viral Genotypic

Table 4.3

Summary of Emergent Pre-specified INSTI Substitutions at Time of Confirmed Virologic Withdrawal During the Randomisation Phase

Region: INSTI

| Codon | Mutation | DTG<br>(N=XX) | LPV/RTV<br>(N=XX) |
|-------|--------------|---------------|-------------------|
| Any | Any Mutation | XX (XX%) | XX (XX%) |
| 51 | n | XX (XX%) | 0 |
| | Any Change | XX (XX%) | 0 |
| | H51H/Y | XX (XX%) | 0 |

Note: Pre-specified INSTI Substitutions Associated with Development of Resistance to INSTI Class: H51Y, T66A, T66I, T66K, L74M, E92Q, E92V, E92G, Q95K, T97A, G118R, F121Y, E138A, E138K, G140A, G140C, G140S, Y143C, Y143H, Y143R, Y143K, Y143S, Y143G, Y143A, P145S, Q146P, S147G, Q148N, Q148K, Q148K, V151I, V151L, V151A, S153F,S153Y, N155H, N155S, N155T, E157Q, G163R, G163K, S230R, R263K, L68V\*, L68I\*, L74I\*, E138T\*, G193E\*
Note: Decision tree for Monogram resistance data has been used
Note: Subject PPD was randomised to LPV/RTV but actually received DTG treatment and included in the LPV/RTV treatment group.

#### Table 4.5 Viral Phenotypic Continuation

#### Summary of Participant Accountability: Phenotype Available - Continuation phase

Protocol: 200304 

Population: Viral Phenotypic Continuation

Table 4.5

Summary of Participant Accountability: Phenotypes Available - Continuation phase

| Phenotype<br>Assessment | DTG<br>(N=XX) |
|---|---|
| INSTI Screening Sample Baseline Sample On-Treatment CVW Sample On-Treatment Non-CVW Sample Baseline & On-Treatment CVW Sample Baseline & On-Treatment CVW Sample | XX (<1%)<br>XX (XX%)<br>XX (XX%)<br>XX (<1%)<br>XX (XX%)<br>XX (<1%) |
| NRTI PI NNRTI | |

Note: 'On-treatment CVW' is at the time of confirmed virologic withdrawal.

Note: Decision tree for Monogram resistance data has been used

Note: Baseline is set to latest pre-treatment assessment. If Day 1 sample is not available,

screening sample will be used as baseline.

Table 4.8 Viral Phenotypic Continuation
Phase Reference sailing table 12.8 Summary of Fold Change to DTG at Baseline and Time of CVW - Continuation


Population: Viral Phenotypic Continuation

| Drug | Timepoint | | DTG<br>(N=11) | LPV/RTV (N=29) |
|------|-----------|---------------------|---------------|----------------|
| DTG | Baseline | Fold Change | | |
| | | n | 11 | 27 |
| | | <1 | 5 (45%) | 17 (59%) |
| | | 1-<2 | 6 (55%) | |
| | | 2-<4 | 0 | 0 |
| | | 4-<8 | 0 | 0 |
| | | >=8 | 0 | 0 |
| | | Fold Change (class) | | |
| | | n | 11 | 27 |
| | | Geom. Mean | 0.99 | 0.94 |
| | | CV (%) | 20.180 | 24.976 |
| | | Median | 1.02 | 0.94 |
| | | Q1 | 0.84 | 0.78 |
| | | Q3 | 1.08 | 1.12 |
| | | Min. | 0.68 | 0.65 |
| | | Max. | 1.41 | 1.91 |
| DTG | CVW | Fold Change | | |

Note: CV (Coefficient of Variation) =  $100*sqrt(exp((SD on log scale)^2)-1)$ .

Note: Decision tree for Monogram resistance data has been used

#### Listing Other 77 ITT-E Listing of All Genotypic Data

#### Reference Sailing Listing 34

- Show all available PFGRPID test results, for example PSGT AA, and PSGTIN AA for the same visit.

Protocol: 200304 Page 1 of x

Population: ITT-E

Listing 77

Listing of All Genotypic Data

Treatment: DTG

Date/

Week 36

Sched. Visit/

| Site ID./Unique Subj. | Actual Visit/<br>Phase | Protease | - | Integrase | Clade | IN<br>assay | PRO/RT<br>Assay |
|---|---|---|---|---|---|---|---|
| 200304.PPD | • | H69K, I93L,<br>L19T, L63L/V,<br>L89M, M36I, | A272P, C162S, D123G, D177E, E291D, E36E/A, I135V, I159I/V, I202V, *K103K/N, K122E, K173A/T, P176P/S, Q102K, Q174K, Q207E, R211R/K, S163S/T, S48T, T165T/I, T200A, T286T/A, T39E, V245Q, V292I, V35T, V60I, V8V/INR= Not Rep | D25E, D278A, I84M, K136Q, K173R, K219Q, L101I, S283S/G, T112V, T124A, T218I, V113I, V201I, V234I, V31I, V72I | С | GSIN | PSGT |
| WEEK | 36/ NR | NR | | NR | PSGTI | I PSGTII | N |

L77: where parcd in ("FOLDCHG", "IC50", "PSASM") and parcatl="PHENOTYPE" and PHENFL="Y";

L78: where paramcd ="AA" and dnareg in ("INTEGRASE", "PROTEASE", "REVERSE TRANSCRIPTASE") and GENFL="Y";

<sup>&#</sup>x27;\*' These represent the known INSTI mutations as defined in table 1 and major mutations for Protease and Reverse Transcriptase as defined in table 2 from EOS RAP.

#### Listing Other 78 ITT-E Listing of All Phenotypic Data Reference Sailing Listing 35


Population: ITT-E

Listing 78

Listing of All Phenotypic Data

Treatment: DTG

| Site ID./Unique<br>Subj. | Time Point<br>Phase | Drug<br>Class | Drug<br>Drug Name | IC50<br>(NMOL/L) | Fold<br>Change | Sensitivity [1] | PRO/RT<br>Assay | IN<br>Assay |
|---|---|---|---|---|---|---|---|---|
| PPD<br>200304.PPD | DAY 1/<br>Day 1/<br>Randomised | INI | DOLUTEGRAVIR | 2.728 | 1.02 | Sensitive | | PSIN |
| | Randomised | | ELVITEGRAVIR | 2.02 | 0.96 | Sensitive | | PSIN |
| | | | RALTEGRAVIR | 4.96 | 0.81 | Sensitive | | PSIN |
| | | NNRTI | DELAVIRDINE | > 5000 | >120.52 | Resistant | PSGT | |
| 200304 PPD | DAY 1/<br>Day 1/ | INI | DOLUTEGRAVIR | NR | | PSGTIN | PSGTIN | |

Note: Subject  $\stackrel{\text{PPD}}{=}$  was randomised to LPV/RTV but actually received DTG treatment and included

in the LPV/RTV treatment group.

Note: NR= Not Reported.

Listing Other 80 ITT-E Listing of Virology Data for Participants with CVW, Display data in both randomised and continuation phases, separating by phases.

Listing Other 82 ITT-E Listing of Virology Data for Participants with On-Treatment Virology Results at Non-CVW timepoints

- Pick test results with decision tree


Population: Intent-to-Treat Exposed

Listing 80

Listing of Virology Data for Participants with CVW

Treatment: DTG

| Site Id. Unique Subject Id./ CVW Visit/ CVW Date/ CVW Type/ Bkgd. ART Phase | Susc. Score Bkgd. ART at BL PSSf/ PSSp/ GSS | Susc. Score Bkgd. ART at CVW PSSf/ | Susc.<br>Score<br>DTG<br>at<br>BL<br> | Susc.<br>Score<br>DTG<br>at<br>CVW | INSTI | PR/RT<br>RC | Mut | INSTI<br>Mutations | | Major<br>NNRTI | Major<br>PI | Clade | Switch<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CVW Type/<br>Bkgd. ART | | PSSp/ PSSp/ | PSSp/<br>GSS | PSSf/<br>PSSp/<br>GSS | | BL/<br>CVW | BL<br>CV | ./ | BL/<br>CVW | BL/<br>CVW | BL/<br>CVW | | VISIC |
| PPD / 200304.0000XX/ | 2/<br>2/<br>1.25 | 2/<br>2/<br>1.5 | 1/<br>1/<br>1 | 1/<br>1/<br>1 | 1/<br>1/<br>1 | 1/<br>1 | 93/<br>108 | 101/<br>136 | NA/<br>None | NA/<br>None | NA/<br>A123C | В | Week 52 |

Rebound/ ATV/r,TDF Randamized phase

#### Treatment: LPV/r

| | CVM | ect Id./<br>Visit/<br>Date/<br>Type/<br>ART | Susc. Score Bkgd. ART at BL PSSf/ PSSp/ GSS | Susc.<br>Score<br>Bkgd.<br>ART<br>at<br>CVW<br><br>PSSf/<br>PSSp/<br>GSS | Susc.<br>Score<br>LPV/r<br>at<br>BL<br><br>PSSf/<br>PSSp/<br>GSS | Susc. Score LPV/r at CVW PSSf/ PSSp/ GSS | INSTI | PR/RT<br>RC<br><br>BL/<br>CVW | INSTI<br>Mutations<br><br>BL/<br>CVW | Major<br>NRTI<br>BL/<br>CVW | Major<br>NNRTI<br>BL/<br>CVW | Major<br>PI<br>BL/<br>CVW | Clade | Switch<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | PPD | | | | | | | | | | | | - | |
| | | A DDD | 2/ | 2/ | 1/ | 1/ | 93/ | 101/ | | | | | | |
| | Week | 4.PPD / | 2/<br>1.25 | 2/<br>1.5 | 1/ | 1/ | 108 | 136 | | | | | | |
| | PPD | 32/ | 1.25 | 1.5 | 1 | 1 | | | | | | | | |
| | Rebou | nd/ | | | | | | | | | | | | |
| | ATV/r | | | | | | | | | | | | | |
| | | mized phase | e | | | | | | | | | | | |
| SV | W | PPD | | | | | | | | | | | | |
| CV<br>PF | W<br>DTC | | within 4 wee | | right da | te PPD | is s | ame as SV | W date. | | | | | |

Note: CVW Visit = Actual visit window of the initial suspected viral load sample, which was subsequently confirmed. NR= Not Reported, FC = Fold Change in IC50 relative to Wild-Type, RC = Replication Capacity.

Note: INSTI mutations include the specified known INSTI mutations listed in EOS RAP Table 1.

Note: NA indicates either assay failed or not done.

Note: \* indicate that tests results are picked using decision tree.

Listing 83: Participant Level Summary of Key Virologic Data of Background Regimens for Participants with On-Treatment Virology Results at CVW Timepoints

Listing 84: Participant Level Summary of Key Virologic Data of Background Regimens for Participants with On-Treatment Virology Results at Non-CVW Timepoints


Population: Intent-to-Treat Exposed

Listing 83

Participant level summary of Key virologic Data of background regimens for Participant with on-treatment Virology results at CVW timepoint

| Treatmen<br>Site | iit. Dio | | | | | _Backgroun | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Id./<br>Unique<br>Subject<br>Id. | Time point/<br>CVW/<br>Phase | Actual<br>Visit/<br>Visit date | Drug Name | GSS** | PSS* | Fold<br>change | Stanford<br>Sens./<br>Genotypic<br>Sens. | Phenotypic<br>Sens. | Net<br>Assess. | Switch<br>Visit |
| PPD<br>PD | Baseline/ | Day 1/ | EMTRICITABINE | 1 | 1 | 1.08 | Sensitive/<br>Sensitive | Susceptible | Susceptible | У |
| | | | TENOFOVIR | 1 | 1 | 0.96 | Sensitive | Susceptible | | |
| | CVW/<br>Randomised | Week 36/<br>PPD | EMTRICITABINE | 1 | 1 | 0.89 | Sensitive | Susceptible | Y | |
| | Treatment | | TENOFOVIR | 1 | 1 | 0.79 | Sensitive | Susceptible | | |

<sup>\*:</sup> individual drug susceptibility score using PSSF.

Note: Not per-protocol resistance testing (genotype only) was performed at Q2 Solutions for Subject PPD after subject withdrawal.

# 11.18. Appendix 18 –List of Data Displays

## 11.18.1. **Data Display Numbering**

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacokinetic / Pharmacodynamic | 6.1 to 6.n | 6.1 to 6.n |
| Section | Listi | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to | ) Z |

## 11.18.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in a separate document.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Virology | VI_Fn | VI _Tn | VI _Ln |
| Health Outcome | HO_Fn | HO_Tn | HO_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 11.18.3. **Deliverable**

| Delivery | Description |
|----------|------------------------------------------------|
| 24 Week | Interim Analysis Statistical Analysis Complete |
| 48 Week | Primary Statistical Analysis Complete |

The following phases are defined: R=Randomised Phase and RC=Randomised Phase and ContinuationPhase.

Phase of the deliverable labelled as R/RC means that the output will initially be created based on the Randomised Phase only then repeated based on the Randomised Phase and Continuation Phase. Deliverables without a Phase are assumed to be for the Randomised phase only

# 11.18.4. **Study Population**

# 11.18.4.1. Tables

| Stud | y Population | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| Subj | ect dispositio | n | | | |
| 1.1. | All<br>Subjects<br>Screened | SP1 | Summary of Study<br>Populations | CS CORE | 24wk, 48wk |
| 1.2. | All<br>Subjects<br>Screened | NS1 | Summary of Subjects by Country and Investigator | CS CORE | 24wk, 48wk |
| 1.3. | ITT-E | EudraCT age<br>DM11 | Summary of Age<br>Categories | CS CORE | 24wk, 48wk |
| 1.4. | All<br>Subjects<br>Screened | ES6 | Summary of Reasons for Screen Failure | CS CORE | 24wk, 48wk |
| 1.5. | ITT-E | ES1 | Summary of Subject<br>Accountability: Study<br>Conclusion Record | | 24wk, 48wk |
| 1.6. | ITT-E | ES1 | Summary of Subject<br>Accountability:<br>Randomised Phase<br>Conclusion Record | | 24wk, 48wk |
| 1.7. | ITT-E | ES1 | Summary of Subject<br>Accountability:<br>Continuation Phase<br>Conclusion Record | | 24wk, 48wk |

| Stud | y Population | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.8. | ITT-E | HIV_ES1 | Summary of Subject<br>Accountability:<br>Withdrawals by Visit | | 24wk, 48wk |
| 1.9. | ITT-E | SD1 | Summary of Treatment Status | | |
| 1.10. | ITT-E | DV1 | Summary of Important Protocol Deviations | CS CORE | 24wk, 48wk |
| 1.11. | ITT-E | SP2 | Summary of Protocol Deviations Leading to Exclusion from the Per- Protocol Population | CS CORE. Only deviations occurring in the period of interest can lead to exclusion from the PP Population. | 24wk, 48wk |
| 1.12. | ITT-E | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | 24wk, 48wk |
| Dem | ography | | 1 | 1 | " |
| 1.13. | ITT-E | DM1 | Summary of Demographic Characteristics | CS CORE | 24wk, 48wk |
| 1.14. | ITT-E | DM5 | Summary of Race and Racial Combinations | CS CORE | 24wk, 48wk |
| 1.15. | ITT-E | DM6 | Summary of Race and Racial Combinations Details | CS CORE | 24wk, 48wk |
| 1.16. | ITT-E | DM8 | Summary of All<br>Indicated Races | | |

| Stud | y Population | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.17. | ITT-E | CDC1 | Summary of CDC<br>Classification of HIV<br>Infection at Baseline | | 24wk, 48wk |
| 1.18. | ITT-E | Shell POP_T1 gsk2619619/ing117172/week48/drivers/cr_t_cvrf.sas | Summary of Baseline<br>Cardiovascular Risk<br>Assessments | | 24wk, 48wk |
| 1.19. | ITT-E | Shell POP_T2<br>gsk2619619/ing117172/week48/drivers/vl_t_scrnbl_hivrna.sas | Distribution of Quantitative Plasma HIV-1 RNA Results at Screening and Baseline | Include a category of viral load <400 especially for screening (ie to identify screening failure). Added <400 at baseline too. | 24wk, 48wk |
| 1.20. | ITT-E | Shell POP_T3 gsk2619619/ing117172/week48/drivers/vl_t_scrnbl_cd4.sas | Distribution of CD4+ Cell<br>Count (cells/mm^3)<br>Results at Screening<br>and Baseline | | 24wk, 48wk |
| 1.21. | ITT-E | Shell POP_T4 gsk2619619/ing117172/week48/drivers/lb_t_hep.sas | Summary of Hepatitis<br>Status at Entry | | 24wk, 48wk |
| Medi | ical Condition | & Concomitant Medications | | | |
| 1.22. | ITT-E | MH1 | Summary of Current<br>Medical Conditions | CS CORE | 24wk, 48wk |
| 1.23. | ITT-E | MH1 | Summary of Past<br>Medical Conditions | CS CORE | 24wk, 48wk |

| Stud | ly Population | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.24. | ITT-E | MH4 | Summary of Current<br>Cardiac,<br>Gastrointestinal,<br>Metabolism and<br>Nutrition, Psychiatric,<br>Renal and Urinary, and<br>Nervous System<br>Conditions | | 24wk, 48wk |
| 1.25. | . ITT-E | MH4 | Summary of Past Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions | | 24wk, 48wk |
| 1.26. | ITT-E | CM1 | Summary of Concomitant Medication by Ingredient ATC Level 1 | CS CORE | 24wk, 48wk |
| 1.27. | ITT-E | CM8 | Summary of Concomitant Medication Ingredient Combinations | | 24wk, 48wk |
| 1.28. | . ITT-E | CM1b | Summary of Concomitant Medication by Combination Term ATC Level 1 | | 24wk, 48wk |

| Stud | y Population | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.29. | ITT-E | Shell POP_T5 gsk1349572/ing111762/week48/drivers/cm_t_prior.sas | Summary of Prior<br>Antiretroviral Therapy at<br>the time of Screening | | 24wk, 48wk |
| 1.30. | ITT-E | Use shell for POP_T5 | Summary of Prior Antiretroviral Therapy discontinued prior to Screening | | 24wk, 48wk |
| 1.31. | ITT-E | Shell POP_T6 | Summary of Prior Antiretroviral Therapy at the time of screening – First line combination | New output | 24wk, 48wk |
| 1.32. | ITT-E | Shell POP_T7 /arenv/arprod/gsk1349572/ing111762/week48/drivers/cm_t_prinum.sas | Summary of Prior<br>Antiretroviral Therapy<br>Classes at time of<br>Screening | Only create if we have more than 10 subjects with a prior ART other than NNRTI+NRTI. | 24wk, 48wk |
| 1.33. | ITT-E | Shell POP_T8 gsk1349572/ing111762/week48/drivers/cm_t_pridur.sas | Summary of Duration of<br>Prior Antiretroviral<br>Therapy at time of<br>Screening | | 24wk, 48wk |
| 1.34. | ITT-E | Shell POP_T9 gsk1349572/ing111762/week48/drivers/cm_t_day1.sas | Summary of Background Antiretroviral Therapy Received at Time of IP Start by Agent Combination | | 24wk, 48wk |
| 1.35. | ITT-E | Shell POP_T10<br>gsk1349572/ing111762/week48/drivers/cm_t_lipid_bl.sas | Summary of Lipid<br>Modifying Agent Use at<br>Baseline | | 24wk, 48wk |

| Stud | y Population 1 | Fables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.36. | ITT-E | Shell POP_T11 gsk1349572/ing111762/week48/drivers/cm_t_lipid_postbl.sas | Summary of Lipid<br>Modifying Agent Use<br>Starting Post-Baseline | | 24wk, 48wk |
| Virol | ogy | | <u>-</u> | | |
| 1.37. | ITT-E | Shell POP_T12 ing111762/week48/drivers/cm_t_classres.sas | Summary of the Number of Baseline Major Mutations Associated with the Resistance to NRTI, NNRTI, and PI drug classes | | 24wk, 48wk |
| 1.38. | ITT-E | Shell POP_T13<br>gsk1349572/ing111762/week48/drivers/mu_t_bl_maj_oth.sas | Summary of the Number of<br>Baseline Major<br>Substitution to NRTI,<br>NNRTI and PI Drug<br>Classes | | |
| 1.39. | All<br>Screened<br>Subjects | Shell POP_T14 | Proportion of subjects without at least 1 fully active NRTI | | 24wk, 48wk |
| 1.40. | All<br>Screened<br>Subjects | Shell POP_T15 ing111762/week48/drivers/cm_t_classres.sas | Summary of the Number of Screening Major Mutations Associated with the Resistance to NRTI, NNRTI, and PI drug classes | Screening genotypic data is all from Q2. There may be some subtle differences to discuss with programmers compared with the Monogram data. For Q2 if there is an insertion it may not be possible to determine precise order. | 24wk, 48wk |

| Study Population Tables | | | | | 1 |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.41. | All<br>Screened<br>Subjects | Shell POP_T16<br>gsk1349572/ing111762/week48/drivers/mu_t_bl_maj_oth.sas | Summary of the Number<br>of Screening Major<br>Substitution to NRTI,<br>NNRTI and PI Drug<br>Classes | Screening genotypic data is all from Q2. There may be some subtle differences to discuss with programmers compared with the Monogram data. For Q2 if there is an insertion it may not be possible to determine precise order. | 24wk, 48wk |

| Stuc | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.42 | . ITT-E | Shell POP_T17 | Summary of Baseline Major NNRTI and NRTI Mutations | New table which includes: Number of thymidine analogue-associated mutations (TAMS): 1, 2, >2 Prevalence of L65A or L70G 69 insertion complex 151 insertion complex Other major NRTI mutations Prevalence of M184V only M184V with any other major NRTI mutation [proposed new output to match that of the SECONDLINE Kirby manuscript] | 24wk, 48wk |

| Stud | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.43. | . ITT-E | Shell POP_T18 gsk1349572/ing111762/week24/drivers/ph_t_bl_geno_gssd11.sas | Summary of Stanford<br>Baseline GSS to<br>Background ART<br>Regimen | | 24wk, 48wk |
| 1.44. | . ITT-E | Shell POP_T19 gsk1349572/ing111762/week24/drivers/ph_t_bl_geno_gssd11.sas | Summary of Monogram<br>Baseline GSS to<br>Background ART<br>Regimen | New table. Use summary of Stanford GSS summary as a shell. | 24wk, 48wk |
| 1.45. | . ITT-E | Shell POP_T20<br>gsk1349572/ing112574/week48/drivers/ph_t_bossfbng_d8.sas | Summary of Baseline<br>OSS (Net Assessment)<br>to Background Therapy | Viking T12.71 | 24wk, 48wk |
| 1.46. | . ITT-E | Shell POP_T21 sk1349572/ing111762/week24/drivers/ph_t_basepss.sas | Summary of Baseline<br>PSS to Background<br>ART Regimen | | 24wk, 48wk |
| 1.47. | . ITT-E | Shell POP_T22<br>gsk1349572/ing111762/week24/drivers/mu_t_hiv_clades.sas | Summary of the<br>Prevalence of HIV-1<br>Clades at Baseline by<br>Frequency | Use Monogram Testing For W24, for <u>China</u> we will have mostly Q2 genotype and just a few Monogram testings of the samples that we were able to export for testing. | 24wk, 48wk |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 1.48 | . ITT-E | Shell POP_T23 | Summary of First Line<br>Regimen and Expected<br>Second Line Regimen<br>Using the WHO<br>Algorithm | New table | 24 wk, 48<br>wk |
| 1.49 | . ITT-E | Shell POP_T24 | Summary of Expected WHO Second Line vs. Background Regimen actually Taken | New table | 24 wk, 48<br>wk |
# 11.18.5. **Efficacy**

### 11.18.5.1. Tables

| Effic | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| Prim | ary | | | | |
| 2.1. | ITT-E | Shell EFF_T1<br>gsk2619619/ing117172/week48/drivers/t_ef_analprop.sas | Summary of Analysis of<br>Proportion of Subjects with<br>Plasma HIV-1 RNA <50 c/mL<br>at Week 24/48 – Snapshot<br>Analysis | | 24wk, 48wk |
| 2.2. | Per-<br>Protocol | Shell EFF_T2 | Summary of Analysis of Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 24/48 – Snapshot Analysis | | 24wk48wk |
| 2.3. | Intent to treat | Shell EFF_T3 | Summary of Analysis of Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 24/48 – Snapshot Analysis | | 24wk, 48wk |
| 2.4. | ITT-E | Shell EFF_T4 gsk2619619/ing117172/week48/drivers/t_sn_studout.sas | Summary of Study Outcomes<br>(<50 c/mL) at Week 24/48 –<br>Snapshot Analysis | | 24wk, 48wk |
| 2.5. | ITT-E | Shell EFF_T6 gsk2619619/ing117172/week48/drivers/t_snap_sum_prop_p.sas | Treatment by Strata Tests of Homogeneity for the Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 24/48-Snapshot Analysis | | 24wk, 48wk |

| Effic | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 2.6. | ITT-E | Shell EFF_T7 gsk2619619/ing117172/week48/drivers/t_sn_studout.sas | Summary of Study Outcomes<br>(<50 c/mL) at Week 24/48 –<br>by number of fully active<br>background NRTIs | | 24wk, 48wk |
| 2.7. | ITT-E | Shell EFF_T8 gsk2619619/ing117172/week48/drivers/t_snap_sum_prop.sas | Proportion of Subjects with<br>Plasma HIV-1 RNA <50 c/mL<br>at Week 24/48by Subgroup -<br>Snapshot Analysis | Note: only present by<br>ABC+3TC vs non<br>ABC+3TC if more<br>than 10 subjects took<br>ABC+3TC | 24wk, 48wk |
| 2.8. | ITT-E | Shell EFF_T9 gsk2619619/ing117172/week48/drivers/t_snap_prop_50.sas | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit - Snapshot Analysis | | 24wk, 48wk |
| 2.9. | ITT-E | Shell EFF_T10<br>gsk2619619/ing117172/week48/drivers/t_snap_prop_50.sas | Proportion of Subjects with Plasma HIV-1 RNA<50 c/mL by Visit and Subgroup – Snapshot Analysis | Adapt program to include subgroups | 24wk, 48wk |
| 2.10. | ITT-E | Shell EFF_T11 gsk2619619/ing117172/week48/drivers/t_snap_prop_400.sas | Proportion of Subjects with<br>Plasma HIV-1 RNA <400 c/mL<br>by Visit - Snapshot Analysis | | 24wk, 48wk |
| 2.11. | ITT-E | Shell EFF_T12<br>gsk2619619/ing117172/week48/drivers/t_sn_studout_400.sas | Summary of Study Outcomes<br>(<400 c/mL) at Week X –<br>Snapshot Analysis | | 24wk, 48wk |
| 2.12. | . ITT-E | Shell EFF_T13 gsk2619619/ing117172/week48/drivers/t_ef_km_trdf.sas | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal Criteria at Week 48 - Treatment Related Discontinuation = Failure | TTE6 | 24wk, 48wk |

| Effic | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 2.13. | ITT-E | Shell EFF_T14 gsk2619619/ing117172/week48/drivers/t_ef_km_erdf.sas | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal Criteria at Week 48 - Efficacy Related Discontinuation = Failure | TTE6 | 24wk, 48wk |
| 2.14. | ITT-E | Shell EFF_T15 /arenv/arprod/gsk1349572/ing114467/week48/drivers/ef_t_pdvf_vis.sas | Proportion of Subjects Meeting<br>Confirmed Virologic<br>Withdrawal Criteria by Visit | | 24wk, 48wk |
| 2.15. | ITT-E | Shell EFF_T16 /arenv/arprod/gsk1349572/ing111762/week48/drivers/ef_t_pdvf_vis.sas | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Withdrawal Criteria by<br>Visit by Type of Virologic<br>Failure | | 24wk, 48wk |
| 2.16. | ITT-E | Shell EFF_T17 gsk1349572/ing111762/week48/drivers/ef_t_pdvf_dist.sas | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Virologic Withdrawal Criteria | | 24wk, 48wk |
| 2.17. | ITT-E | Shell EFF_T18 gsk1349572/ing114915/week48/drivers/ef_t_km_timeto_sup50.sas | Summary of Kaplan-Meier<br>Estimates of Time to Viral<br>Suppression (HIV-1 RNA <50<br>c/mL) | | 24wk, 48wk |
| 2.18. | ITT-E | Shell EFF_T19 | Proportion of Subjects With<br>Detectable Viral Load Below<br>the Limit of Quantification at<br>Week 24/48 | | 24wk, 48wk |

| Effic | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 2.19. | ITT-E | HIV1 | Summary of Post-Baseline<br>HIV-1 Associated Conditions<br>Including Recurrences | | 24wk, 48wk |
| 2.20. | ITT-E | HIV1 | Summary of Post-Baseline<br>HIV-1 Associated Conditions<br>Excluding Recurrences | | 24wk, 48wk |
| 2.21. | ITT-E | HIV2 | Summary of Post-Baseline<br>HIV-1 Disease Progressions | | 24wk, 48wk |
| 2.22. | ITT-E | Shell EFF_T19 gsk2619619/ing117172/week48/drivers/ef_t_cd4_chg.sas | Summary of Change from<br>Baseline in CD4+ Cell Count<br>(cells/mm^3) by Visit | | 24wk, 48wk |
| 2.23. | ITT-E | Shell EFF_T20 gsk2619619/ing117172/week48/drivers/t_ef_hv1rn_chg.sas | Summary of Change from<br>Baseline in Plasma HIV-1 RNA<br>(log10 c/mL) by Visit | | 24wk, 48wk |
| 2.24. | ITT-E | Shell EFF_T21<br>gsk2619619/ing117172/week48/drivers/t_sn_studout.sas | Summary of Study Outcomes<br>(<50 c/mL) at Week X by<br>[Subgroup] – Snapshot<br>Analysis | As Needed. Modify program to present by subgroups. | 24wk, 48wk |
| 2.25. | ITT-E | Shell EFF_T1<br>gsk2619619/ing117172/week48/drivers/t_ef_analprop.sas | Summary of Analysis of Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 – Snapshot Analysis – Additional Estimand 1 | | 48wk |
| 2.26. | ITT-E | Shell EFF_T4 gsk2619619/ing117172/week48/drivers/t_sn_studout.sas | Summary of Study Outcomes<br>(<50 c/mL) at Week 48 –<br>Snapshot Analysis – Additional<br>Estimand 1 | | 48wk |

| Effic | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 2.27. | ITT-E | Shell EFF_T1<br>gsk2619619/ing117172/week48/drivers/t_ef_analprop.sas | Summary of Analysis of<br>Proportion of Subjects with<br>Plasma HIV-1 RNA <50 c/mL<br>at Week 48 – Snapshot<br>Analysis – Additional Estimand<br>2 | | 48wk |
| 2.28. | ITT-E | Shell EFF_T4 gsk2619619/ing117172/week48/drivers/t_sn_studout.sas | Summary of Study Outcomes<br>(<50 c/mL) at Week 48 –<br>Snapshot Analysis – Additional<br>Estimand 2 | | 48wk |
| 2.29. | MITT-E-36 | Shell EFF_T1<br>gsk2619619/ing117172/week48/drivers/t_ef_analprop.sas | Summary of Analysis of<br>Proportion of Subjects with<br>Plasma HIV-1 RNA <50 c/mL<br>at Week 36 – Snapshot<br>Analysis | | 24wk |
| 2.30. | MITT-E-36 | Shell EFF_T4 gsk2619619/ing117172/week48/drivers/t_sn_studout.sas | Summary of Study Outcomes<br>(<50 c/mL) at Week 36 –<br>Snapshot Analysis | | 24wk |
| 2.31. | MITT-E-48 | Shell EFF_T1<br>gsk2619619/ing117172/week48/drivers/t_ef_analprop.sas | Summary of Analysis of Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 – Snapshot Analysis | | 24wk |
| 2.32. | MITT-E-48 | Shell EFF_T4<br>gsk2619619/ing117172/week48/drivers/t_sn_studout.sas | Summary of Study Outcomes<br>(<50 c/mL) at Week 48 –<br>Snapshot Analysis | | 24wk |

| Effic | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 2.33. | MITT-E-36 | Shell EFF_T13 gsk2619619/ing117172/week48/drivers/t_ef_km_trdf.sas | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal Criteria at Week 36 - Treatment Related Discontinuation = Failure | TTE6 | 24wk |
| 2.34. | MITT-E-48 | Shell EFF_T13 gsk2619619/ing117172/week48/drivers/t_ef_km_trdf.sas | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal Criteria at Week 48 - Treatment Related Discontinuation = Failure | TTE6 | 24wk |
| 2.35. | ITT-E | Shell EFF_T13 gsk2619619/ing117172/week48/drivers/t_ef_km_trdf.sas | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal Criteria at Week 48 - Treatment Related Discontinuation = Failure — Sensitvity Analysis | TTE6 | 48wk |

| Effic | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 2.36. | ITT-E | Shell EFF_T14 gsk2619619/ing117172/week48/drivers/t_ef_km_erdf.sas | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal Criteria at Week 48 - Efficacy Related Discontinuation = Failure — Sensitvity Analysis | TTE6 | 48wk |
| 2.37. | . ITT-E | Shell EFF_T1<br>gsk2619619/ing117172/week48/drivers/t_ef_analprop.sas | Summary of Analysis of Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 – Snapshot Analysis – Projected Estimate | | 24wk |
| 2.38. | . ITT-E | Shell EFF_T4 gsk2619619/ing117172/week48/drivers/t_sn_studout.sas | Summary of Study Outcomes<br>(<50 c/mL) at Week 48 –<br>Snapshot Analysis – Projected<br>Estimate | | 24wk |

# 11.18.5.2. Efficacy Figures

| Effic | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 2.1. | ITT-E | Shell EFF_F1 gsk2619619/ing117172/week48/drivers/ef_f_p50.sas | Proportion (95% CI) of Subjects with HIV-<br>1 RNA <50 c/mL by Visit – Snapshot<br>Analysis | Week 24: Up to Week 24<br>Data<br>Week 48: Up to Week 48<br>Data | 24wk, 48wk |
| 2.2. | ITT-E | Shell EFF_F2 gsk2619619/ing117172/week48/drivers/ef_f_diffprop.sas | Unadjusted Treatment Difference in Proportion (95%) of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 24/48 by Subgroup – Snapshot Analysis | | 24wk, 48wk |
| 2.3. | ITT-E | Shell EFF_F3<br>gsk2619619/ing117172/week48/drivers/ef_f_p50.sas | Proportion (95% CI) of Subjects with HIV-<br>1 RNA <400 c/mL by Visit – Snapshot<br>Analysis | Use <400 cut-off instead<br>of <50 cut-off<br>Week 24: Up to Week 24<br>Data<br>Week 48: Up to Week 48<br>Data | 24wk, 48wk |
| 2.4. | ITT-E | Shell EFF_F4 gsk1349572/ing111762/week48/drivers/ef_f_km_trdf.sas | Kaplan-Meier Plot of Time to Failure by<br>Week 24– Treatment Related<br>Discontinuation = Failure | | 24wk, 48wk |
| 2.5. | MITT-E-36 | Shell EFF_F4 gsk1349572/ing111762/week48/drivers/ef_f_km_trdf.sas | Kaplan-Meier Plot of Time to Failure by<br>Week 36– Treatment Related<br>Discontinuation = Failure | | 24wk |
| 2.6. | MITT-E-48 | Shell EFF_F4 gsk1349572/ing111762/week48/drivers/ef_f_km_trdf.sas | Kaplan-Meier Plot of Time to Failure by<br>Week 48 – Treatment Related<br>Discontinuation = Failure | | 24wk |
| 2.7. | ITT-E | Shell EFF_F5 gsk1349572/ing111762/week48/drivers/ef_f_km_erdf.sas | Kaplan-Meier Plot of Time to Failure –<br>Efficacy Related Discontinuation = Failure | | 24wk, 48wk |

| Effic | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 2.8. | ITT-E | Shell EFF_F6 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit | | 24wk, 48wk |
| 2.9. | ITT-E | Shell EFF_F7 | Change from Baseline in CD4+ Cell Count (cells/mm^3) by visit | New figure | 24wk, 48wk |

## 11.18.6. **Safety**

### 11.18.6.1. Tables

| Safe | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| Adve | erse Events | | | | |
| 3.1. | Safety | Shell SAFE_T1 gsk2619619/ing117172/week48/drivers/ex_t_exposure_rand.sas | Summary of Extent of Exposure to Investigational Product for the Randomised Phase | CS Core | 24wk, 48wk |
| 3.2. | Safety | Shell SAFE_T2 gsk2619619/ing117172/week48/drivers/ex_t_exposure.sas | Summary of Extent of Exposure to Investigational Product for the Randomised and Continuation Phases | | 24wk, 48wk |
| 3.3. | Safety | Shell SAFE_T3 gsk1349572/ing114467/week48/drivers/ae_t_stats_neuro_psych.sas | Statistical Analysis of Grade 2 or greater Drug-Related Diarrhoea | New output. | 24wk, 48wk |
| 3.4. | Safety | ÄE1 | Summary of All Adverse Events<br>by System Organ Class | CS Core (optional) | 24wk, 48wk<br>R, RC |
| 3.5. | Safety | AE5B | Summary of All Adverse Events<br>by System Organ Class and<br>Maximum Toxicity | CS Core | 24wk, 48wk<br>R, RC |
| 3.6. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | CS Core | 24wk, 48wk |
| 3.7. | Safety | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events by Overall Frequency | CS Core | 24wk, 48wk |
| 3.8. | Safety | AE1 | Summary of All Grade 2-4 Adverse Events by System Organ Class | | 24wk, 48wk |

| Safe | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 3.9. | Safety | AE5B | Summary of All Drug-Related<br>Adverse Events by System Organ<br>Class and Maximum Toxicity | CS Core | 24wk, 48wk<br>R, RC |
| 3.10. | Safety | AE1 | Summary of All Drug-Related<br>Adverse Events by System Organ<br>Class | CS Core | 24wk, 48wk |
| 3.11. | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency | CS Core | 24wk, 48wk |
| 3.12. | Safety | AE1 | Summary of All Drug-Related<br>Grade 2-4 Adverse Events by<br>System Organ Class | | 24wk, 48wk |
| 3.13. | Safety | AE1 | Summary of Serious Adverse<br>Events by System Organ Class | CS Core | 24wk, 48wk<br>R, RC |
| 3.14. | Safety | AE3 | Summary of Drug-Related Fatal Serious Adverse Events | | 24wk, 48<br>wk |
| 3.15. | Safety | AE1 | Summary of Drug-Related<br>Serious Adverse Events by<br>System Organ Class | CS Core | 24wk, 48wk |
| 3.16. | Safety | AE3 | Summary of Non-Fatal Serious<br>AEs | | 24wk, 48wk |
| 3.17. | Safety | AE3 | Summary of Drug-Related Non-<br>Fatal Serious Adverse Events | | 24wk, 48wk |
| 3.18. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product | CS Core | 24wk, 48wk<br>R, RC |

| Safe | ty : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 3.19 | . Safety | AE1 | Summary of Common (>5%) Non-<br>Serious Adverse Events | CS Core FDAAA 'Common' to be defined by study/project team, in accordance with FDAAA requirements. Use >5% cut-off | 24wk, 48wk |
| 3.20 | Safety | EudraCT Non-serious AE<br>AE15 | Summary of Subjects and<br>Number of Occurrences of<br>Common Non-Serious Adverse<br>Events by System Organ Class | CS Core EudraCT For studies with very few events/subjects listing is sufficient. | 24wk, 48wk |
| 3.21 | . Safety | EudraCT SAE<br>AE16 | Summary of Subjects and<br>Number of Occurrences of<br>Serious, Drug-Related Serious,<br>Fatal, and Drug-Related Serious<br>Adverse Events | CS Core EudraCT For studies with very few SAEs/subjects listing is sufficient. | 24wk, 48wk |

| Safe | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| | | AE3 | Summary of Fatal Serious<br>Adverse Events | CS Core<br>GSK CTR | 24wk, 48wk |
| 3.22. | Safety | | | For studies with very few fatal SAEs, listing is sufficient | |
| 3.23. | Safety | AE3 | Summary of Most Frequent<br>Adverse Events by Overall<br>Frequency | | 24wk, 48wk |
| 3.24. | Safety | Shell SAFE_T4 gsk3365791/mid_dori_ph3/week48/drivers/t_ae_cum_er_srd1.sas | Summary of Cumulative Adverse Events by Visit | See DORI | 24wk, 48wk |

| Safe | ty : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| Labo | ratory Values | 5 | | | |
| 3.25. | Safety | Shell SAFE_T5 Use the non standard program in the ARIA study gsk2619619/ing117172/week48/drivers/t_stat_trig_mar.sas | Statistical analysis of Change from Baseline in fasting LDL cholesterol at Weeks 24/48 (Multiple imputations – MAR) | | 24wk, 48wk |
| 3.26. | Safety | Shell SAFE_T6 From ARIA: gsk2619619/ing117172/week48/drivers/t_stat_trig_oc.sas | Statistical analysis of Change from Baseline in fasting LDL cholesterol at Weeks 24/48 by Visit – ANCOVA – Observed Case | | 24wk, 48wk |
| 3.27. | Safety | Shell SAFE_T7 From ARIA gsk2619619/ing117172/week48/drivers/t_stat_trig_locf.sas | Statistical analysis of Change from Baseline in fasting LDL cholesterol at Weeks 24/48 by Visit – ANCOVA – LOCF | | 24wk, 48wk |
| 3.28. | Safety | Shell SAFE_T8 Use the non standard program in the ARIA study gsk2619619/ing117172/week48/drivers/t_stat_trig_mar.sas | Statistical analysis Change from<br>Baseline in fasting TC/HDL ratio<br>at Weeks 24/48 (Multiple<br>imputations – MAR) | Use Shell SAFE_T5 | 24wk, 48wk |
| 3.29. | Safety | Shell SAFE_T9 From ARIA gsk2619619/ing117172/week48/drivers/t_stat_trig_oc.sas | Statistical analysis Change from<br>Baseline in fasting TC/HDL ratio<br>at Weeks 24/48 by Visit -<br>ANCOVA – Observed Case | Use Shell SAFE_T6 | 24wk, 48wk |
| 3.30. | Safety | Shell SAFE_T10 From ARIA gsk2619619/ing117172/week48/drivers/t_stat_trig_locf.sas | Statistical analysis Change from<br>Baseline in fasting TC/HDL ratio<br>at Weeks 24/48 by Visit -<br>ANCOVA – Lipids LOCF | Use Shell SAFE_T7 | 24wk, 48wk |

| Safe | ty : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 3.31. | Safety | Shell SAFE_T11 (Famingo SAS code may be useful - gsk1349572/ing114915/week48/drivers/lb_t_stats_incid_grad2_ldl.sas) | Statistical analysis of Maximum post-Baseline emergent Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Weeks 24/48 | New output | 24wk, 48wk |
| 3.32. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit | CS Core | 24wk, 48wk |
| 3.33. | Safety | LB1 | Summary of Chemistry Changes<br>from Baseline by Visit – Sensitivity<br>Analysis Excluding Suspect<br>Creatinine Samples | CS Core | 24wk, 48wk |
| 3.34. | Safety | LB1 | Summary of Chemistry Changes<br>from Baseline by Visit – Lipids<br>and Glucose in Conventional<br>Units | | 24wk, 48wk |
| 3.35. | Safety | LB1 | Summary of Hematology<br>Changes From Baseline by Visit | CS Core | 24wk, 48wk |
| 3.36. | Safety | Shell SAFE_T12<br>gsk2619619/ing117172/week48/drivers/lb_t_max_tox_rand.sas | Summary of Maximum Post-<br>Baseline Emergent Chemistry<br>Toxicities | CS Core | 24wk, 48wk<br>R, RC |
| 3.37. | Safety | Repeat SAFE_T12 | Summary of Maximum Post-<br>Baseline Emergent Chemistry<br>Toxicities - Sensitivity Analysis<br>Excluding Suspect Creatinine<br>Samples | CS Core | 24wk, 48wk |
| 3.38. | Safety | Shell SAFE_T13 gsk2619619/ing117172/week48/drivers/lb_t_max_tox_haem_rand.sas | Summary of Maximum Post-<br>Baseline Emergent Hematology<br>Toxicities | CS Core | 24wk, 48wk<br>R, RC |

| Safe | ty : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 3.39. | Safety | Shell SAFE_T14<br>gsk2619619/ing117172/week48/drivers/lb_t_ncep_tri.sas | Summary of Changes in NCEP<br>Lipid Baseline Category to<br>Maximum Post-Baseline Category<br>- Triglycerides | | 24wk, 48wk |
| 3.40. | Safety | Shell SAFE_T15 gsk2619619/ing117172/week48/drivers/lb_t_ncep_tot.sas | Summary of Changes in NCEP Lipid Baseline Category to Maximum Post-Baseline Category – Total Cholesterol | | 24wk, 48wk |
| 3.41. | Safety | Shell SAFE_T16 gsk2619619/ing117172/week48/drivers/lb_t_ncep_hdl.sas | Summary of Changes in NCEP<br>Lipid Baseline Category to<br>Maximum Post-Baseline Category<br>– HDL Cholesterol | | 24wk, 48wk |
| 3.42. | Safety | Shell SAFE_T17 gsk2619619/ing117172/week48/drivers/lb_t_ncep_ldl.sas | Summary of Changes in NCEP Lipid Baseline Category to Maximum Post-Baseline Category – LDL Cholesterol | | 24wk, 48wk |
| 3.43. | Safety | VS1 | Summary of Vital Signs | | 24wk, 48wk |
| 3.44. | Safety | VS1 | Summary of Change From<br>Baseline in Vital Signs by Visit | CS Core Will only be produced if post- baseline data collected | 24wk, 48wk |
| 3.45. | Safety | LIVER10 | Summary of Hepatobiliary<br>Laboratory Abnormalities | | 24wk, 48wk |
| 3.46. | Safety | LIVER10 | Summary of Hepatobiliary<br>Laboratory Abnormalities<br>Including the Continuation phase | | 24wk, 48wk<br>RC |

| Safe | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 3.47. | Safety | LIVER1 | Summary of Liver<br>Monitoring/Stopping Event<br>Reporting | If a liver stopping event is reported | 24wk, 48wk |
| 3.48. | Safety | Shell SAFE_T18 gsk3365791/mid_dori_ph3/week48/drivers/t_cssrsib.sas | Summary of C-SSRS Suicidal Ideation or Behaviour during Treatment Excluding Incomplete Calls | Use DORI | 24wk, 48wk |

### 11.18.6.2. Figures

| Safety : | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 3.1. | Safety | AE10 | Plot of Common Adverse Events and Relative Risk | CS CORE | 24wk, 48wk |
| 3.2. | Safety | Shell SAFE_F1 /arenv/arprod/g sk1349572/ing1 14467/wk144/dr ivers/ef_f_cd4cf b_bywk.sas | Line Plot of Adjusted Mean (95% CI) Change From Baseline in Fasting LDL Cholesterol (units) Over Time - Repeated Measure Mixed Model | | 24wk, 48wk |
| 3.3. | Safety | Shell SAFE_F2<br>/arenv/arprod/g<br>sk1349572/ing1<br>14467/wk144/dr<br>ivers/ef_f_cd4cf<br>b_bywk.sas | Line Plot of Adjusted Mean (95% CI) Change From Baseline in Fasting TC/HDL ratio (units) Over Time - Repeated Measure Mixed Model | | 24wk, 48wk |
| 3.4. | Safety | LIVER9 | Scatter Plot of Maximum vs. Baseline for ALT | CS CORE. Add line of equality. | 24wk, 48wk |
| 3.5. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin | CS CORE. Lloyd would like to see theALT on the horizontal axis and Bilirubin on the vertical axis, is it possible to update the standard? | 24wk, 48wk |

| Safety : | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 3.6. | Safety | Shell SAFE_F3<br>/arenv/arprod/g<br>sk2619619/ing1<br>17172/wk48/dri<br>vers/sff_f_bar_t<br>rig.sas | Bar Chart of Triglycerides (mmol/L) NCEP categories at Week 24/48 vs Baseline | Copy from ARIA | 24wk, 48wk |
| 3.7. | Safety | Shell SAFE_F4<br>/arenv/arprod/g<br>sk2619619/ing1<br>17172/wk48/dri<br>vers/sff_f_bar_c<br>hol.sas | Bar Chart of Total Cholesterol (mmol/L) NCEP categories at Week 24/48 vs Basline | | |
| 3.8. | Safety | Shell SAFE_F5<br>/arenv/arprod/g<br>sk2619619/ing1<br>17172/wk48/dri<br>vers/sff_f_bar_<br>hdl.sas | Bar Chart of HDL Cholesterol (mmol/L) NCEP categories at Week 24/48 vs Baseline | | |

| Safety : | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 3.9. | Safety | Shell SAFE_F6<br>/arenv/arprod/g<br>sk2619619/ing1<br>17172/wk48/dri<br>vers/sff_f_bar_I<br>dl.sas | Bar Chart of LDL Cholesterol (mmol/L) NCEP categories at Week 24/48 vs Baseline | | |
| 3.10. | Safety | Shell SAFE_F7 /arenv/arprod/g sk1349572/ing_ psap/trii_iss_m ar/drivers/lb_f_lf t_prof.sas | Liver Chemistry Profile Plots for Subjects with Elevations at Any Post-Baseline Visit | | 24wk, 48wk |

## 11.18.7. **Virology**

### 11.18.7.1. Tables

| Virol | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| Gene | otype | | | | |
| 4.1. | ITT- E | Shell VI_T1<br>gsk1349572/ing111762/week48/drivers/mu_t_gen_acc_48.sas | Summary of Subject<br>Accountability:<br>Genotypes Available | We might want<br>to note the China<br>data in this<br>dataset since is<br>different assay | 24wk, 48wk |
| 4.2. | CVW<br>Genotypic | Shell VI_T2 /arenv/arprod/gsk1349572/ing114467/week48/drivers/mu_t_othmut_emrg.sas | Summary of Treatment<br>Emergent Major<br>Mutations of NRTI,<br>NNRTI and PI Classes | | 24wk, 48wk |
| 4.3. | CVW<br>Genotypic | Shell VI_T3<br>/arenv/arprod/gsk1349572/ing111762/week48/drivers/mu_t_ini_te_pss48.sas | Summary of Pre-<br>specified Treatment<br>Emergent IN<br>Substitutions at Time<br>of Confirmed Virologic<br>Withdrawal | Replace<br>columns:<br>Baseline PSSf to<br>Background<br>Regimen with<br>treatment arms | 24wk, 48wk |

| Viro | logy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>& phase<br>[Priority] |
| 4.4. | CVW<br>Genotypic | Shell VI_T4 /arenv/arprod/gsk1349572/ing111762/week48/drivers/ph_t_bl_geno_gsspdvf_48.sas | Summary of Changes<br>in Genotypic<br>Susceptibility (GSS) to<br>Background ART<br>Therapy at Time of<br>Confirmed Virologic<br>Withdrawal | | 24wk, 48wk |
| Pher | notype | | | | |
| 4.5. | CVW<br>Phenotypic | Shell VI_T5 Arenv/arprod/gsk1349572/ing111762/week48/drivers/mu_t_phen_acc_48.sas | Summary of Subject<br>Accountability:<br>Phenotype Available | | 24wk, 48wk |
| 4.6. | CVW<br>Phenotypic | Shell VI_T6 arenv/arprod/gsk1349572/ing114467/week48/drivers/ph_t_ot_sus_572ral.sas | Summary of Fold Change to DTG and LPV/RTV at Baseline and Time of Confirmed Virologic Withdrawal | | 24wk, 48wk |
| 4.7. | CVW<br>Phenotypic | Shell VI_T7<br>gsk1349572/ing111762/week48/drivers/ph_t_pss_shift_48.sas | Summary of Changes<br>in Phenotypic<br>Resistance (PSS <sub>f</sub> ) to<br>Background ART<br>Regimen at Time of<br>Confirmed Virologic<br>Withdrawal | | 24wk, 48wk |

#### 11.18.8. **Health Outcomes**

### 11.18.8.1. Tables

| Heal | th Outcome | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| HIV- | Treatment Sat | tisfaction Questionnaire | | | |
| | ITT-E | Shell HO_T1 gsk2619619/ing117172/week48/drivers/t_qs_indiv_locf.sas | Summary of HIV-Treatment Satisfaction<br>Questionnaire Individual Item Scores | Modify program to use OC rather than LOCF & include all items from 14-item HIVTSQ. For Health Outcome SUMMARY tables use TU_FREQ | 24wk, 48wk |
| | ITT-E | Shell HO_T2 gsk2619619/ing117172/week48/drivers/t_qs_indiv_locf.sas | Summary of HIV-Treatment Satisfaction Questionnaire Treatment Satisfaction Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T3 gsk2619619/ing117172/week48/drivers/t_qs_indiv_locf.sas | Summary of HIV-Treatment Satisfaction<br>Questionnaire Pain/Discomfort<br>Satisfaction Item Score | Use Shell HO_T2. This is item 12 only. | 24wk, 48wk |
| | ITT-E | Shell HO_T4 | Summary of HIV-Treatment Satisfaction<br>Questionnaire Change from Baseline in<br>Individual Item Scores | Use Shell HO_T2 | 24wk, 48wk |
| | ITT-E | Shell HO_T5 | Summary of HIV-Treatment Satisfaction<br>Questionnaire Change from Baseline in<br>Treatment Satisfaction Score | Use Shell HO_T2 | 24wk, 48wk |
| | ITT-E | Shell HO_T6 | Summary of HIV-Treatment Satisfaction<br>Questionnaire Change from Baseline in<br>Pain/Discomfort Satisfaction Item Score | Use Shell HO_T2 | 24wk, 48wk |

| Heal | Ith Outcome | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| | ITT-E | Shell HO_T7 | Statistical Analysis of HIV-Treatment<br>Satisfaction Questionnaire Change<br>from Baseline in Treatment Satisfaction<br>Score by visit – Repeated Measure<br>Mixed Model Analysis | | 24wk, 48wk |
| | ITT-E | Shell HO_T8 | Statistical Analysis of HIV-Treatment<br>Satisfaction Questionnaire Change<br>from Baseline in Treatment Satisfaction<br>Score at Week 24/48 - Repeated<br>Measures Mixed Model Analysis | | 24wk, 48wk |
| | ITT-E | Shell HO_T9 | Summary of HIV-Treatment Satisfaction<br>Questionnaire in Individual Item Scores<br>Change | Use Shell HO_T1 | 48wk |
| | ITT-E | Shell HO_T10 | Summary of HIV-Treatment Satisfaction Questionnaire in Treatment Satisfaction Score Change | Use Shell HO_T2 | 48wk |
| | ITT-E | Shell HO_T11 | Summary of HIV-Treatment Satisfaction<br>Questionnaire in Pain/Discomfort Item<br>Score Change | Use Shell HO_T2 | 48wk |
| | ITT-E | Shell HO_T12 | Statistical Analysis of HIV-Treatment<br>Satisfaction Questionnaire in Treatment<br>Satisfaction Score Change at Week 48 | New output | 48wk |
| Mori | isky Medicatio | n Adherence Scale – 8 | | | |
| | ITT-E | Shell HO_T13 | Summary of the Morisky 8-Item<br>Medication Adherence Scale - Total<br>Score | | 24wk, 48wk |

| Heal | th Outcome | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| | ITT-E | Shell HO_T14 | Summary of the Morisky 8-Item<br>Medication Adherence Scale -<br>Adherence Level | | 24wk, 48wk |
| | ITT-E | Shell HO_T15 | Statistical Analysis of the Morisky 8-<br>Item Medication Adherence Scale –<br>Adherence Level | New output | 24wk, 48wk |
| Gast | trointestinal Sy | ymptom Rating Scale | | | |
| | ITT-E | Shell HO_T16 | Summary of Gastrointestinal Symptom<br>Rating Scale – Individual Item Scores | | 24wk, 48wk |
| | ITT-E | Shell HO_T17 | Summary of Gastrointestinal Symptom<br>Rating Scale - Diarrhoea Syndrome<br>Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T18 | Summary of Gastrointestinal Symptom<br>Rating Scale – Indigestion Syndrome<br>Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T19 | Summary of Gastrointestinal Symptom Rating Scale Constipation Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T20 | Summary of Gastrointestinal Symptom<br>Rating Scale - Abdominal Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T21 | Summary of Gastrointestinal Symptom<br>Rating Scale – Reflux Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T22 | Summary and Statistical Analysis of<br>Change from Baseline in<br>Gastrointestinal Symptom Rating Scale<br>- Diarrhoea Syndrome Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T23 | Summary and Statistical Analysis of Change from Baseline in Gastrointestinal Symptom Rating Scale | | 24wk, 48wk |

| Hea | Ith Outcome | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| | | | - Indigestion Syndrome Score | | |
| | ITT-E | Shell HO_T24 | Summary and Statistical Analysis of<br>Change from Baseline in<br>Gastrointestinal Symptom Rating Scale<br>Constipation Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T25 | Summary and Statistical Analysis of<br>Change from Baseline in<br>Gastrointestinal Symptom Rating Scale<br>- Abdominal Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T26 | Summary and Statistical Analysis of of Change from Baseline in Gastrointestinal Symptom Rating Scale – Reflux Score | | 24wk, 48wk |
| | ITT-E | Shell HO_T27 | Statistical Analysis of Change from<br>Baseline in Gastrointestinal Symptom<br>Rating Scale - Diarrhoea Syndrome<br>Score at Week 24/48 | | 24wk, 48wk |
| | ITT-E | Shell HO_T28 | Statistical Analysis of Change from<br>Baseline in Gastrointestinal Symptom<br>Rating Scale - Indigestion Syndrome<br>Score at Week 24/48 | | 24wk, 48wk |
| | ITT-E | Shell HO_T29 | Statistical Analysis of Change from<br>Baseline in Gastrointestinal Symptom<br>Rating Scale – Constipation Score at<br>Week 24/48- | | 24wk, 48wk |
| | ITT-E | Shell HO_T30 | Statistical Analysis of Change from Baseline in Gastrointestinal | | 24wk, 48wk |

| Heal | Health Outcome | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| | ITT-E | Shell HO_T31 | Statistical Analysis of Change from<br>Baseline in Gastrointestinal Symptom<br>Rating Scale – Reflux Score at Week<br>24/48 | | 24wk, 48wk |

# 11.18.9. **ICH Listings**

| ICH | : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| Stud | ly Population | | | | |
| 1. | All Subjects<br>Screened | ES7 | Listing of Reasons for Screen Failure | CS CORE | 24wk, 48wk |
| 2. | Randomised | Shell POP_L1 gsk2619619/ing117172/week48/drivers/sa_l_rand_notrt.sas | Listing of Subjects Randomised<br>But Not Treated | CS CORE (related to 'Listing for exclusion from any population) | 24wk, 48wk |
| 3. | Randomised | TA1 | Listing of Randomised and Actual Strata and Treatment Assignment | CS CORE | 24wk, 48wk |
| 4. | ITT-E | ES2 | Listing of Reasons for Study<br>Withdrawal | CS CORE | 24wk, 48wk |
| 5. | ITT-E | SD3 | Listing of Study Treatment Discontinuation Record | | |
| 6. | ITT-E | BL1 | Listing of Subjects for Whom the<br>Treatment Blind Was Broken | CS CORE | 24wk, 48wk |
| 7. | ITT-E | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | CS CORE | 24wk, 48wk |
| 8. | ITT-E | DV2 | Listing of Important Protocol Deviations | CS CORE | 24wk, 48wk |
| 9. | ITT-E | Shell POP_L2 gsk2619619/ing117172/week48/drivers/pd_l_protdev_expp.sas | Listing of Important Protocol Deviations Leading to Exclusion from the Per-Protocol Population | CS CORE | 24wk, 48wk |
| 10. | ITT-E | DM2 | Listing of Demographic Characteristics | CS CORE | 24wk, 48wk |
| 11. | ITT-E | DM9 | Listing of Race | CS CORE | 24wk, 48wk |

| ICH | : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| Effic | асу | | | | |
| 12. | ITT-E | Shell EFF_L1 gsk2619619/ing117172/week48/drivers/l_eff_hivrna.sas | Listing of Qualitative and<br>Quantitative Plasma HIV-1 RNA<br>Data | Include the interpretation of whether the virus is detected or not ('Detected' or 'Not Detected') by the assay | 24wk, 48wk<br>RC |
| 13. | ITT-E | Shell EFF_L2<br>gsk2619619/ing117172/week48/drivers/l_so_01.sas | Listing of Study Outcome (<50 c/mL) at Week X – Snapshot Analysis | | 24wk, 48wk |
| 14. | ITT-E | Shell EFF_L3 gsk2619619/ing117172/week48/drivers/l_so_02.sas | Listing of Study Outcome (<400 c/mL) at Week X – Snapshot Analysis | | 24wk, 48wk |
| Safe | ty | | | | |
| 15. | Safety | HIV_IP5 | Listing of Investigational Product Exposure Data | CS CORE | 24wk, 48wk<br>RC |
| 16. | Safety | HIV_IP5 | Listing of Investigational Product Exposure Data – Mexican Subjects | CS CORE | EOS<br>RC |
| 17. | Safety | AE7 | Listing of Subject Numbers for<br>Individual Adverse Events | CS CORE | 24wk, 48wk<br>RC |
| 18. | Safety | AE8 | Listing of All Adverse Events | CS CORE | 24wk, 48wk<br>RC |
| 19. | Safety | AE8 | Listing of Adverse Events Potentially Related to Torsades de Pointes | | 24wk, 48wk<br>RC |
| 20. | Safety | AE8 | Listing of Fatal Adverse Events | CS CORE | 24wk, 48wk<br>RC |

| ICH | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example Shell | Title | Programming Notes | Deliverable<br>& phase<br>[Priority] |
| 21. | Safety | AE8 | Listing of Fatal Serious Adverse Events | | 24wk, 48wk<br>RC |
| 22. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | CS CORE | 24wk, 48wk<br>RC |
| 23. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product | CS CORE | 24wk, 48wk<br>RC |
| 24. | Safety | AE2 | Listing of Relationship of Adverse<br>Event System Organ Classes,<br>Preferred Terms, and Verbatim<br>Text | CS CORE | 24wk, 48wk<br>RC |
| 25. | Safety | SAE Reasons<br>AE14 | Listing of Reasons for Considering as a Serious Adverse Event | CS CORE<br>FDA | 24wk, 48wk<br>RC |
| 26. | Safety | LB5 | Listing of Clinical Chemistry Laboratory Data for Subjects with Laboratory Abnormalities of Potential Clinical Concern | CS CORE | 24wk, 48wk<br>RC |
| 27. | Safety | LB5 | Listing of Hematology Laboratory Data for Subjects with Laboratory Abnormalities of Potential Clinical Concern | CS CORE | 24wk, 48wk<br>RC |
| 28. | Safety | UR2a | Listing of Urinalysis Data for<br>Subjects with Abnormalities of<br>Potential Clinical Concern | CS CORE | 24wk, 48wk<br>RC |

## 11.18.10. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| Study F | Population | | | · | |
| 29. | All Subjects<br>Screened | Shell POP_L3<br>gsk2619619/ing<br>117172/week48<br>/drivers/sa_I_po<br>p.sas | Listing of Study Populations | | 24wk, 48wk |
| 30. | All Subjects<br>Screened | Shell POP_L4<br>gsk2619619/ing<br>117172/week48<br>/drivers/l_subre<br>c c.sas | Listing of Subject Recruitment by Country and Site Number | | 24wk, 48wk |
| 31. | ITT-E | Shell POP_L5<br>gsk2619619/ing<br>117172/week48<br>/drivers/sa_l_vi<br>sits.sas | Listing of Visit Dates | | 24wk, 48wk<br>RC |
| 32. | ITT-E | Shell POP_L6<br>gsk2619619/ing<br>117172/week48<br>/drivers/lb_l_he<br>ptst.sas | Listing of Hepatitis Test Results | | 24wk, 48wk |
| 33. | ITT-E | CDC3 | Listing of CDC Classification of HIV Infection at Baseline | | 24wk, 48wk |
| 34. | ITT-E | MH2 | Listing of Current and Past Medical Conditions at Baseline | | 24wk, 48wk |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 35. | ITT-E | Shell POP_L7<br>gsk2619619/ing<br>117172/week48<br>/drivers/l_card_<br>risk.sas | Listing of Baseline Cardiovascular Risk Assessment Data | | 24wk, 48wk |
| 36. | ITT-E | Shell POP_L8<br>gsk2619619/ing<br>117172/week48<br>/drivers/l_hist_c<br>ardiac.sas | Listing of History of Cardiac Therapeutic Procedures | | 24wk, 48wk |
| 37. | ITT-E | Shell POP_L9<br>gsk2619619/ing<br>117172/week48<br>/drivers/invp_I_<br>acct.sas | Listing of Investigational Product Accountability | | 24wk, 48wk<br>RC |
| 38. | ITT-E | CM2 | Listing of Concomitant Medications | CS CORE | 24wk, 48wk<br>RC |
| 39. | ITT-E | CM6 | Listing of Relationship Between ATC Level 1, Ingredient and Verbatim Text | | 24wk, 48wk<br>RC |
| 40. | ITT-E | CA3 | Listing of Prior Antiretroviral Therapy | | 24wk, 48wk |
| 41. | ITT-E | CA5 | Listing of Concomitant and Post-treatment Antiretroviral Therapy | | 24wk, 48wk<br>RC |
| 42. | ITT-E | CA5 | Listing of Subjects with Changes in Background Antiretroviral Therapy | | 24wk, 48wk<br>RC |
| 43. | ITT-E | CA7 | Listing of Relationship Between ATC Level 4, Combination, and Verbatim Text for ART | | 24wk, 48wk<br>RC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| Efficac | y | | | | |
| 44. | ITT-E | Shell EFF_L4<br>gsk2619619/ing<br>117172/week48<br>/drivers/lb_cd4c<br>c.sas | Listing of CD4+ Cell Count Data | | 24wk, 48wk<br>RC |
| 45. | ITT-E | HIV4 | Listing of HIV-1 Associated Conditions | | 24wk, 48wk<br>RC |
| 46. | ITT-E | Shell EFF_L5<br>gsk1349572/ing<br>111762/week48<br>/drivers/ef_I_hv<br>1rn_olpdvf.s | Listing of Viral Load over time for Subjects with Confirmed Virologic Withdrawal Criteria | Other Listing 71 from SAILING | 24wk, 48wk |
| 47. | ITT-E | Shell EFF_L6<br>gsk1349572/ing<br>111762/week48<br>/drivers/ef_I_hv<br>1rn_olpdvf.s | Listing of Viral Load over time for Subjects with Confirmed Virologic Withdrawal Criteria During the Continuation Phase | Other Listing 71 from SAILING | 24wk, 48wk<br>RC |

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 48. | ITT-E | Shell EFF_L7 Listing 48 - gsk2619619/ing 117172/week48 /drivers/ef_I_cv w.sas Listing 77 - gsk2619619/in g117172/week 48/drivers/mu _I_geno_resist .sas | Listing of Viral Load over time for Subjects with on-treatment virology results at non-CVWC timepoints | Use non-ICH listing 48 (for the format) and 77 (for the subjects to be included) | 24wk, 48wk<br>RC? |
| 49. | ITT-E | Shell EFF_L8<br>gsk1349572/ing<br>111762/week48<br>/drivers/mu_t_vl<br>cd4_pdvf.sas | Plasma HIV-1 RNA and CD4+ Cell Count at Confirmed Virologic Withdrawal Criteria | Use table 12.60, update as a listing, update population and program name | 24wk, 48wk<br>RC? |

| Non-IC | Non-ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| Safety | | | | | |
| 50. | Safety | AE8 | Listing of Non-Serious AEs of Mexican Subjects | | EOS, RC |
| 51. | Safety | AE8 | Listing of SAEs of Mexican Subjects | | EOS, RC |
| 52. | Safety | AE8 | Listing of SAEs of non-Mexican Subjects | | EOS, RC |
| 53. | Safety | PREG1a | Listing of Subjects Who Became Pregnant During the Study | | 24wk, 48wk<br>RC |
| 54. | Safety | LB5 | Listing of Clinical Chemistry Data | | 24wk, 48wk<br>RC |
| 55. | Safety | LB5 | Listing of Hematology Data | | 24wk, 48wk<br>RC |
| 56. | Safety | LB5 | Listing of Laboratory Data for Subjects with Grade 3 or 4 Post-Baseline Emergent Toxicities | See for the shell arenv/arprod/gsk1349572/ing11176 2/week48/drivers/lb maxaltbil.sas | 24wk, 48wk<br>RC |
| 57. | Safety | LB5 | Listing of Urinalysis Concentration Data | | 24wk, 48wk<br>RC |
| 58. | Safety | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory Criteria<br>Post-Baseline | | 24wk, 48wk<br>RC |
| 59. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | If a liver stopping event is reported | 24wk, 48wk<br>RC |
| 60. | Safety | Shell SAFE_L1<br>gsk2619619/ing<br>117172/week48<br>/drivers/lb_l_ma<br>xaltbil.sas | Listing of Post Baseline Maximum ALT and Maximum Bilirubin | | 24wk, 48wk<br>RC |
| 61. | Safety | EG5 | Listing of ECG Findings | Only collected for CV events | 24wk, 48wk<br>RC |

| Non-IC | Non-ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 62. | Safety | VS4 | Listing of Vital Signs | | 24wk, 48wk<br>RC |
| 63. | Safety | ABC_HSR<br>_EXPO2 | Listing of Abacavir Hypersensitivity Reaction Record - Exposure to Abacavir | | 24wk, 48wk<br>RC |
| 64. | Safety | ABC_HSR<br>DRUG2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject History of Drug Allergies | | 24wk, 48wk<br>RC |
| 65. | Safety | ABC_HSR<br>COND2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject and Family Conditions | | 24wk, 48wk<br>RC |
| 66. | Safety | ABC_HSR<br>RASH2 | Listing of Abacavir Hypersensitivity Reaction Record - Skin Rash Details | | 24wk, 48wk<br>RC |
| 67. | Safety | ABC_HSR<br>SYMP4 | Listing of Abacavir Hypersensitivity Reaction Record - Symptoms | | 24wk, 48wk<br>RC |
| 68. | Safety | VS4 | Listing of Abacavir Hypersensitivity Reaction Record - Vital Signs | | 24wk, 48wk<br>RC |
| 69. | Safety | ABC_HSR<br>_SYMP6 | Listing of Abacavir Hypersensitivity Reaction Record - Individual Symptoms and Diagnostic Category Assignments (Excluding Other Symptoms) | | 24wk, 48wk<br>RC |
| 70. | Safety | ABC_HSR<br>_SYMP7 | Listing of Abacavir Hypersensitivity Reaction Record - Individual Symptoms and Diagnostic Category Assignments (Other Symptoms) | | 24wk, 48wk<br>RC |
| 71. | Safety | LIVER5 | Listing of Liver Event Results and Time of Event Relative to<br>Treatment | | 24wk, 48wk<br>RC |
| 72. | Safety | LIVER6 | Listing of Liver Event Information for RUCAM Score | | 24wk, 48wk<br>RC |
| 73. | Safety | LIVER7 | Listing of Liver Biopsy Details | | 24wk, 48wk<br>RC |
| 74. | Safety | LIVER8 | Listing of Liver Imaging Details | | 24wk, 48wk<br>RC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 75. | Safety | MH2 | Listing of Past and Current Liver Disease Medical Conditions | | 24wk, 48wk |
| 76. | Safety | LB5 | Listing of Laboratory Data from Liver Event Follow-Up | | 24wk, 48wk<br>RC |
| Virolog | Virology | | | | |
| 77. | ITT-E | Shell VI_L1<br>gsk1349572/ing<br>111762/week48<br>/drivers/mu_I_g<br>eno_all.sas | Listing of All Genotypic Data | Baseline and on study genotypes are MAINLY Monogram, but some Q2 will be in there. We need to note when it is from Q2 versus Monogram to assist with potential subtle differences in how the resistance data is annotated and provided | 24wk, 48wk<br>RC |
| 78. | ITT-E | Shell VI_L2<br>gsk1349572/ing<br>111762/week48<br>/drivers/ph_I_ph<br>eno_all.sas | Listing of All Phenotypic Data | | 24wk, 48wk<br>RC |
| 79. | All Subjects<br>Screened | Shell VI_L3 gsk1349572 /ing111762 /week48/dr ivers/mu_l _geno_all. sas | Listing of All Screening Genotype Data from Quest | New (study specific) | 24wk, 48wk |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 80. | ITT-E | Shell VI_L4<br>gsk1349572/ing<br>111762/week48<br>/drivers/mu_t_vi<br>rology_pdvf | Listing of Genotypic and Phenotypic Data for Subjects with Confirmed Virologic Withdrawal Criteria | Use T12.59 from SAILING. Update as a listing and also title and population Potentially different assays,phenotypic assay for RT PRO and Integrase. Can we identify this in the listing | 24wk, 48wk<br>RC |
| 81. | ITT-E | Shell VI_L5<br>gsk1349572/ing<br>111762/week48<br>/drivers/mu_t_vi<br>rology_pdvf.sas | Listing of Genotypic and Phenotypic Data for Subjects with Confirmed Virologic Withdrawal Criteria During the Continuation Phase | Use T12.59 from SAILING. Update as a listing and also title and population | 24wk, 48wk<br>C |
| 82. | ITT-E | Shell VI_L6<br>gsk1349572/ing<br>111762/week48<br>/drivers/mu_t_vi<br>rology_last | Listing of Genotypic and Phenotypic Data for Subjects with ontreatment virology results at non-CVW timepoints | Use T12.59 from SAILING. Update as a listing and also title and population | 24wk, 48wk<br>RC |
| 83. | ITT-E | Shell VI_L7<br>gsk1349572/ing<br>111762/week48<br>/drivers/ph_I_ph<br>eno_bg_pdvf.sa<br>s | Subject Level Summary of Key Virologic Data for Subjects with Confirmed Virologic Withdrawal or Last On-treatment VL >400 c/mL | As in Table 12.62 (SAILING) but add columns for DTG FC, LPV FC, IN substitutions, Major PI mutations, mutations, Major NRTI, Major NNRTI mutations; flag for CVW/Last VL >400. | |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| Health | Health Outcome Listings | | | | |
| 84. | ITT-E | Shell HO_L1<br>gsk2619619/ing<br>117172/week48<br>/drivers/l_hivtre<br>at_sat.sas | Listing of HIV-Treatment Satisfaction Questionnaire in Individual Item Scores and Treatment Satisfaction Score | Use TU_LIST for all Health Outcome Listings Change SAS program to exclude Lifestyle Ease Score and General Satisfaction Clinical Score | 24wk, 48wk |
| 85. | ITT-E | Shell HO_L2<br>gsk2619619/ing<br>117172/week48<br>/drivers/l_hivtre<br>at_sat.sas | Listing of HIV-Treatment Satisfaction Questionnaire in Individual Item Scores Change and Treatment Satisfaction Score Change | Modify program to use HIVTSQc | 48wk |
| 86. | ITT-E | Shell HO_L3 | Listing of Morisky 8-Item Medication Adherence Scale Individual Items, Total Score and Adherence Level | New output but can use TSQ listing SAS code – Shell HO_L1 | 24wk, 48wk |
| 87. | ITT-E | Shell HO_L4 | Listing of Gastrointestinal Symptom Rating Scale – Individual Item Scores | New output but can use TSQ listing SAS code – Shell HO_L1 | 24wk, 48wk |
| 88. | ITT-E | Shell HO_L5 | Listing of Gastrointestinal Symptom Rating Scale - Syndrome Scores | New output but can use TSQ listing SAS code – Shell HO_L1 | 24wk, 48wk |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable & phase [Priority] |
| 89. | | | Patient profiles for subjects meeting protocol defined liver stopping criteria, | Example in /arenv/arprod/gsk1349572/ing_idmc /interim1/drivers/dm_l_patproflist2.s as or /arwork// <study>/profiles/profile.s as Include: Investigator, country, tmt, sex, DOB, age, race, medical history, IP start and end date, reasons for discontinuation, AE, conmeds, prior ART, labs, viral loads, vital signs.</study> | 24wk, 48wk |
| 90. | | | Patient profiles for subjects with virological failures | | 24wk, 48wk |